Official Title: A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN

NCT Number: NCT02510261

Document Date: Protocol, Version 3.0, 05 January 2017

# **Protocol Administrative Change 2**

#### ALN-TTR02-006

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### Purpose:

As noted in protocol version 3.0 dated 05 January 2017, skin punch biopsies of the thigh and leg for evaluation of intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD) will be collected at the 52 Week visit, and annually thereafter. The samples have been and are being quantified through stereologic evaluation of the immunostained nerve fibers.

This letter is to clarify that skin punch biopsies collected under this protocol will also be stained for amyloid to determine amyloid burden. Characterization of amyloid burden will serve as an additional exploratory assessment. Amyloid burden assessment will be performed on all collected skin punch biopsies by the same laboratory performing the IENFD and SGNFD assessments.

As the study-specific informed consent form (ICF) does not describe the specific analyses being performed on these biopsies, and as such, the ICF does not require any updating.

The changes in the protocol are specified below; added text is indicated by **bold** font:

# <u>Section 8.1.3: Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density, Page 37</u>

For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD and amyloid burden characterization will be obtained at each time point.

| PPD | |
|-----|-------------|
| | 02 may 2017 |
| | Date |

# PATISIRAN (ALN-TTR02)

### **ALN-TTR02-006**

A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN

Protocol Version:

Version 3.0 (Incorporating Amendment 2)

Protocol Date

05 January 2017

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

# **INVESTIGATOR'S AGREEMENT**

I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

# **Version History:**

| Version Number | Date | Comment |
|---|---|---|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 – Global | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 – Japan | 14 October 2015 | Incorporating Japan-specific Amendment 1 |
| 2.1 – Taiwan | 10 December 2015 | Incorporating Taiwan-specific Amendment 1 |
| 2.1 – France/Germany | 17 December 2015 | Incorporating France/Germany-specific |
| | | Amendment 1 |
| 2.2 – Japan | 14 March 2016 | Incorporating Japan-specific Amendment 2 |
| 3.0 - Global | 05 January 2017 | Incorporating Global Amendment 2 (including |
| | | Japan-, Taiwan- and France/Germany-specific |
| | | changes) |

## **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

# **Name of Investigational Product:**

Patisiran

## Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

## **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

## Methodology:

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 (±3) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days. Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm 5$ ) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and vearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may

occur if deemed necessary by the study personnel.

## Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤2 x ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

## Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

## **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography (as regionally applicable)
- Cardiac structure and function through echocardiograms and serum levels of terminal

prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid stimulating hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; ophthalmology examinations; and assessment of suicidal ideation and behavior.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | X° | X° |
| Weight | | Prior 1 | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | X <sup>d</sup> | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | | $[X]^{f}$ |
| Vital Signs <sup>g</sup> | | Prior t | X<br>to Each Dose | | | | |
| Safety Laboratory Assessments <sup>h</sup> | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | X <sup>i</sup> | | X | X | X | X | X |
| C-SSRS Questionnaire | | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TTR Protein (ELISA) | X <sup>d</sup> | | X | X | X | X | X |
| TSH and Vitamin A | | | | X | X | Xº | Xº |
| Blood Sample for Long-term Storage | X | X | X | X | X | X | X |
| mNIS+7 <sup>j</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS+7 <sup>k</sup> | X <sup>d</sup> | | | X | | | $[X]^f$ |
| NIS only | | | | | X <sup>l</sup> | X <sup>m</sup> | X <sup>m</sup> |
| Grip Strength Test <sup>n</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| 10-Meter Walk Test <sup>p</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| Ophthalmology Examination <sup>q</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>r</sup> | | | | X | X | X° | Xº |
| MR Neurography <sup>s</sup> (Germany & France only) | X | | X | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | X° | Xº |
| Norfolk QOL-DN <sup>t</sup> | X <sup>d</sup> | | | X | X | X° | Xº |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| EQ-5D QOL | $X^d$ | | | X | X | X° | X° |
| Echocardiogram | $X^{d,u}$ | | | X | | | $[X]^f$ |
| Troponin I and NT-proBNP | $X^d$ | | | X | | | $[X]^{f}$ |
| Anti-Drug Antibody Testing <sup>v</sup> | | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Premedication / Patisiran Administration <sup>w</sup> | X | X | | | | | |
| Phone Contact <sup>x</sup> (In applicable regions only) | | | X | | | | |
| Adverse Events | X <sup>b</sup> Continuous Monitoring | | | | | | |
| Concomitant Medications | X <sup>b</sup> Continuous Monitoring | | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: C-SSRS = Columbia-Suicide Severity Rating Scale; COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- a. Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- b. Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- c. Assessment does not need to be repeated. Information will be obtained from parent study.
- d. Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- e. mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f. Assessment/procedure required only if patient withdraws before the 52-week visit.
- g. Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- h. Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- i. Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.


- j. The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- k. The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- 1. One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- m. Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- n. Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- o. Assessment does not need to be repeated if done within the previous 26 weeks.
- p. The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- q. Examination will include visual acuity, visual fields, and slit-lamp evaluation. An electroretinogram may also be performed, as described in Section 9.1.6
- r. Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- s. MR neurography will only be conducted at sites in Germany and France. In these countries, neurography may be conducted for patients who had MR neurography in the parent study and for a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Patients who had imaging in the parent study should have Day 0 imaging if they did not undergo MR neurography within the past 3 months.
- t. Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- u. Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- v. Serum samples for anti-drug antibodies will be collected as specified.
- w. Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study in the 21 (±3) day timeframe. Doses may be administered at the clinical site or, where applicable country and local regulations allow, at home by a healthcare professional trained in the protocol.
- x. Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use. During phone contact, patients may also be asked additional questions about their general experience receiving infusions at home.


# **TABLE OF CONTENTS**

# SYNOPSIS3

| TABLE | OF CONTENTS | 11 |
|---|---|---|
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| • | Infusion-Related Reactions | 20 |
| • | Liver function test abnormalities | 20 |
| • | Vitamin A Lowering | 20 |
| • | Osteoporosis | 20 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |

| 6.1. | Study Drug Packaging and Labeling | 31 |
|---|---|---|
| 6.2. | Study Drug Storage | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |
| 6.4.1. | Premedication | 32 |
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | |
| 8.1.4. | Magnetic Resonance Neurography (Germany and France Only) | |
| 8.1.5. | Modified Body Mass Index | |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test. | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | |
| 8.1.11. | Rasch-built Overall Disability Scale | |
| 8.1.12. | Pharmacoeconomics Questionnaire | 39 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | |
| 8.1.15. | Thyroid-Stimulating Hormone | 39 |
| 8.1.16. | Vitamin A | 39 |
| 8.1.17. | Anti-Drug Antibodies | 39 |

| 8.1.18. | Blood Sample for Long-term Storage | 39 |
|----------|-------------------------------------------|----|
| 9. | ASSESSMENT OF SAFETY | 41 |
| 9.1. | Safety Parameters | 41 |
| 9.1.1. | Demographic and Medical History | 41 |
| 9.1.2. | Vital Signs | 41 |
| 9.1.3. | Weight and Height | 41 |
| 9.1.4. | Physical Examination | 41 |
| 9.1.5. | Laboratory Assessments | 41 |
| 9.1.5.1. | Hematology | 42 |
| 9.1.5.2. | Blood Chemistry | 42 |
| 9.1.5.3. | Urinalysis | 42 |
| 9.1.5.4. | Coagulation | 43 |
| 9.1.5.5. | Pregnancy Screen | 43 |
| 9.1.6. | Ophthalmology Examination | 43 |
| 9.1.7. | Columbia-Suicide Severity Rating Scale | 43 |
| 9.2. | Adverse Events and Serious Adverse Events | 43 |
| 9.2.1. | Definition of Adverse Events | 43 |
| 9.2.1.1. | Adverse Event | 43 |
| 9.2.1.2. | Serious Adverse Event | 43 |
| 9.3. | Relationship to Study Drug | 44 |
| 9.4. | Recording Adverse Events | 44 |
| 9.5. | Reporting Adverse Events | 45 |
| 9.5.1. | Serious Adverse Event Reporting. | 45 |
| 9.5.2. | Pregnancy Reporting | 47 |
| 10. | STATISTICS | 48 |
| 10.1. | Sample Size | 48 |
| 10.2. | Statistical Methodology | 48 |
| 10.2.1. | Populations to be Analyzed | 48 |
| 10.2.2. | Baseline Evaluations | 48 |
| 10.2.3. | Efficacy Analyses | 48 |
| 10.2.4. | Safety Analyses | 49 |
| 10.2.5. | Healthcare Utilization Assessments | 49 |

| 10.2.6. | Interim Analysis | 49 |
|---------|--------------------------------------------|----|
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 50 |
| 11.1. | Study Monitoring | 50 |
| 11.2. | Audits and Inspections | 50 |
| 11.3. | Institutional Review Board | 50 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 51 |
| 13. | ETHICS | 52 |
| 13.1. | Ethics Review | 52 |
| 13.2. | Ethical Conduct of the Study | 52 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 52 |
| 13.3. | Written Informed Consent | 53 |
| 13.4. | Compensation for Health Damages | 53 |
| 14. | DATA HANDLING AND RECORD KEEPING | 54 |
| 14.1. | Case Report Forms | 54 |
| 14.2. | Confidentiality | 54 |
| 14.3. | Inspection of Records | 55 |
| 14.4. | Retention of Records | 55 |
| 15. | PUBLICATION POLICY | 56 |
| 16. | LIST OF REFERENCES | 57 |
| 17. | APPENDICES | 58 |

# LIST OF TABLES

| Tabla 1 | Schedule of Assessments | ranga da kanana da k |
|---|---|---|
| Table I | Schedille of Assessments | , and the same of the same |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RBP | retinol binding protein |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WT | wild type |

## 1. INTRODUCTION

## 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

## 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran Investigator's Brochure.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

## 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

## • Vitamin A Lowering

The suppression of serum levels of TTR and retinol binding protein (RBP) is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

## Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone

mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the Investigator's Brochure.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

# 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study. Patients in this study will have completed "parent" study ALN-TTR02-003 or ALN-TTR02-004. Note that Study ALN-TTR02-003 is not being conducted in Japan.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 \ (\pm 3)$  days. Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30 \ (\pm 5)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments

after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

# 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor (Alnylam Pharmaceuticals, Inc).

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or Medpace, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

## 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

# 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

# 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study

conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

In Japan it is recommended that the Investigators select appropriate contraception methods, as available.

Pregnancy reporting guidelines are provided in Section 9.5.2.

# 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

# **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan, the clinical sites will provide patients with a prescription for vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or (in applicable regions) trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

# 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

# 6. STUDY DRUG MATERIALS AND MANAGEMENT

# 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

## 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

## **6.4.2.** Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every  $21 (\pm 3)$  days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A . Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan the clinical sites will provide the subjects with a prescription for vitamin A..

## 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower

infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - 1) If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The Investigator or designee (or in Japan, the responsible pharmacist designated according to the Japan local regulations) will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

# 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.
# 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

# 8. ASSESSMENT OF EFFICACY

# 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place at the CAS. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

# 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

# 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

#### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

# 8.1.4. Magnetic Resonance Neurography (Germany and France Only)

Magnetic resonance (MR) neurography will only be performed at sites in Germany and France. Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity may be imaged for patients in Germany and France who have previously had MR neurography in the parent study and for a subset of patients providing informed consent who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

# 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

# 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

# 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

# 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

# 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

## 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

# 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

## 8.1.12. Pharmacoeconomics Ouestionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

# 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

# 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

## **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.16. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A

## 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1.

## 8.1.18. Blood Sample for Long-term Storage

To permit exploratory investigations and the application of novel approaches to bioanalysis that may further elucidate the outcomes of this study, or potentially advance understanding of the safety, mechanism of action and/or efficacy of patisiran, blood samples will be collected for long-term storage. These samples will be securely stored in a central biorepository for up to 10

years following the last patient last visit in this clinical study. After 10 years have elapsed, samples will be destroyed.

Details regarding the collection, processing, storage, and shipping of samples will be provided in the Laboratory Manual.

Exploratory analysis of these biospecimens will be performed by Alnylam Pharmaceuticals or its designees.

All study participants will be advised during the informed consent process of these biobanking details and the potential for exploratory investigation of their samples. Those who do not wish to contribute specimens to the biorepository will be asked to sign an "opt out" form. Moreover, patients who subsequently decide to withdraw consent for the utilization of such stored samples will be able to do so, with the understanding that any data arising from samples already analyzed will be the property of Alnylam Pharmaceuticals.

# 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

# 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

# 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

## 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

## 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

#### 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

# 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

# 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

# **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

# 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

# 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

# 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

# 9.1.7. Columbia-Suicide Severity Rating Scale

The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess each patient's mental status as it relates to suicidal ideation and behavior.

## 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs.

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

## 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.

Medpace SAE hotline – USA:

Telephone: PPD ext. PPD or PPD ext. PPD

Facsimile: PPD or PPD

Medpace SAE hotline – Europe:

Telephone: PPD

Facsimile: PPD

Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that

transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

# 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

# 10. STATISTICS

# 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

# 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### **10.2.2.** Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

## 10.2.3. Efficacy Analyses

Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory

and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

## 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

A listing of healthcare utilization data will be presented.

## 10.2.6. Interim Analysis

Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

# 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator and the site will permit study-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

# 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

# 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

The Investigator should not start any study procedure with the patient until documentation of the approval by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator and Alnylam Pharmaceuticals, Inc.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Medical Association Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA) in the US, and all other applicable medical privacy laws and regulations.

#### 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

# 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

# 13.4. Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required per local regulations.

## 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

# 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

# 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| necucu. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

# **Appendix 2: New York Heart Association Classification of Heart Failure**

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

# **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

# **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (18.6)^a$ |
| | | <ul> <li>Sural SNAP, tibial motor n. distal latency, peroneal<br/>CMAP/motor n. conduction velocity/motor n. distal<br/>latency</li> </ul> |
| | | • Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (10)^a$ |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | • Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

#### ALN-TTR02-006 Protocol Amendment 2

Summary of Changes (dated 05 January 2017) compared to Protocol Amendment 1 (dated 08 September 2015)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

## **Rationale for Protocol Amendment**

The primary purpose of this amendment is to add the Columbia-Suicide Severity Rating Scale (C-SSRS) to the study assessments, which was inadvertently left out of previous versions of the protocol. The inclusion of the C-SSRS addresses a regulatory requirement to prospectively assess suicidality in clinical trials involving all drugs for neurological indications. Overall, this amendment includes the following changes:

- The Columbia-Suicide Severity Rating Scale has been added as an assessment of suicidal ideation and behavior.
- Country-specific versions of the protocol have been integrated in order to increase consistency in the execution of the clinical study globally
- Electroretinograms are now recommended to be performed in the case of suspected retinal disease.
- The premedication regimen has been updated to align with commercially available doses.
- Blood samples for long-term storage have been added in order to permit future exploratory investigations.
- During scheduled phone contact, clinical sites may now ask patients who are receiving home infusions about their general experience receiving these infusions

A detailed summary of the above changes, in addition to changes made for clarity, is provided in Table 1. Corrections to abbreviations, typographical errors and formatting are not detailed.

# Table 1: Protocol Amendment 2 Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose: Added Columbia-Suicide Severity Rating Scale to the study assessments

The primary change occurs in Table 1 Schedule of Assessments

Added text: Added row to Schedule of Assessments indicating that the Columbia-Suicide Severity Rating Scale is to be

collected at 26 weeks and 52 weeks after baseline and annually thereafter, as well as at the End of Study and Early

Withdrawal visits.

Section(s) also containing this change or similar changes:

• Synopsis, Criteria for Evaluation, Safety

• Section 9.1.7 Columbia-Suicide Severity Rating Scale (section added)

Purpose: As part of global protocol integration, specified that home infusions are allowed only where applicable country and local regulations allow.

The primary change occurs in Section 3.1 Overall Study Design

Added text: After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 (±3) days, or.

Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a

healthcare professional trained on the protocol and delivery of premedications and patisiran.

Section(s) also containing this change or similar changes:

- Synopsis, Methodology
- Table 1, Schedule of Assessments
- Section 5.3 Treatment Compliance
- Section 6.4.2 Study Drug Administration

Purpose: As part of global protocol integration, specified that MR neurography is only to be conducted in Germany and France

The primary change occurs in Table 1 Schedule of Assessments, footnote s

Now reads:

Required only forMR neurography will only be conducted at sites in Germany and France. In these countries, neurography may be conducted for patients who had MR neurography in the parent study and may be imaged for consentingfor a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Patients who had imaging in the parent study should have Day 0 imaging if they did not undergo MR neurography within the past 3 months.

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for evaluation, Efficacy
- Section 8.1 Efficacy Parameters
- Section 8.1.4 Magnetic Resonance Neurography (Germany and France Only) (Section has been added)

Purpose: As part of global protocol integration, specified which studies patients may roll in from, and that the ALN-TTR02-003 study is not being conducted in Japan.

The primary change occurs in Section 3.1 Overall Study Design

Added text: Patients in this study will have completed "parent" study ALN-TTR02-003 or ALN-TTR02-004. Note that Study ALN-TTR02-003 is not being conducted in Japan.

Purpose: As part of global protocol integration, added Japan-specific recommendations regarding contraception.

The primary change occurs in Section 4.4 Pregnancy and Breastfeeding Restrictions / Contraception Requirements

Added text: In Japan it is recommended that the Investigators select appropriate contraception methods, as available.

Purpose: As part of global protocol integration, added Japan-specific instructions regarding duties related to study drug accountability.

The primary change occurs in Section 6.5 Study Drug Accountability

Added text: The Investigator or designee (or in Japan, the responsible pharmacist designated according to the Japan local

regulations) will maintain accurate records of receipt and the condition of the patisiran supplied for this study,

including dates of receipt.

Purpose: As part of global protocol integration, added statement on compensation for health damages as per local regulations.

The primary change occurs in Section 13.4 Compensation for Health Damages (section added)

Added text:

# 13.4 Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required per local regulations

Purpose: To update premedication regimen so that it aligns with commercially available doses.

The primary change occurs in Section 6.4.1 Premedication

Now reads: Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site).

Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg

PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Section(s) also containing this change or similar changes:

• Synopsis, Investigational product, dosage and mode of administration

Purpose: Added recommendation to collect an electroretinogram in the case of suspected retinal injury

The primary change occurs in Section 9.1.6 Ophthalmology Examination

Added text:

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Updated description of statistical analysis to align with currently planned analytic approach.

The primary change occurs in Section 10.2.3 Efficacy Analyses

Now reads:

Efficacy analyses will examine between and within patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm$ SE) values over time for each location (hip, knee, etc.).

Section(s) also containing this change or similar changes:

- Synopsis, Statistical Methods
- Section 10.2.5 Healthcare Utilization Assessments
- Section 10.2.6 Interim Analysis

Purpose: Added blood sampling for long-term storage in order to permit future exploratory investigations.

The primary change occurs in Table 1 Schedule of Assessments

Added text:

Added row to Schedule of Assessments indicating a blood sample for long-term storage is to be collected at each clinic visit.

Section(s) also containing this change or similar changes:

• Section 8.1.18 Blood Sample for Long-term Storage (section added)

Purpose: Added questionnaire regarding experience of home infusions to scheduled phone contact for home infusion patients.

The primary change occurs in Table 1 Schedule of Assessments, footnote x

Added text: x. Patients who are receiving pat

x. Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every  $30 \ (\pm 5)$  days for assessment of adverse events and concomitant medication use. **During phone contact, patients** may also be asked additional questions about their general experience receiving infusions at home.

Purpose: Added a definition of "woman of child-bearing potential".

The primary change occurs in Section 4.4 Pregnancy and Breastfeeding Restrictions / Contraception Requirements

Added text:

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

Purpose: Clarified language on Vitamin A dosing and added Japan-specific instructions.

The primary change occurs in Section 5.2 Concomitant Medications

Now reads:

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan, the clinical sites will provide patients with a prescription for vitamin A

Section(s) also containing this change or similar changes:

- Section 6.4.2 Study Drug Administration
  - Section 8.1.16 Vitamin A

Purpose: Clarified procedures for efficacy assessments, adding the location at which to conduct assessments, and removing specified duration.

The primary change occurs in Section 8.1 Efficacy Parameters

Now reads: Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days at the CAS.

Purpose: Removed language indicating that anti-drug antibodies would only be analyzed if clinically indicated.

The primary change occurs in Section 8.1.17 Efficacy Parameters

Deleted text: Serum samples for anti-drug antibodies will be collected as specified in Table 1.—Samples may be analyzed, if

clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Clarified that no study procedures may occur until approval is granted by all appropriate parties.

The primary change occurs in Section 13.1 Ethics Review

Added text: The Investigator should not start any study procedure with the patient until documentation of the approval

by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator

and Alnylam Pharmaceuticals, Inc.

# PATISIRAN (ALN-TTR02)

# **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN


Version 2.0 (Incorporating Amendment 1)

Protocol Date

08 September 2015

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



Date

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.
### **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agramaintain the confidentiality of all information received or developed in connection with this protocol. |
|---|
| Printed Name of Investigator |
| Signature of Investigator |

### **Version History:**

Date

|----------------|-------------------|----------------------------------|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |

### **SYNOPSIS**

### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

#### Name of Investigational Product:

Patisiran

#### Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

### **Methodology:**

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study. Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 (±3) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study. unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0. After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm 5$ ) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

### Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

### Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

### Reference therapy, dosage and mode of administration:

Not applicable.

#### Criteria for evaluation:

### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography

- Cardiac structure and function through echocardiograms and serum levels of terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I
- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid Stimulating Hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of anti-drug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | Xº | Xº |
| Weight | | Prior t | X<br>o Each Dose | | | Xº | Xº |
| mBMI <sup>e</sup> | X <sup>d</sup> | | | X | X | Xº | Xº |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | X <sup>d</sup> | | | X | X | Xº | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | $[X]^f$ | $[X]^{\mathrm{f}}$ |
| Vital Signs <sup>g</sup> | | Prior t | X<br>o Each Dose | | | | |
| Safety Laboratory Assessmentsh | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | X <sup>k</sup> | | X | X | X | X | X |
| TTR Protein (ELISA) | X | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TSH and Vitamin A | | | | X | X | Xº | Xº |
| mNIS+7 <sup>1</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS+7 <sup>m</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS only | | | | | X <sup>n</sup> | $X^{n,p}$ | X <sup>n,p</sup> |
| Grip Strength Test <sup>q</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| 10-Meter Walk Test <sup>r</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| Ophthalmology Examination <sup>s</sup> | X <sup>d</sup> | | | X | X | Xº | Xº |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | | X | X | Xº | Xº |
| MR Neurography <sup>u</sup> | | | | X | X | Xº | Xº |
| Pharmacoeconomics Questionnaire | X | | | X | X | Xº | Xº |
| Norfolk QOL-DN <sup>v</sup> | X <sup>d</sup> | | | X | X | Xº | Xº |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | [X] <sup>f</sup> | $[X]^f$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | Xº | Xº |
| Echocardiogram | $X^{d,w}$ | | | X | | $[X]^{\mathrm{f}}$ | $[X]^f$ |
| Troponin I and NT-proBNP | X <sup>d</sup> | | | X | | $[X]^{\mathrm{f}}$ | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>x</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration | X <sup>y</sup> | | X <sup>y</sup> | • | | | |
| Phone Contact | | | Xz | | | | |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Adverse Events | X <sup>b</sup> Continuous Monitoring | | | | | | |
| Concomitant Medications | X <sup>b</sup> Continuous Monitoring | | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- <sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- <sup>d</sup> Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- <sup>e</sup> mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- $^{\rm f}$  Assessment/procedure required only if patient withdraws before the 52-week visit.
- <sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- <sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- k Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.
- The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on

79

separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.

- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- P Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.
- Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- <sup>u</sup> Required only for patients who had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in their parent study.
- <sup>v</sup> Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- w Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>x</sup> Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- y Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study within the 21 (±3) days timeframe. Doses may be administered at the clinical site or at home by a healthcare professional trained in the protocol.
- <sup>z</sup> Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use.

### **TABLE OF CONTENTS**

| SYNOP | SIS | 3 |
|---|---|---|
| TABLE | OF CONTENTS | 11 |
| LIST OF | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 1.4.1. | Infusion-Related Reactions. | 20 |
| 1.4.2. | Vitamin A Lowering | 20 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage | 31 |

| 6.3. | Study Drug Preparation | 31 |
|---|---|---|
| 6.4. | Administration | 32 |
| 6.4.1. | Premedication | 32 |
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | 37 |
| 8.1.4. | Magnetic Resonance Neurography | 37 |
| 8.1.5. | Modified Body Mass Index | 38 |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.11. | Rasch-built Overall Disability Scale | 39 |
| 8.1.12. | Pharmacoeconomics Questionnaire | 39 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | 39 |
| 8.1.15. | Vitamin A | 39 |
| 8.1.16. | Anti-Drug Antibodies | 39 |
| 9. | ASSESSMENT OF SAFETY | 40 |
| 9.1. | Safety Parameters | 40 |
| 9.1.1. | Demographic and Medical History | 40 |

| 9.1.2. | Vital Signs | 40 |
|----------|-------------------------------------------|----|
| 9.1.3. | Weight and Height | 40 |
| 9.1.4. | Physical Examination | 40 |
| 9.1.5. | Laboratory Assessments | 40 |
| 9.1.5.1. | Hematology | 41 |
| 9.1.5.2. | Blood Chemistry | 41 |
| 9.1.5.3. | Urinalysis | 41 |
| 9.1.5.4. | Pregnancy Screen. | 42 |
| 9.1.6. | Ophthalmology Examination | 42 |
| 9.2. | Adverse Events and Serious Adverse Events | 42 |
| 9.2.1. | Definition of Adverse Events | 42 |
| 9.2.1.1. | Adverse Event | 42 |
| 9.2.1.2. | Serious Adverse Event | 42 |
| 9.3. | Relationship to Study Drug | 43 |
| 9.4. | Recording Adverse Events | 43 |
| 9.5. | Reporting Adverse Events | 44 |
| 9.5.1. | Serious Adverse Event Reporting | 44 |
| 9.5.2. | Pregnancy Reporting | 46 |
| 10. | STATISTICS | 47 |
| 10.1. | Sample Size | 47 |
| 10.2. | Statistical Methodology | 47 |
| 10.2.1. | Populations to be Analyzed | 47 |
| 10.2.2. | Baseline Evaluations | 47 |
| 10.2.3. | Efficacy Analyses | 47 |
| 10.2.4. | Safety Analyses | 48 |
| 10.2.5. | Healthcare Utilization Assessments | 48 |
| 10.2.6. | Interim Analysis | 48 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 49 |
| 11.1. | Study Monitoring | 49 |
| 11.2. | Audits and Inspections | 49 |
| 11.3. | Institutional Review Board | 49 |
| 12 | OUALITY CONTROL AND OUALITY ASSURANCE | 50 |

| 13. | ETHICS | 51 |
|---------|--------------------------------------------|----|
| 13.1. | Ethics Review | |
| 13.2. | Ethical Conduct of the Study | 51 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 51 |
| 13.3. | Written Informed Consent | 51 |
| 14. | DATA HANDLING AND RECORD KEEPING | 53 |
| 14.1. | Case Report Forms | 53 |
| 14.2. | Confidentiality | 53 |
| 14.3. | Inspection of Records | 53 |
| 14.4. | Retention of Records | 54 |
| 15. | PUBLICATION POLICY | 55 |
| 16. | LIST OF REFERENCES | 56 |
| 17. | APPENDICES | 57 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| НР | heat pain |
| HRdb | heart rate response to deep breathing |

| ICF informed consent form ICH International Conference on Harmonization IEC Independent Ethics Committee IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous INP lipid nanoparticle IBMI modified body mass index INP modified body mass index IMEDRA Medical Dictionary for Regulatory Activities IMIS Modified Neuropathy Impairment Score IMIS Modified Neuropathy Impairment Score IMIS Neuropathy Impairment Score INP NIS Neuropathy Impairment Score INP NIS Neuropathy Impairment Score INS Neuropathy Impairment Score INS Neuropathy Impairment Score INS Neuropathy Impairment Score INS-W Neuropathy Impairment S | Abbreviation | Definition |
|---|---|---|
| ICH International Conference on Harmonization IEC Independent Ethics Committee IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous ILNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | IB | Investigators Brochure |
| IEC Independent Ethics Committee IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous ILNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | ICF | informed consent form |
| IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | ICH | International Conference on Harmonization |
| INN International Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous ILNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | IEC | Independent Ethics Committee |
| INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IENFD | intraepidermal nerve fiber density |
| IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score WIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | INN | International Nonproprietary Name |
| IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | INR | international normalized ratio |
| IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IRB | Institutional Review Board |
| IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IRR | infusion-related reaction |
| IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IRS | interactive response system |
| IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IUD | intrauterine device |
| LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IUS | intrauterine system |
| mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IV | intravenous |
| MedDRA Medical Dictionary for Regulatory Activities Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- NES-W | LNP | lipid nanoparticle |
| mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | mBMI | modified body mass index |
| mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | MedDRA | Medical Dictionary for Regulatory Activities |
| MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | mNIS | Modified Neuropathy Impairment Score |
| NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | mRNA | messenger RNA |
| NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | MR | magnetic resonance |
| NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NCS | nerve conduction studies |
| NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NHP | non-human primate |
| NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NIS | Neuropathy Impairment Score |
| NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NIS-W | Neuropathy Impairment Score- Weakness |
| NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NSAID | nonsteroidal anti-inflammatory drug |
| OTC over-the-counter PCS Patient Care Sites | NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| PCS Patient Care Sites | NYHA | New York Heart Association |
| | OTC | over-the-counter |
| PD pharmacodynamic | PCS | Patient Care Sites |
| | PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WHO | World Health Organization |
| WT | wild type |

### 1. INTRODUCTION

### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR.<sup>1,2</sup> The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset.<sup>3</sup> There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC).<sup>4,5,6</sup> The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States.<sup>7,8</sup> The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.<sup>9</sup>

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. <sup>10</sup> The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in

serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

### 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

### 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the circulating amyloidogenic protein could impact the clinical course of the disease. Based on

nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

### • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### • Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone mineralization. If there are no medical contraindications, and per investigator judgment and

local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

### 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

### 3. INVESTIGATIONAL PLAN

### 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 \ (\pm 3)$  days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30 \ (\pm 5)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for

which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

### 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

### 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

### 4. SELECTION AND WITHDRAWAL OF PATIENTS

### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study

6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development.<sup>14</sup> It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters,

or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2,

CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

### 5. TREATMENT OF PATIENTS

### 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

### **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

### **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

### 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

### 6. STUDY DRUG MATERIALS AND MANAGEMENT

### 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

### **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

### 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

### 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

### **6.4.2.** Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every  $21 \pm 3$  days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done according to a site-specific plan by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window ( $\pm 3$  days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of

patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - 1) If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

### 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

### 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

### 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

### 8. ASSESSMENT OF EFFICACY

### 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

## 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

#### 8.1.4. Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.
## 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

## 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

# 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

## 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

## 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

## 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

#### **8.1.12.** Pharmacoeconomics Ouestionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

## 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

## 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

#### **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.16. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

#### 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

## 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

## 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

#### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

#### 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the

Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

## 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

## **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

## 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

## 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

# 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

## 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity

- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

## 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the

completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

## 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

#### 10. STATISTICS

# **10.1.** Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

## **10.2.1.** Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### 10.2.2. Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

## 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma 5$  NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm SE$ ) values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

## 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### **10.2.5.** Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

### 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

## 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

## 13. ETHICS

## 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

#### 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes

requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

## 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the

drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

#### 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

## 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- 5 Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| Able to carry on normal activity and to work; no special care needed. | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed. | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

**Appendix 2: New York Heart Association Classification of Heart Failure** 

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

# **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

# **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NISa) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | <ul> <li>Nerve conduction studies ∑5 (18.6)<sup>a</sup></li> </ul> |
| | | <ul> <li>Sural SNAP, tibial motor n. distal latency, peroneal<br/>SNAP/motor n. conduction velocity/motor n. distal<br/>latency</li> </ul> |
| | | • Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies ∑5 (10) <sup>a</sup> |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | • Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

## **ALN-TTR02-006 Amendment 1 Summary of Changes:**

# Protocol Version 2.0 (Amendment 1), dated 08 September 2015, compared to Protocol Version 1.0 (Original Protocol), dated 06 November 2014

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Amendment 1**

The changes in this amendment have been made to the following sections as indicated below; a rationale for the changes is also provided, followed by a detailed summary of changes.

## Modification of Premedication Regimen

To date, per the ALN-TTR02-004/ALN-TTR02-006 protocol, patients in this study were to receive a premedication regimen that included 8 mg of dexamethasone or equivalent the night before and 20 mg IV dexamethasone or equivalent the day of the infusion. Some patients on this premedication regimen for an extended amount of time in the ongoing Phase 2 open-label extension (OLE) study (Study ALN-TTR02-003) have reported recurrent episodes of flushing after the infusion that the Investigator(s) reported as an infusion-related reaction (IRR) and/or related to the premedication dexamethasone. In a prior Phase 2 multi-dose study (Study ALN-TTR02-002), a less intensive premedication regimen was tested, consisting of 10 mg of dexamethasone given only on the day of infusion in 9 FAP patients, which did not lead to an increase in IRRs. Based on the prior Phase 2 experience in Study ALN-TTR02-002, the premedication regimen for the 9 patients in the OLE study (Study ALN-TTR02-003) who were experiencing post infusion flushing was reduced to include only 10 mg dexamethasone on the day of infusion. In addition, after discussion with the investigator two additional patients without flushing also received the lower dose of dexamethasone in the OLE study (Study ALN-TTR02-003). These 11 patients in the OLE study (Study ALN-TTR02-003) have been followed for a mean (range) of 6 (1-8) months on this less intensive premedication regimen and appeared to tolerate the infusions without any worsening or increased frequency of IRRs, and some reported less flushing. Based on this information, it is appropriate to change to the less intensive premedication regimen for patients in Study ALN-TT02-004/TTR02-006.

In addition, after consultation with the medical monitor, specified patients who are intolerant of 10 mg IV dexamethasone or equivalent on the day of infusion may be considered for further step-wise reduction in dexamethasone or equivalent as specified in the protocol (See Protocol Section 6.4.1). Alternatively, after consultation with the medical monitor, if the patient develops infusion related reactions on 10 mg IV or less of dexamethasone, even after slowing of the infusion, that patient will be allowed to increase the steroid premeditation dose in a step-wise manner as indicated per protocol (See Protocol Section 6.4.3).

#### Clarification of Risk Benefit Assessment

The risk benefit assessment has been updated to reflect liver function test abnormalities and risk for osteoporosis. Because patients with FAP may be at risk for osteoporosis, it has been added that, if there is no medical contraindication, and per investigator judgment and local standard of care, study

participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

#### Clarification of the Inclusion Criterion about Total Bilirubin

The inclusion criterion about total bilirubin has been updated to be consistent with the inclusion critierion about total bilirubin in Study ALN-TTR02-004. Specifically the updated criterion states that patients must have total bilirubin within normal limits, but states that a patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.

## Clarification about Exclusion Criterion about Uncontrolled Cardiac Arrhythmia and Unstable Angina

This amendment also clarified that patients with any uncontrolled cardiac arrhythmia or unstable angina are not permitted to enroll in the study (Exclusion Criterion #3). Patients with uncontrolled clinically significant cardiac arrhythmia or unstable angina were not permitted to enroll in this study in the previous version of the protocol; the change was made to remove the subjective determination of clinical significance from the criterion.

#### Clarification about the Duration of the Study

This amendment also clarified that the duration of the study was determined to allow the collection for long-term safety, tolerability, and efficacy data of patisiran.

#### **Additional Clarifications**

The following clarifications have also been made in this amendment:

- The collection of thyroid stimulating hormone (TSH) is an efficacy assessment in Section 8.
- Blood for serum vitamin A level will be collected before the administration of vitamin A supplementation (and not before patisiran administration because these assessments are performed at non-dosing visits).
- Magnetic resonance neurography is to be performed in the subset of patients who completed it in their parent study and may be performed for patients who did not complete it in their parent study.
- The same examiner should perform the mNIS+7 and NIS+7 assessments at the Week 52 visit as in the patient's parent study.
- All clinical laboratory samples will be processed by the central laboratory.
- Concomitant medications that continue from the parent study should be entered into the database.
- Added INR assessment as a safety laboratory assessment.
- Added a 12-Week visit to collect samples for safety laboratory assessments.
- Added to the Schedule of Events that inclusion and exclusion criteria are to be evaluated at the Day 0 Visit.
- Separated the End of Study Visit and the Early Withdrawal Visits on the Schedule of Events.
- Clarified study drug preparation.

• Clarified the follow-up for SAEs

A detailed summary of changes is provided in Table 1. Corrections to typographical errors, punctuation, grammar, abbreviations, and formatting are not detailed.

# **Table 1:** Amendment 1 Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in this amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose:

To explore tolerability of patients with lower dexamethasone in premedication regimen

Primary change (1 of 3):

Section 6.4.1 Premedication

Formerly read:

Prior to dosing, patients will receive 2 sets of premedications in order to reduce the risk of experiencing an IRR.

For all patients, the first set of premedications will be administered on the evening before patisiran administration as follows:

- Oral dexamethasone (8 mg) or equivalent
- Oral paracetamol/ acetaminophen (500 mg) or equivalent
- Oral H2 blocker (ranitidine 150 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Oral H1 blocker, 10 mg cetirizine (hydroxyzine 25 mg, fexofenadine, or equivalent may be substituted if patient does not tolerate cetirizine)

If the evening premedications (first set) are missed, they should be administered a minimum of 6 hours before the second set (see below) of premedications on the day of dosing (ie, at least 7 hours before patisiran dosing).

Prior to each dose of patisiran, patients will also receive the following premedications (ie, second set) at least 60 minutes before the infusion:

- Intravenous dexamethasone (20 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Modifications to the premedication regimen may be allowed due to lack of tolerability of one or more of the premedications by the patient (eg, lowering of the corticosteroid dose if a patient develops uncontrolled hyperglycemia or altered mental status). Such modifications may be allowed for that patient only after consultation with the Medical Monitor. If the premedication regimen was already modified for this reason on the parent study, the modification for that particular patient will be carried over into this study.

Now reads:

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps must be followed:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of intravenous dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

Primary change (2 of 3):

Section 6.4.2 Study Drug Administration

Formerly read:

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

The infusion time may be extended up to 3 hours in the event of a mild or moderate IRR; patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor (see Section 6.4.3). If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor. For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

Now reads:

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

Primary change (3 of 3):

Section 6.4.3 Suggested Guidelines for Management of Infusion-Related Reactions

#### **Added Text:**

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.
- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are recommended:
  - 1) If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

Section(s) also containing this change:

- Synopsis
- Section 3.1 Overall Design

Purpose:

Provide updated risk benefit language

Primary change:

Section 1.4 Risk-Benefit Assessment

Formerly read:

#### 1.4 Risk-Benefit Assessment

Please see the IB for an expanded risk/benefit assessment.

#### 1.4.1 Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran or placebo. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### 1.4.2 Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take continue taking daily supplement containing the recommended daily allowance of vitamin A.

#### **Now Reads:**

#### 1.4 Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed.<sup>40</sup> This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP.<sup>41</sup> Provided there is adequate

Now Reads: Section(s) also

containing this change:

vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>42</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

3. Has uncontrolled cardiac arrhythmia or unstable angina

Synopsis

| Purpose | Clarify inclusion criterion about total bilirubin level to align with Study TTR02-004 |
|---|---|
| Primary Change | Section 4.1 Patient Inclusion Criteria |
| Formerly Read: | 4. Have a total bilirubin ≤1.5 × ULN, unless greater elevation above normal limits is due to Gilbert's syndrome |
| Now Reads: | 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges. |
| Section(s) also containing this change: | • Synopsis |
| Purpose | Clarification about exclusion criterion about uncontrolled cardiac arrhythmia and unstable angina |
| Primary change: | Section 4.2 Patient Exclusion Criteria |
| Formerly Read: | 3. Has uncontrolled elinically significant cardiac arrhythmia or unstable angina |
Purpose:

Clarified that the duration of the study was determined to allow the collection for long-term safety, tolerability, and efficacy data of

patisiran

Primary change:

Section 1.3

Formerly Read:

This study will allow patients to receive treatment with patisiran until it becomes commercially available in their region, or until the study is otherwise terminated by the Sponsor.

**Now Reads:** 

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

Section(s) also containing this change:

Synopsis

• Section 3.1 Overall Study Design

Purpose:

Clarified that the collection of thyroid stimulating hormone (TSH) is an efficacy assessment

Primary change:

Deleted from Section 9.1.5.2 Blood Chemistry; Added to Section 8.1.15 Thyroid Stimulating Hormone

Formerly Read:

9.1.5.2 Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

Aspartate transaminase (AST)

• Alanine transaminase (ALT)

Sodium

Potassium

Blood urea nitrogen (BUN)

Creatinine

Thyroid stimulating hormone

**Now Reads:** 

8.1.15 Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

Section(s) also containing this change:

Synopsis

- Alkaline phosphatase
- Bilirubin (total and direct)

Glucose

Phosphate

Albumin

Calcium

| Purpose: | Clarification that blood for serum vitamin $A$ level will be collected before the administration of vitamin $A$ supplementation (and not before patisiran administration because these assessments are performed at non-dosing visits). |
|---|---|
| Primary change: | Section 8.1.16 Vitamin A |
| Now Reads: | Blood for serum vitamin A levels will be collected at scheduled visits before the administration of patisiran and vitamin A supplementation. |
| Purpose: | Clarification that magnetic resonance neurography is to be performed only in the subset of patients who completed it in their parent study and may be performed for patients who did not complete it in their parent study |
| Primary change: | Section 8.1.4 Magnetic Resonance Neurography (Subset of Patients) |
| Added Text: | Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. <sup>1</sup> This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in their parent study. A central reader will be used for MR neurography. |
| Section(s) also containing this change: | <ul> <li>Synopsis</li> <li>Table 1 Schedule of Assessments, footnote u</li> </ul> |

Purpose:

Clarification that the same examiner should perform the mNIS+7 and NIS+7 assessments at the Week 52 visit as in the patient's parent study

Primary change:

Section 8.1.1.1

Formerly read:

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Each site will make every effort to have these assessments performed by the same study personnel, who will be different from the Investigator and other personnel managing the patient. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment.

Now reads:

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

Section(s) also containing this change:

Table 1 Schedule of Events, footnotes l, m, and n

Purpose:

Clarification that all clinical laboratory samples will be processed by the central laboratory.

Primary change:

Section 9.1.5 Laboratory Assessments

Formerly read:

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. Samples collected at the Day 0, 26 week, and 52 week visits will be sent to a central laboratory for analysis. Samples collected at the annual visits and End of Study or Early Withdrawal visits will be analyzed at the local laboratory. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

Now reads:

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a

Laboratory Manual.

Section(s) also

Table 1 Schedule of Assessment, footnotes i and j (deleted)

containing this change:

Purpose: Concomitant medications that continue from the parent study should be entered into the database.

Primary change: Section 5.2 Concomitant Medications

Now reads: Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all

> concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from

the parent study will be entered into the database.

Section(s) also Table 1 Schedule of Assessments, footnote b containing this change:

Added INR assessment as a safety laboratory assessment. Purpose:

Primary change: Section 9.1.5.4 Coagulation (new section)

9.1.5.4 Coagulation Now reads:

A sample for INR assessment will be collected.

Section(s) also containing this change: • Table 1 Schedule of Events

Purpose: Added a 12-Week visit to collect samples for safety laboratory assessments

Primary change: Table 1 Schedule of Events

**Description of** Change:

A 12-Week visit column was added to the Schedule of Events to denote the collection of samples for safety laboratory assessments at

Week 12.

Section(s) also

**Synopsis** 

containing this change:

Section 3.1 Overall Study Design

Clarified on the Schedule of Events that inclusion and exclusion criteria are to be evaluated at the Day 0 Visit Purpose:

Primary change: Table 1 Schedule of Events

**Description of** Change:

A row was added to the Schedule of Events to denote that inclusion and exclusion criteria must be reviewed on the Day 0 visit.

| Purpose: | Separated the End of Study Visit and the Early Withdrawal Visits on the Schedule of Events |
|---|---|
| Primary change: Table 1 Schedule of Events | |
| <b>Description of</b> Separate columns were added for the End of Study and Early Withdrawal Visits. <b>Change:</b> | |
| Purpose: | Clarification about study drug preparation |
| Primary change: | Section 6.3 Study Drug Preparation |
| Now reads: | Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag. |
| Purpose: | Clarification of follow-up time for SAEs |
| Primary change: | Section 9.5 Reporting Adverse Events |
| Formerly read: | For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. Serious AEs will be followed through 28 days from the last dose of patisiran, or until satisfactory resolution, or until the SAE is considered by the Investigator to be chronic or the patient is stable, whichever occurs first. |
| Now reads: | For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whicheve occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. |

Purpose: Correct typographical errors, punctuation, grammar, and formatting

These changes are not listed individually.

# PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN

Final Protocol:

Version 1.0, 06 November 2014

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

Sponsor Contact:



The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

Date

# **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and maintain the confidentiality of all information protocol. | l agree to conduct the study as outlined. I agree received or developed in connection with this | e to |
|---|---|---|
| Printed Name of Investigator | | |
| Signature of Investigator | | |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

#### Name of Investigational Product:

Patisiran

#### Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

#### Methodology:

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every  $21 \text{ (\pm 3)}$  days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm$ 5) days. Patients will also have visits at the clinical site at approximately 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### **Number of patients (planned):**

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

#### Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin  $\leq$ 1.5 × ULN, unless greater elevation above normal limits is due to Gilbert's syndrome
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled clinically significant cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive 2 sets of premedications as described below, unless changes were approved by the Medical Monitor.

On the evening before patisiran administration (or at least 6 hours before administration of the second set of premedications on the day of dosing), patients will receive the following:

- Oral dexamethasone (8 mg) or equivalent
- Oral paracetamol/ acetaminophen (500 mg) or equivalent
- Oral H2 blocker (ranitidine 150 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Oral H1 blocker, 10 mg cetirizine (hydroxyzine 25 mg, fexofenadine, or equivalent may be substituted if patient does not tolerate cetirizine)

Patients will also receive the following premedications (ie, second set) at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (20 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

It is anticipated that a patient on this study will receive treatment with open-label patisiran until the patient is able to obtain commercially available patisiran in their respective country. The study will be completed when all patients are receiving commercially available patisiran. The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor. The Sponsor also reserves the right to discontinue the study for clinical or administrative reasons at any time.

#### Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

#### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (OOL-DN) and the EuroOOL (EO-5D) questionnaires

- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography (only for patients having this assessment in the parent study)
- Cardiac structure and function through echocardiograms and serum levels of terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I
- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 26 Week Visit | 52 Week Visit | Annual Visit | End of Study / Early<br>Withdrawal Visit |
|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±6 Weeks | 4 (+1) Weeks from<br>Last Dose |
| Procedure | | | | | |
| Informed Consent | X | | | | |
| Medical History | $X^b$ | | | | |
| Demographics | $X^{c}$ | | | | |
| Physical Examination | $X^d$ | | X | X | Xº |
| Weight | X<br>Prior to Each Dose | | | | Xº |
| mBMI <sup>e</sup> | $X^d$ | | X | X | X° |
| Height | $X^{c}$ | | | | |
| FAP Stage and PND Score | $X^d$ | | X | X | Xº |
| Karnofsky Performance Status | X | | | | |
| NYHA Classification | X | | X | | $[X]^f$ |
| Vital Signs <sup>g</sup> | | X<br>Prior to E | | | |
| Safety Laboratory Assessments <sup>h</sup> | $X^{d,i}$ | Xi | Xi | $X^{j}$ | X <sup>j</sup> |
| Pregnancy Test (urine) | $X^k$ | X | X | X | X |
| TTR Protein (ELISA) | X | X | X | X | X |
| TSH and Vitamin A | | | X | X | X° |
| mNIS+7 <sup>1</sup> | $X^d$ | | X | | $[X]^f$ |
| NIS+7 <sup>m</sup> | $X^d$ | | X | | $[X]^f$ |
| NIS only | | | | X <sup>n</sup> | $X^{n,p}$ |
| Grip Strength Test <sup>q</sup> | $X^d$ | | X | | $[X]^f$ |

| | Day 0 Visit | 26 Week Visit | 52 Week Visit | Annual Visit | End of Study / Early<br>Withdrawal Visit |
|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±6 Weeks | 4 (+1) Weeks from<br>Last Dose |
| Procedure | | | | | |
| 10-Meter Walk Test <sup>r</sup> | $X^d$ | | X | | $[X]^f$ |
| Ophthalmology Examination <sup>s</sup> | $X^d$ | | X | X | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | X | X | X° |
| MR Neurography <sup>u</sup> | | | X | X | X° |
| Pharmacoeconomics<br>Questionnaire | X | | X | X | X° |
| Norfolk QOL-DN <sup>v</sup> | $X^d$ | | X | X | X° |
| COMPASS 31 Questionnaire | $X^d$ | | X | | $[X]^f$ |
| R-ODS Disability | $X^d$ | | X | | $[X]^{f}$ |
| EQ-5D QOL | $X^d$ | | X | X | X° |
| Echocardiogram | $X^{d,w}$ | | X | | $[X]^f$ |
| Troponin I and NT-proBNP | $X^d$ | | X | | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>x</sup> | | X | X | X | X |
| Premedication / Patisiran<br>Administration | X <sup>y</sup> | | | | |
| Phone Contact | X <sup>z</sup> | | | | |
| Adverse Events | X<br>Continuous Monitoring | | | | |
| Concomitant Medications | X<br>Continuous Monitoring | | | | |

156

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- <sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF).
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- d Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- <sup>e</sup> mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f Assessment/procedure required only if patient withdraws before the 52-week visit.
- <sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- <sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific safety laboratory assessments.
- <sup>1</sup> Analysis of blood samples obtained at Day 0, 26 weeks, and 52 weeks will be performed at a central laboratory. Urinalysis is not required at Day 0.
- Analysis of blood samples obtained at the Annual visits and the End of Study or Early Withdrawal visit will be performed at the local laboratory.
- <sup>k</sup> Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.
- The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- <sup>p</sup> Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.

Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

ALN-TTR02-006

Version 1.0

- <sup>u</sup> Required only for patients who had MR neurography in the parent study.
- Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- <sup>w</sup> Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- x Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study within the 21 (±3) days timeframe. Doses may be administered at the clinical site or at home by a healthcare professional trained in the protocol.
- Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use.

# **TABLE OF CONTENTS**

| SYNOP | SIS | 3 |
|---|---|---|
| TABLE | OF CONTENTS | 11 |
| LIST OF | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 1.4.1. | Infusion-Related Reactions. | 19 |
| 1.4.2. | Vitamin A Lowering | 20 |
| 2. | STUDY OBJECTIVES | 21 |
| 3. | INVESTIGATIONAL PLAN | 22 |
| 3.1. | Overall Study Design | 22 |
| 3.2. | Number of Patients | 23 |
| 3.3. | Treatment Assignment | 23 |
| 3.4. | Criteria for Study Termination | 23 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 24 |
| 4.1. | Patient Inclusion Criteria | 24 |
| 4.2. | Patient Exclusion Criteria | 24 |
| 4.3. | Patient Withdrawal Criteria | 25 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 25 |
| 5. | TREATMENT OF PATIENTS | 28 |
| 5.1. | Description of Study Drug | 28 |
| 5.2. | Concomitant Medications | 28 |
| 5.3. | Treatment Compliance | 28 |
| 5.4. | Randomization and Blinding | 29 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 30 |
| 6.1. | Study Drug Packaging and Labeling | 30 |
| 6.2. | Study Drug Storage | 30 |

Version 1.0

| 6.3. | Study Drug Preparation | 30 |
|---|---|---|
| 6.4. | Administration | 31 |
| 6.4.1. | Premedication | 31 |
| 6.4.2. | Study Drug Administration | 31 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 32 |
| 6.5. | Study Drug Accountability | 32 |
| 6.6. | Study Drug Handling and Disposal | 33 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 34 |
| 8. | ASSESSMENT OF EFFICACY | 35 |
| 8.1. | Efficacy Parameters | 35 |
| 8.1.1. | Neurological Testing | 35 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 35 |
| 8.1.1.2. | Neurological Impairment Score | 36 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 36 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | 36 |
| 8.1.4. | Magnetic Resonance Neurography | 36 |
| 8.1.5. | Modified Body Mass Index | 37 |
| 8.1.6. | Timed 10-meter Walk Test | 37 |
| 8.1.7. | Grip Strength Test | 37 |
| 8.1.8. | Composite Autonomic Symptom Score | 37 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 37 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 37 |
| 8.1.11. | Rasch-built Overall Disability Scale | 38 |
| 8.1.12. | Pharmacoeconomics Questionnaire | 38 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 38 |
| 8.1.14. | Transthyretin | 38 |
| 8.1.15. | Vitamin A | 38 |
| 8.1.16. | Anti-Drug Antibodies | 38 |
| 9. | ASSESSMENT OF SAFETY | 39 |
| 9.1. | Safety Parameters | 39 |
| 9.1.1. | Demographic and Medical History | 39 |

| 9.1.2. | Vital Signs | 39 |
|----------|-------------------------------------------|----|
| 9.1.3. | Weight and Height | 39 |
| 9.1.4. | Physical Examination | 39 |
| 9.1.5. | Laboratory Assessments | 39 |
| 9.1.5.1. | Hematology | 40 |
| 9.1.5.2. | Blood Chemistry | 40 |
| 9.1.5.3. | Urinalysis | 40 |
| 9.1.5.4. | Pregnancy Screen. | 41 |
| 9.1.6. | Ophthalmology Examination | 41 |
| 9.2. | Adverse Events and Serious Adverse Events | 41 |
| 9.2.1. | Definition of Adverse Events | 41 |
| 9.2.1.1. | Adverse Event | 41 |
| 9.2.1.2. | Serious Adverse Event | 41 |
| 9.3. | Relationship to Study Drug | 42 |
| 9.4. | Recording Adverse Events | 42 |
| 9.5. | Reporting Adverse Events | 43 |
| 9.5.1. | Serious Adverse Event Reporting | 43 |
| 9.5.2. | Pregnancy Reporting | 44 |
| 10. | STATISTICS | 46 |
| 10.1. | Sample Size | 46 |
| 10.2. | Statistical Methodology | 46 |
| 10.2.1. | Populations to be Analyzed | 46 |
| 10.2.2. | Baseline Evaluations | 46 |
| 10.2.3. | Efficacy Analyses | 46 |
| 10.2.4. | Safety Analyses | 47 |
| 10.2.5. | Healthcare Utilization Assessments | 47 |
| 10.2.6. | Interim Analysis | 47 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 48 |
| 11.1. | Study Monitoring | 48 |
| 11.2. | Audits and Inspections | 48 |
| 11.3. | Institutional Review Board | 48 |
| 12. | OUALITY CONTROL AND OUALITY ASSURANCE | 49 |

| 13. | ETHICS | 50 |
|---------|--------------------------------------------|----|
| 13.1. | Ethics Review | 50 |
| 13.2. | Ethical Conduct of the Study | 50 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 50 |
| 13.3. | Written Informed Consent | 50 |
| 14. | DATA HANDLING AND RECORD KEEPING | 52 |
| 14.1. | Case Report Forms | 52 |
| 14.2. | Confidentiality | 52 |
| 14.3. | Inspection of Records | 53 |
| 14.4. | Retention of Records | 53 |
| 15. | PUBLICATION POLICY | 54 |
| 16. | LIST OF REFERENCES | 55 |
| 17. | APPENDICES | 56 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| ТР | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WHO | World Health Organization |
| WT | wild type |

#### 1. INTRODUCTION

#### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). A.5.6 The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. <sup>10</sup> The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

#### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. This study will allow patients to receive treatment with patisiran until it becomes commercially available in their region, or until the study is otherwise terminated by the Sponsor.

#### 1.4. Risk-Benefit Assessment

Please see the IB for an expanded risk/benefit assessment.

#### 1.4.1. Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran or

placebo. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### 1.4.2. Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take continue taking daily supplement containing the recommended daily allowance of vitamin A.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

#### 3. INVESTIGATIONAL PLAN

### 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

It is anticipated that a patient on this study will receive treatment with open-label patisiran until the patient is otherwise able to obtain commercially available patisiran in their respective country. The study will be completed when all patients are receiving commercially available patisiran.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive 2 sets of premedications before dosing with patisiran in order to reduce the risk of experiencing an IRR. The first set of premedications will be administered the evening before patisiran administration (or at least 6 hours before the second set of premedications on the day of dosing). The second set of premedications will be administered at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21~(\pm 3)$  days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30~(\pm 5)$  days. Patients will also have visits at the clinical site at approximately 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to

the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

### 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 ( $\pm$ 3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

#### 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin ≤1.5 × ULN, unless greater elevation above normal limits is due to Gilbert's syndrome
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

#### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled clinically significant cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study

6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters,

or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2,

CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

#### 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

#### **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for

scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

# 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

#### 6. STUDY DRUG MATERIALS AND MANAGEMENT

# 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran and placebo will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# **6.3.** Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm$  3 days). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions.

#### 6.4. Administration

#### 6.4.1. Premedication

Prior to dosing, patients will receive 2 sets of premedications in order to reduce the risk of experiencing an IRR.

For all patients, the first set of premedications will be administered on the evening before patisiran administration as follows:

- Oral dexamethasone (8 mg) or equivalent
- Oral paracetamol/ acetaminophen (500 mg) or equivalent
- Oral H2 blocker (ranitidine 150 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Oral H1 blocker, 10 mg cetirizine (hydroxyzine 25 mg, fexofenadine, or equivalent may be substituted if patient does not tolerate cetirizine)

If the evening premedications (first set) are missed, they should be administered a minimum of 6 hours before the second set (see below) of premedications on the day of dosing (ie, at least 7 hours before patisiran dosing).

Prior to each dose of patisiran, patients will also receive the following premedications (ie, second set) at least 60 minutes before the infusion:

- Intravenous dexamethasone (20 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Modifications to the premedication regimen may be allowed due to lack of tolerability of one or more of the premedications by the patient (eg, lowering of the corticosteroid dose if a patient develops uncontrolled hyperglycemia or altered mental status). Such modifications may be allowed for that patient only after consultation with the Medical Monitor. If the premedication regimen was already modified for this reason on the parent study, the modification for that particular patient will be carried over into this study.

#### 6.4.2. Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every 21  $(\pm 3)$  days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where
applicable country and local regulations allow. Home administration of patisiran will be done according to a site-specific plan by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

The infusion time may be extended up to 3 hours in the event of a mild or moderate IRR; patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor (see Section 6.4.3). If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor. For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window ( $\pm 3$  days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

#### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.

Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion. Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much

patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

# 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

# 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

#### 8. ASSESSMENT OF EFFICACY

# 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

#### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Each site will make every effort to have these assessments performed by the same study personnel, who will be different from the Investigator and other personnel managing the patient. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment.

#### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

# 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

#### 8.1.4. Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders.<sup>15</sup> This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for those patients who had MR neurography in the parent study. A central reader will be used for MR neurography.

#### 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

#### 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

# 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

#### 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

#### 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

#### 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

#### 8.1.12. Pharmacoeconomics Questionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

# 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

#### 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

#### 8.1.15. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of patisiran and vitamin A supplementation.

#### 8.1.16. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

#### 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

# 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

#### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

## 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. Samples collected at the Day 0, 26-week, and 52-week visits will be sent to a central laboratory for analysis. Samples collected at the annual visits and End of Study or Early Withdrawal visits will be analyzed at the local laboratory. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

#### 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

#### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine
- Thyroid stimulating hormone (TSH)

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

#### **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

#### 9.1.5.4. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

#### 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

# 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to

prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day

should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. Serious AEs will be followed through 28 days from the last dose of patisiran, or until satisfactory resolution, or until the SAE is considered by the Investigator to be chronic or the patient is stable, whichever occurs first.

#### 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC

system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

#### 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the

pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

#### 10. STATISTICS

# 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

#### **10.2.1.** Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### **10.2.2.** Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

# 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean  $(\pm SE)$  values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

#### 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

#### 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

#### 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

#### 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

#### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

# 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

#### 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

#### 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

#### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- 3 Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- 5 Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, HK, et al. Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou V, et al. Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci USA, 1993. 90: p. 2375-2379.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

**Appendix 2: New York Heart Association Classification of Heart Failure** 

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

# **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

# **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NISa) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (18.6)^a$ |
| | | <ul> <li>Sural SNAP, tibial motor n. distal latency, peroneal<br/>SNAP/motor n. conduction velocity/motor n. distal<br/>latency</li> </ul> |
| | | • Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (10)^a$ |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

# PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN


Version 3.1-Argentina (Incorporating Amendment

2)

Protocol Date

20 January 2017

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

Sponsor Contact:



Date

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

# **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to |
|---|
| maintain the confidentiality of all information received or developed in connection with this |
| protocol. |

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| <br>Date |

# **Version History:**

|---|---|---|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 – Global | 08 September 2015 | Incorporating Global Amendment 1 |
| 3.1 – Argentina | 20 January 2017 | Incorporating Global Amendment 2 and |
| | | Argentina-specific clarification letter dated |
| | | 03 November 2016 |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

#### **Name of Investigational Product:**

Patisiran

#### Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

# **Methodology:**

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV)

once every 21 (±3) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0.

Eligibility for this study will be confirmed before administration of the first dose on Day 0. After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

#### Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤2 x ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

#### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Cardiac structure and function through echocardiograms and serum levels of terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid stimulating hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; ophthalmology examinations; and assessment of suicidal ideation and behavior.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.
Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Windo | ≤45 Days from<br>W Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | $X^d$ | | | X | X | X° | X° |
| Weight | | Prior | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | X <sup>d</sup> | | | X | X | Xº | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | X <sup>d</sup> | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | | $[X]^f$ |
| Vital Signs <sup>g</sup> | X<br>Prior to Each Dose | | | | | | |
| Safety Laboratory Assessments <sup>h</sup> | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | | 1 | I | X <sup>i</sup> | I | | l |
| C-SSRS Questionnaire | | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TTR Protein (ELISA) | $X^{d}$ | | X | X | X | X | X |
| TSH and Vitamin A | | | | X | X | X° | X° |
| mNIS+7 <sup>j</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS+7 <sup>k</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS only | | | | | $X^{l}$ | X <sup>m</sup> | X <sup>m</sup> |
| Grip Strength Test <sup>n</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| 10-Meter Walk Test <sup>p</sup> | X <sup>d</sup> | | | X | | | $[X]^f$ |
| Ophthalmology Examination <sup>q</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>r</sup> | | | | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | Xº | Xº |
| Norfolk QOL-DN <sup>s</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | X° | X° |
| Echocardiogram | $X^{d,t}$ | | | X | | | $[X]^f$ |
| Troponin I and NT-proBNP | X <sup>d</sup> | | | X | | | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>u</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration <sup>v</sup> | X | | X | | | | |

217

| | | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|---|
| | Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | | |
| Adverse Events | | X <sup>b</sup> Continuous Monitoring | | | | | | |
| Concomitant Medications | | X <sup>b</sup> Continuous Monitoring | | | | | | |

#### Table 1 Footnotes:

Abbreviations: C-SSRS = Columbia-Suicide Severity Rating Scale; COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- a. Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- b. Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- c. Assessment does not need to be repeated. Information will be obtained from parent study.
- d. Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- e. mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f. Assessment/procedure required only if patient withdraws before the 52-week visit.
- g. Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- h. Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- i. Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose. Pregnancy testing will be done on a monthly basis during study duration.
- j. The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days

- after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- k. The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- 1. One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- m. Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- n. Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- o. Assessment does not need to be repeated if done within the previous 26 weeks.
- p. The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- q. Examination will include visual acuity, visual fields, and slit-lamp evaluation. An electroretinogram may also be performed, as described in Section 9.1.6
- r. Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- s. Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- t. Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- u. Serum samples for anti-drug antibodies will be collected as specified.
- v. Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study in the 21 (±3) day timeframe.

# **TABLE OF CONTENTS**

#### SYNOPSIS3

| <b>TABLE</b> | OF CONTENTS | 11 |
|---|---|---|
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |

| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | 37 |
| 8.1.4. | Modified Body Mass Index | 37 |
| 8.1.5. | Timed 10-meter Walk Test | 37 |
| 8.1.6. | Grip Strength Test | 38 |
| 8.1.7. | Composite Autonomic Symptom Score | 38 |
| 8.1.8. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.9. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.10. | Rasch-built Overall Disability Scale | 38 |
| 8.1.11. | Pharmacoeconomics Questionnaire | 38 |
| 8.1.12. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.13. | Transthyretin | 39 |
| 8.1.14. | Thyroid-Stimulating Hormone | 39 |
| 8.1.15. | Vitamin A | 39 |
| 8.1.16. | Anti-Drug Antibodies | 39 |
| 9. | ASSESSMENT OF SAFETY | 40 |
| 9.1. | Safety Parameters | 40 |
| 9.1.1. | Demographic and Medical History | 40 |
| 9.1.2. | Vital Signs | |
| 9.1.3. | Weight and Height | 40 |

| 9.1.4. | Physical Examination | 40 |
|----------|-------------------------------------------|----|
| 9.1.5. | Laboratory Assessments | 40 |
| 9.1.5.1. | Hematology | 41 |
| 9.1.5.2. | Blood Chemistry | 41 |
| 9.1.5.3. | Urinalysis | 41 |
| 9.1.5.4. | Coagulation | 42 |
| 9.1.5.5. | Pregnancy Screen | 42 |
| 9.1.6. | Ophthalmology Examination | 42 |
| 9.1.7. | Columbia-Suicide Severity Rating Scale | 42 |
| 9.2. | Adverse Events and Serious Adverse Events | 42 |
| 9.2.1. | Definition of Adverse Events | 42 |
| 9.2.1.1. | Adverse Event | 42 |
| 9.2.1.2. | Serious Adverse Event | 42 |
| 9.3. | Relationship to Study Drug | 43 |
| 9.4. | Recording Adverse Events | 43 |
| 9.5. | Reporting Adverse Events | 44 |
| 9.5.1. | Serious Adverse Event Reporting | 44 |
| 9.5.2. | Pregnancy Reporting | 46 |
| 10. | STATISTICS | 47 |
| 10.1. | Sample Size | 47 |
| 10.2. | Statistical Methodology | 47 |
| 10.2.1. | Populations to be Analyzed | 47 |
| 10.2.2. | Baseline Evaluations | 47 |
| 10.2.3. | Efficacy Analyses | 47 |
| 10.2.4. | Safety Analyses | 48 |
| 10.2.5. | Healthcare Utilization Assessments | 48 |
| 10.2.6. | Interim Analysis | 48 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 49 |
| 11.1. | Study Monitoring | 49 |
| 11.2. | Audits and Inspections | 49 |
| 11.3. | Institutional Review Board | 49 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 5( |

| 13. | ETHICS | 51 |
|---------|--------------------------------------------|----|
| 13.1. | Ethics Review | 51 |
| 13.2. | Ethical Conduct of the Study | 51 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 51 |
| 13.3. | Written Informed Consent | 51 |
| 14. | DATA HANDLING AND RECORD KEEPING | 53 |
| 14.1. | Case Report Forms | 53 |
| 14.2. | Confidentiality | 53 |
| 14.3. | Inspection of Records | 54 |
| 14.4. | Retention of Records | 54 |
| 15. | PUBLICATION POLICY | 55 |
| 16. | LIST OF REFERENCES | 56 |
| 17. | APPENDICES | 57 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RBP | retinol binding protein |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| ТР | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WT | wild type |

#### 1. INTRODUCTION

#### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). A,5,6 The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

#### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran Investigator's Brochure.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### • Vitamin A Lowering

The suppression of serum levels of TTR and retinol binding protein (RBP) is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone

mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the Investigator's Brochure.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

#### 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 (±3) days Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

# 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

#### 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\le 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\le 2.0$  (patients on anticoagulant therapy with an INR of  $\le 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

#### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study

conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9,

CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

#### 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

#### **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

# 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

#### 6. STUDY DRUG MATERIALS AND MANAGEMENT

# 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

#### 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

#### 6.4.2. Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every 21 ( $\pm$ 3) days.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

#### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.
- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.

- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

# 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

# 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

#### 8. ASSESSMENT OF EFFICACY

### 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place at the CAS. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

#### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

#### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

#### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

#### 8.1.4. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

#### 8.1.5. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

#### 8.1.6. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

#### 8.1.7. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

#### 8.1.8. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.9. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

#### 8.1.10. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

#### 8.1.11. Pharmacoeconomics Questionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

#### 8.1.12. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

#### 8.1.13. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

#### **8.1.14.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.15. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

#### 8.1.16. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1.

#### 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

#### 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

#### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

#### 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

#### 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

#### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

### **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

#### 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

#### 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

# 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

#### 9.1.7. Columbia-Suicide Severity Rating Scale

The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess each patient's mental status as it relates to suicidal ideation and behavior.

#### 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:
- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs.

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

## 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.

```
Medpace SAE hotline – USA:
Telephone: PPD ext. PPD or PPD ext. PPD
Facsimile: PPD or PPD

Medpace SAE hotline – Europe:
Telephone: PPD
Facsimile: PPD
Facsimile: PPD
```

Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that

transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

## 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

## 10. STATISTICS

# 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

# 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### **10.2.2.** Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

## 10.2.3. Efficacy Analyses

Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory

and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

## 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

A listing of healthcare utilization data will be presented.

## 10.2.6. Interim Analysis

Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator and the site will permit study-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

## 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

## 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Medical Association Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

# 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

## 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

## 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

## 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| inceded. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| assistance needed. | 50 | Requires considerable assistance and frequent medical care. |
| | 40 | Disabled; requires special care and assistance. |
| Unable to care for self; requires | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| equivalent of institutional or hospital care; disease may be progressing rapidly. | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

# **Appendix 2: New York Heart Association Classification of Heart Failure**

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

# **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | <ul> <li>Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS<sup>a</sup>)</li> <li>Weakness (192)</li> <li>Sensation (32)</li> <li>Reflexes (20)</li> <li>Nerve conduction studies ∑5 (18.6)<sup>a</sup></li> <li>Sural SNAP, tibial motor n. distal latency, peroneal CMAP/motor n. conduction velocity/motor n. distal latency</li> <li>Vibration detection threshold (3.7)</li> <li>Heart rate response to deep breathing (3.7)</li> </ul> |
| Modified NIS+7 | 304 | <ul> <li>Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS<sup>a</sup>)</li> <li>Weakness (192)</li> <li>Reflexes (20)</li> <li>Nerve conduction studies ∑5 (10)<sup>a</sup></li> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP, peroneal CMAP</li> <li>Quantitative sensory testing: QST-BSA<sub>TP+HP5</sub> (80)</li> <li>Postural blood pressure (2)</li> </ul> |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

## **ALN-TTR02-006 Protocol Version 3.1 Argentina**

Summary of Changes (dated 20 January 2017) compared to Protocol Version 2 (dated 08 September 2015)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

## **Rationale for Protocol Amendment**

The primary purpose of this amendment is to add the Columbia-Suicide Severity Rating Scale (C-SSRS) to the study assessments, which was inadvertently left out of previous versions of the protocol. The inclusion of the C-SSRS addresses a regulatory requirement to prospectively assess suicidality in clinical trials involving all drugs for neurological indications. Overall, this amendment includes the following changes:

- The Columbia-Suicide Severity Rating Scale has been added as an assessment of suicidal ideation and behavior.
- Electroretinograms are now recommended to be performed in the case of suspected retinal disease.
- The premedication regimen has been updated to align with commercially available doses.
- Reference to home infusions and to magnetic resonance neurography have been removed as they will not be performed in Argentina.
- The protocol was updated to include changes specified in the clarification letter dated 03 November 2016, clarifying the timing of pregnancy testing.

A detailed summary of these changes, in addition to changes made for clarity, is provided in Table 1. Corrections to abbreviations, typographical errors and formatting are not detailed.

## Table 1: Protocol Version 3.1 Argentina Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by bold font.

Purpose: Added Columbia-Suicide Severity Rating Scale to the study assessments

The primary change occurs in Table 1 Schedule of Assessments

Added text: Added row to Schedule of Assessments indicating that the Columbia-Suicide Severity Rating Scale is to be

collected at 26 weeks and 52 weeks after baseline and annually thereafter, as well as at the End of Study and Early

Withdrawal visits.

Section(s) also containing this change or similar changes:

• Synopsis, Criteria for Evaluation, Safety

• Section 9.1.7 Columbia-Suicide Severity Rating Scale (section added)

Purpose: Added clarity on timing of pregnancy testing, per clarification letter dated 03 November 2016.

The primary change occurs in Table 1 Schedule of Assessments, footnote i

Added text: X. Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the

first dose. Pregnancy testing will be done on a monthly basis during study duration.

Section(s) also containing this change or similar changes:

• Table 1 Schedule of Assessments, Pregnancy Test row

Purpose: To remove reference to home infusions as this will not be performed in Argentina.

The primary change occurs in Section 3.1 Overall Study Design

Deleted text: After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 (±3)

days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 (±5) days. Patients will also have visits at the clinical site at

approximately 12, 26 and 52 weeks, and yearly thereafter.

Section(s) also containing this change or similar changes:

- Synopsis methodology
- Table 1 Schedule of Assessments, Phone Contact row (removed)
- Table 1 Schedule of Assessments, Footnote w and Footnote x
- Section 5.3 Treatment Compliance
- Section 6.4.2 Study Drug Administration

Purpose: To update premedication regimen so that it aligns with commercially available doses.

The primary change occurs in Section 6.4.1 Premedication

Now reads: Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site).

Hydroxyzine or fexofenadine-25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg

PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Section(s) also containing this change or similar changes:

• Synopsis, Investigational product, dosage and mode of administration

Purpose: To remove reference to magnetic resonance neurography as this will not be performed in Argentina.

The primary change occurs in Section 8.1.4 Magnetic Resonance Neurography (removed section)

Deleted Section:

## 8.1.4Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for evaluation, Efficacy
- Table 1 Schedule of Assessments, MR neurography row (deleted)
- Table 1 Schedule of Assessments, footnote u (deleted)
- Section 8.1 Efficacy parameters

Purpose: Added recommendation to collect an electroretinogram in the case of suspected retinal injury

The primary change occurs in Section 9.1.6 Ophthalmology Examination

Added text:

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments, footnote q

Purpose: Updated description of statistical analysis to align with currently planned analytic approach.

The primary change occurs in Section 10.2.3 Efficacy Analyses

Now reads:

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs.—Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the Σ5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean (±SE) values over time for each location (hip, knee, etc.).

Section(s) also containing this change or similar changes:

- Synopsis, Statistical Methods
- Section 10.2.5 Healthcare Utilization Assessments
- Section 10.2.6 Interim Analysis

Purpose: Clarified procedures for efficacy assessments, adding the location at which to conduct assessments, and removing specified duration.

The primary change occurs in Section 8.1 Efficacy Parameters

Now reads: Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days at the CAS.

Purpose: Removed language indicating that anti-drug antibodies would only be analyzed if clinically indicated.

The primary change occurs in Section 8.1.17 Anti-drug Antibodies

Deleted text: Serum samples for anti-drug antibodies will be collected as specified in Table 1.—Samples may be analyzed, if elinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments, footnote u

# PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN

Protocol Version: Version 3.1-Brazil (Incorporating Amendment 2)

Protocol Date 20 January 2017

IND Number: 117395

EUDRACT Number 2014-003877-40

Sponsor: Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

Sponsor Contact:



The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

# **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to |
|---|
| maintain the confidentiality of all information received or developed in connection with this |
| protocol. |

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

# **Version History:**

|----------------|-------------------|-----------------------------------------|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 - Brazil | 16 September 2015 | Incorporating Brazil-Specific Amendment |
| 3.1 - Brazil | 20 January 2017 | Incorporating Global Amendment 2 |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

## **Name of Investigational Product:**

Patisiran

#### Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

## **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

# **Methodology:**

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (Patients).

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 (±3) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

## Reference therapy, dosage and mode of administration:

Not applicable.

#### Criteria for evaluation:

## **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Cardiac structure and function through echocardiograms and serum levels of terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid stimulating hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

## Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; ophthalmology examinations; and assessment of suicidal ideation and behavior.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Windo | ≤45 Days from<br>V Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | Xº | X° |
| Weight | | Prior | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | $X^d$ | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | X <sup>d</sup> | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | | $[X]^{f}$ |
| Vital Signs <sup>g</sup> | | X<br>Prior to Each Dose | | | | | |
| Safety Laboratory Assessments <sup>h</sup> | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test | X <sup>i</sup> | | X <sup>i</sup> (Prior to e | each dose) | <u> </u> | X | X |
| C-SSRS Questionnaire | | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TTR Protein (ELISA) | $X^{d}$ | | X | X | X | X | X |
| TSH and Vitamin A | | | | X | X | X° | Xº |
| Blood Sample for Long-term Storage | X | X | X | X | X | X | X |
| mNIS+7 <sup>j</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS+7 <sup>k</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS only | | | | | $X^{l}$ | $X^{m}$ | X <sup>m</sup> |
| Grip Strength Test <sup>n</sup> | X <sup>d</sup> | | | X | | | $[X]^f$ |
| 10-Meter Walk Test <sup>p</sup> | X <sup>d</sup> | | | X | | | $[X]^f$ |
| Ophthalmology Examination <sup>q</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>r</sup> | | | | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | X° | X° |
| Norfolk QOL-DN <sup>s</sup> | X <sup>d</sup> | | | X | X | X° | Xº |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | X° | Xº |
| Echocardiogram | $X^{d,t}$ | | | X | | | $[X]^f$ |
| Troponin I and NT-proBNP | $X^d$ | | | X | | | $[X]^{f}$ |
| Anti-Drug Antibody Testing <sup>u</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration <sup>v</sup> | X <sup>y</sup> | | X | • | | | |

| | | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|---|
| W | indow | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | | |
| Adverse Events | | | | Continuo | X <sup>b</sup><br>ous Monitorii | ng | | |
| Concomitant Medications | | X <sup>b</sup> Continuous Monitoring | | | | | | |

#### Table 1 Footnotes:

Abbreviations: C-SSRS = Columbia-Suicide Severity Rating Scale; COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- <sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- <sup>d</sup> Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- <sup>e</sup> mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.

Assessment/procedure required only if patient withdraws before the 52-week visit.

<sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.

<sup>h</sup>Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.

A urine-based pregnancy test will be performed on all females of child-bearing potential prior to dosing at all visits. In cases where a positive urine pregnancy test result is observed, a serum pregnancy test will be administered and the dose will be held. No dose will be administered until a negative pregnancy test is observed. Pregnancy test on the Day 0 Visit does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.

- j The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- k The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>m</sup> Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>n</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- <sup>p</sup> The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>q</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation. An electroretinogram may also be performed, as described in Section 9.1.6.
- <sup>r</sup>Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- s Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- <sup>t</sup>Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>u</sup> Serum samples for anti-drug antibodies will be collected as specified.
- Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study in the 21 (±3) day timeframe.

# **TABLE OF CONTENTS**

## SYNOPSIS3

| <b>TABLE</b> | OF CONTENTS | 11 |
|---|---|---|
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |
| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration. | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | |
| 8.1.4. | Modified Body Mass Index | 37 |
| 8.1.5. | Timed 10-meter Walk Test | 37 |
| 8.1.6. | Grip Strength Test | 38 |
| 8.1.7. | Composite Autonomic Symptom Score | 38 |
| 8.1.8. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.9. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.10. | Rasch-built Overall Disability Scale | 38 |
| 8.1.11. | Pharmacoeconomics Questionnaire | 38 |
| 8.1.12. | Echocardiogram and Biomarkers of Cardiac Function | |
| 8.1.13. | Transthyretin | 39 |
| 8.1.14. | Thyroid-Stimulating Hormone | 39 |
| 8.1.15. | Vitamin A | 39 |
| 8.1.16. | Anti-Drug Antibodies | 39 |
| 8.1.17. | Blood Sample for Long-term Storage. | 39 |
| 9. | ASSESSMENT OF SAFETY | 41 |
| 9.1. | Safety Parameters | 41 |
| 9.1.1. | Demographic and Medical History | 41 |
| 9.1.2. | Vital Signs | 41 |
| 9.1.3. | Weight and Height | 41 |
| 9.1.4. | Physical Examination | 41 |
| 9.1.5. | Laboratory Assessments | 41 |

| 9.1.6. | Ophthalmology Examination | 43 |
|---------|---------------------------------------------|----|
| 9.1.7. | Columbia-Suicide Severity Rating Scale | 43 |
| 9.2. | Adverse Events and Serious Adverse Events | |
| 9.2.1. | Definition of Adverse Events | 43 |
| 9.3. | Relationship to Study Drug | 44 |
| 9.4. | Recording Adverse Events | |
| 9.5. | Reporting Adverse Events | 45 |
| 9.5.1. | Serious Adverse Event Reporting | 45 |
| 9.5.2. | Pregnancy Reporting | 47 |
| 10. | STATISTICS | 48 |
| 10.1. | Sample Size | 48 |
| 10.2. | Statistical Methodology | 48 |
| 10.2.1. | Populations to be Analyzed | 48 |
| 10.2.2. | Baseline Evaluations | 48 |
| 10.2.3. | Efficacy Analyses | |
| 10.2.4. | Safety Analyses | 49 |
| 10.2.5. | Healthcare Utilization Assessments | 49 |
| 10.2.6. | Interim Analysis | 49 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 50 |
| 11.1. | Study Monitoring. | |
| 11.2. | Audits and Inspections | 50 |
| 11.3. | Institutional Review Board | 50 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 51 |
| 13. | ETHICS | 52 |
| 13.1. | Ethics Review | 52 |
| 13.2. | Ethical Conduct of the Study | 52 |
| 13.2.1. | Financial Disclosure Reporting Obligations. | 52 |
| 13.3. | Written Informed Consent | 52 |
| 14. | DATA HANDLING AND RECORD KEEPING | 54 |
| 14.1. | Case Report Forms | 54 |
| 14.2. | Confidentiality | 54 |
| 14.3. | Inspection of Records | 55 |

Table 1

14

## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RBP | retinol binding protein |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| ТР | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WT | wild type |

#### 1. INTRODUCTION

#### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). A,5,6 The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

#### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran Investigator's Brochure.

## 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

19

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### • Vitamin A Lowering

The suppression of serum levels of TTR and retinol binding protein (RBP) is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone

mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the Investigator's Brochure.

## 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

Confidential

#### 3. INVESTIGATIONAL PLAN

## 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 (±3) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

## 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

299

#### 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

#### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study

conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9,

CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

#### 5. TREATMENT OF PATIENTS

## 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

#### **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

## **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

## 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

#### 6. STUDY DRUG MATERIALS AND MANAGEMENT

## 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

## 6.2. Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

## 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

#### 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

#### 6.4.2. Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every 21 ( $\pm$ 3) days.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

#### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.
- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.

**Clinical Protocol** 

- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

#### 6.5. **Study Drug Accountability**

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

#### 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

## 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

#### 8. ASSESSMENT OF EFFICACY

### 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place at the CAS. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

#### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

## 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

311

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

#### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

## 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

#### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

#### 8.1.4. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

#### 8.1.5. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

312

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

#### 8.1.6. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

#### 8.1.7. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

#### 8.1.8. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.9. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

#### 8.1.10. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

#### 8.1.11. Pharmacoeconomics Questionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

#### 8.1.12. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

#### 8.1.13. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

#### **8.1.14.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.15. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

#### 8.1.16. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1.

#### 8.1.17. Blood Sample for Long-term Storage

To permit exploratory investigations and the application of novel approaches to bioanalysis that may further elucidate the outcomes of this study, or potentially advance understanding of the safety, mechanism of action and/or efficacy of patisiran, blood samples will be collected for long-term storage. These samples will be securely stored in a central biorepository for up to 10 years following the last patient last visit in this clinical study. After 10 years have elapsed, samples will be destroyed.

Details regarding the collection, processing, storage, and shipping of samples will be provided in the Laboratory Manual.

Exploratory analysis of these biospecimens will be performed by Alnylam Pharmaceuticals or its designees.

All study participants will be advised during the informed consent process of these biobanking details and the potential for exploratory investigation of their samples. Those who do not wish to contribute specimens to the biorepository will be asked to sign an "opt out" form. Moreover, patients who subsequently decide to withdraw consent for the utilization of such stored samples

will be able to do so, with the understanding that any data arising from samples already analyzed will be the property of Alnylam Pharmaceuticals.

#### 9. ASSESSMENT OF SAFETY

## 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

#### 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

#### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

#### 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

#### 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

#### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

## **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

#### 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

#### 9.1.5.5. Pregnancy Testing

A urine-based pregnancy test will be performed on all females of child-bearing potential prior to dosing at all visits, as specified in Table 1. In cases where a positive urine pregnancy test result is observed, a serum pregnancy test will be administered and the dose will be held. No dose will be administered until a negative pregnancy test is observed. Pregnancy test on the Day 0 Visit does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.

### 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

#### 9.1.7. Columbia-Suicide Severity Rating Scale

The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess each patient's mental status as it relates to suicidal ideation and behavior.

#### 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

43

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

## 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs.

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

## 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

## 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

## 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

• Patient's study number

- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or e-mail. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

#### 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.
#### 10. STATISTICS

# 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

#### 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### **10.2.2.** Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

## 10.2.3. Efficacy Analyses

Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory

and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

#### 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

A listing of healthcare utilization data will be presented.

#### 10.2.6. Interim Analysis

Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

## 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

#### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Medical Association Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

# 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

## 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

## 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

## 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

#### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| assistance needed. | 50 | Requires considerable assistance and frequent medical care. |
| | 40 | Disabled; requires special care and assistance. |
| Unable to care for self; requires | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| equivalent of institutional or hospital care; disease may be progressing rapidly. | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

**Appendix 2: New York Heart Association Classification of Heart Failure** 

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

# **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (18.6)^a$ |
| | | Sural SNAP, tibial motor n. distal latency, peroneal CMAP/motor n. conduction velocity/motor n. distal latency |
| | | • Vibration detection threshold (3.7) |
| | | Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies ∑5 (10) <sup>a</sup> |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

#### **ALN-TTR02-006 Protocol Version 3.1 Brazil**

Summary of Changes (dated 20 January 2017) compared to Protocol Version 2.1 Brazil (dated 16 September 2015)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Protocol Amendment**

The primary purpose of this amendment is to add the Columbia-Suicide Severity Rating Scale (C-SSRS) to the study assessments, which was inadvertently left out of previous versions of the protocol. The inclusion of the C-SSRS addresses a regulatory requirement to prospectively assess suicidality in clinical trials involving all drugs for neurological indications. Overall, this amendment includes the following changes:

- The Columbia-Suicide Severity Rating Scale has been added as an assessment of suicidal ideation and behavior.
- Electroretinograms are now recommended to be performed in the case of suspected retinal disease.
- The premedication regimen has been updated to align with commercially available doses.
- Blood samples for long-term storage have been added in order to permit future exploratory investigations.
- Reference to home infusions and to magnetic resonance neurography have been removed as they will not be performed in Brazil.

A detailed summary of the above changes, in addition to changes made for clarity, is provided in Table 1. Corrections to abbreviations, typographical errors and formatting are not detailed.

#### Table 1: Protocol Version 3.1 Brazil Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by bold font.

Purpose: Added Columbia-Suicide Severity Rating Scale to the study assessments

The primary change occurs in Table 1 Schedule of Assessments

Added text: Added row to Schedule of Assessments indicating that the Columbia-Suicide Severity Rating Scale is to be

collected at 26 weeks and 52 weeks after baseline and annually thereafter, as well as at the End of Study and Early

Withdrawal visits.

Section(s) also containing this change or similar changes:

• Synopsis, Criteria for Evaluation, Safety

• Section 9.1.7 Columbia-Suicide Severity Rating Scale (section added)

Purpose: To remove reference to home infusions as this will not be performed in Brazil.

The primary change occurs in Section 3.1 Overall Study Design

Deleted text: After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 (\pm 3)$ 

days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30 (\pm 5)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

Section(s) also containing this change or similar changes:

Synopsis methodology

• Table 1 Schedule of Assessments, Phone Contact row (removed)

• Table 1 Schedule of Assessments, Footnote y and Footnote z

• Section 5.3 Treatment Compliance

• Section 6.4.2 Study Drug Administration

Purpose: To update premedication regimen so that it aligns with commercially available doses.

The primary change occurs in Section 6.4.1 Premedication

Now reads: Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site).

Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg

PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Section(s) also containing this change or similar changes:

• Synopsis, Investigational product, dosage and mode of administration

Purpose: Added recommendation to collect an electroretinogram in the case of suspected retinal injury

The primary change occurs in Section 9.1.6 Ophthalmology Examination

Added text:

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments, footnote q

Purpose: Updated description of statistical analysis to align with currently planned analytic approach.

The primary change occurs in Section 10.2.3 Efficacy Analyses

Now reads:

Efficacy analyses will examine between and within patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma 5$  NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm SE$ ) values over time for each location (hip, knee, etc.).

Section(s) also containing this change or similar changes:

- Synopsis, Statistical Methods
- Section 10.2.5 Healthcare Utilization Assessments
- Section 10.2.6 Interim Analysis

Purpose: Added blood sampling for long-term storage in order to permit future exploratory investigations.

The primary change occurs in Table 1 Schedule of Assessments

Added text:

Added row to Schedule of Assessments indicating a blood sample for long-term storage is to be collected at each clinic visit.

Section(s) also containing this change or similar changes:

• Section 8.1.17 Blood Sample for Long-term Storage (section added)

Purpose: Clarified procedures for efficacy assessments, adding the location at which to conduct assessments, and removing specified duration.

The primary change occurs in Section 8.1 Efficacy Parameters

Now reads: Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days at the CAS.

Purpose: To remove reference to magnetic resonance neurography as this will not be performed in Brazil.

The primary change occurs in Section 8.1.4 Magnetic Resonance Neurography (removed section)

Deleted Section:

#### 8.1.4 Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for evaluation, Efficacy
- Table 1 Schedule of Assessments, MR neurography row (deleted)
- Table 1 Schedule of Assessments, footnote u (deleted)
- Section 8.1 Efficacy parameters

Purpose: Removed language indicating that anti-drug antibodies would only be analyzed if clinically indicated.

The primary change occurs in Section 8.1.16 Anti-drug Antibodies

Deleted text: Serum samples for anti-drug antibodies will be collected as specified in Table 1.—Samples may be analyzed, if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments, footnote u


# PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN


Version 2.1-Brazil (Incorporating Amendment 1)

Protocol Date

15 September 2015

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 

Signature ( & Sept 20 ( ) PPU

Date

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

# **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to |
|---|
| maintain the confidentiality of all information received or developed in connection with this |
| protocol. |

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

# **Version History:**

|----------------|-------------------|-----------------------------------------|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 | 15 September 2015 | Incorporating Brazil-Specific Amendment |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

## Name of Investigational Product:

Patisiran

#### **Title of Study:**

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

## **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

#### **Methodology:**

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study. Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 (±3) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study. unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0. After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm 5$ ) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### **Number of patients (planned):**

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\le 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\le 2.0$  (patients on anticoagulant therapy with an INR of  $\le 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### Reference therapy, dosage and mode of administration:

Not applicable.

#### Criteria for evaluation:

#### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography

- Cardiac structure and function through echocardiograms and serum levels of terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I
- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid Stimulating Hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of anti-drug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | Xº | Xº |
| Weight | | Prior t | X<br>to Each Dose | | | Xº | Xº |
| mBMI <sup>e</sup> | X <sup>d</sup> | | | X | X | Xº | Xº |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | X <sup>d</sup> | | | X | X | Xº | Xº |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | $[X]^f$ | [X] <sup>f</sup> |
| Vital Signs <sup>g</sup> | | Prior t | X<br>to Each Dose | | | | |
| Safety Laboratory Assessmentsh | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test | $X^k$ | | X <sup>k</sup> (Prior to 6 | each dose) | | X | X |
| TTR Protein (ELISA) | X | | X | X | X | X | X |

| | Day 0 Visit ≤45 Days from Last Dose <sup>a</sup> | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit<br>±4<br>Weeks | Annual<br>Visit<br>±6<br>Weeks | End of<br>Study<br>4 (+1)<br>Weeks<br>from<br>Last<br>Dose | Early Withdrawal Visit 4 (+1) Weeks from Last Dose |
|---|---|---|---|---|---|---|---|
| Window | | | | | | | |
| Procedure | | | | | | | |
| TSH and Vitamin A | | | | X | X | Xº | Xº |
| mNIS+7 <sup>1</sup> | $X^d$ | | | X | | $[X]^f$ | $[X]^f$ |
| NIS+7 <sup>m</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS only | | | | | X <sup>n</sup> | $X^{n,p}$ | $X^{n,p}$ |
| Grip Strength Test <sup>q</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| 10-Meter Walk Test <sup>r</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| Ophthalmology Examination <sup>s</sup> | X <sup>d</sup> | | | X | X | Xº | Xº |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | | X | X | Xº | Xº |
| MR Neurography <sup>u</sup> | | | | X | X | Xº | Xº |
| Pharmacoeconomics Questionnaire | X | | | X | X | Xº | Xº |
| Norfolk QOL-DN <sup>v</sup> | X <sup>d</sup> | | | X | X | Xº | Xº |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | Xº | Xº |
| Echocardiogram | $X^{d,w}$ | | | X | | $[X]^{\mathrm{f}}$ | $[X]^f$ |
| Troponin I and NT-proBNP | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>x</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration | Xy | | X <sup>y</sup> | • | | | |
| Phone Contact | | | Xz | | | | |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Adverse Events | | | Continuo | X <sup>b</sup><br>ous Monitori | ng | | |
| Concomitant Medications | | | Continuo | X <sup>b</sup><br>ous Monitori | ng | | |

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- <sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- <sup>d</sup> Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- <sup>e</sup> mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- <sup>f</sup> Assessment/procedure required only if patient withdraws before the 52-week visit.
- <sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- <sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- <sup>k</sup> A urine-based pregnancy test will be performed on all females of child-bearing potential prior to dosing at all visits. In cases where a positive urine pregnancy test result is observed, a serum pregnancy test will be administered and the dose will be held. No dose will be administered until a negative pregnancy test

is observed. Pregnancy test on the Day 0 Visit does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.

- <sup>1</sup> The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- <sup>p</sup> Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.
- <sup>t</sup> Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- <sup>u</sup> Required only for patients who had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in their parent study.
- v Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- w Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>x</sup> Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- y Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study within the 21 (±3) days timeframe. Doses may be administered at the clinical site or at home by a healthcare professional trained in the protocol.
- <sup>z</sup> Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use.

# **TABLE OF CONTENTS**

| SYNOPSIS | | 3 |
|---|---|---|
| TABLE OF CONTENTS. | | |
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |

| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | |
| 8.1.4. | Magnetic Resonance Neurography | 37 |
| 8.1.5. | Modified Body Mass Index | 38 |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.11. | Rasch-built Overall Disability Scale | 39 |
| 8.1.12. | | |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | 39 |
| 8.1.15. | Thyroid-Stimulating Hormone | 39 |
| 8.1.16. | Vitamin A | 39 |
| 8.1.17. | Anti-Drug Antibodies | 39 |
| 9. | ASSESSMENT OF SAFETY | 40 |
| 9.1. | Safety Parameters | 40 |
| 9.1.1. | Demographic and Medical History | 40 |
| 9.1.2. | Vital Signs | 40 |
| 9.1.3. | Weight and Height | 40 |
| 9.1.4. | Physical Examination | 40 |
| 9.1.5. | Laboratory Assessments | 40 |

| 9.1.6. | Ophthalmology Examination | 42 |
|-------------------------|--------------------------------------------|----|
| 9.2. | Adverse Events and Serious Adverse Events | 42 |
| 9.2.1. | Definition of Adverse Events | 42 |
| 9.3. | Relationship to Study Drug | 43 |
| 9.4. | Recording Adverse Events | 43 |
| 9.5. | Reporting Adverse Events | 44 |
| 9.5.1. | Serious Adverse Event Reporting | 44 |
| 9.5.2. | Pregnancy Reporting | 46 |
| 10. | STATISTICS | 47 |
| 10.1. | Sample Size | 47 |
| 10.2. | Statistical Methodology | 47 |
| 10.2.1. | Populations to be Analyzed | 47 |
| 10.2.2. | Baseline Evaluations | 47 |
| 10.2.3. | Efficacy Analyses | 47 |
| 10.2.4. Safety Analyses | | 48 |
| 10.2.5. | Healthcare Utilization Assessments | 48 |
| 10.2.6. | Interim Analysis | 48 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 49 |
| 11.1. | Study Monitoring | |
| 11.2. | | |
| 11.3. | Institutional Review Board | 49 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 50 |
| 13. | ETHICS | 51 |
| 13.1. | Ethics Review | 51 |
| 13.2. | Ethical Conduct of the Study | 51 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 51 |
| 13.3. | Written Informed Consent | 51 |
| 14. | DATA HANDLING AND RECORD KEEPING | 53 |
| 14.1. | Case Report Forms | 53 |
| 14.2. | Confidentiality | 53 |
| 14.3. | Inspection of Records | 53 |
| 14.4. | Retention of Records | 54 |

| Patisiran (ALN-TTR02)<br>Clinical Protocol | | ALN-TTR02-006<br>Version 2.1-Brazil (Amendment 1) |
|---|---|---|
| 15. | PUBLICATION POLICY | 55 |
| 16. | LIST OF REFERENCES | 56 |
| 17. | APPENDICES | 57 |
| | LIST OF TAB | LES |
| Table 1 | Schedule of Assessments | 7 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| НР | heat pain |
| HRdb | heart rate response to deep breathing |
| ICF informed consent form ICH International Conference on Harmonization IEC Independent Ethics Committee IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous INP lipid nanoparticle IBMI modified body mass index INP modified body mass index IMEDRA Medical Dictionary for Regulatory Activities IMIS Modified Neuropathy Impairment Score IMIS Modified Neuropathy Impairment Score IMIS Neuropathy Impairment Score INP NIS Neuropathy Impairment Score INP NIS Neuropathy Impairment Score INS Neuropathy Impairment Score INS Neuropathy Impairment Score INS Neuropathy Impairment Score INS-W Neuropathy Impairment S | Abbreviation | Definition |
|---|---|---|
| ICH International Conference on Harmonization IEC Independent Ethics Committee IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous ILNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | IB | Investigators Brochure |
| IEC Independent Ethics Committee IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous ILNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | ICF | informed consent form |
| IENFD intraepidermal nerve fiber density INN International Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | ICH | International Conference on Harmonization |
| INN International Nonproprietary Name INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous ILNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | IEC | Independent Ethics Committee |
| INR international normalized ratio IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IENFD | intraepidermal nerve fiber density |
| IRB Institutional Review Board IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score WIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | INN | International Nonproprietary Name |
| IRR infusion-related reaction IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter | INR | international normalized ratio |
| IRS interactive response system IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IRB | Institutional Review Board |
| IUD intrauterine device IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IRR | infusion-related reaction |
| IUS intrauterine system IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IRS | interactive response system |
| IV intravenous LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IUD | intrauterine device |
| LNP lipid nanoparticle mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IUS | intrauterine system |
| mBMI modified body mass index MedDRA Medical Dictionary for Regulatory Activities mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | IV | intravenous |
| MedDRA Medical Dictionary for Regulatory Activities Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- NES-W | LNP | lipid nanoparticle |
| mNIS Modified Neuropathy Impairment Score mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | mBMI | modified body mass index |
| mRNA messenger RNA MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | MedDRA | Medical Dictionary for Regulatory Activities |
| MR magnetic resonance NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | mNIS | Modified Neuropathy Impairment Score |
| NCS nerve conduction studies NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score-Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | mRNA | messenger RNA |
| NHP non-human primate NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | MR | magnetic resonance |
| NIS Neuropathy Impairment Score NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NCS | nerve conduction studies |
| NIS-W Neuropathy Impairment Score- Weakness NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NHP | non-human primate |
| NSAID nonsteroidal anti-inflammatory drug NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NIS | Neuropathy Impairment Score |
| NT-proBNP N-terminal prohormone of B-type natriuretic peptide NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NIS-W | Neuropathy Impairment Score- Weakness |
| NYHA New York Heart Association OTC over-the-counter PCS Patient Care Sites | NSAID | nonsteroidal anti-inflammatory drug |
| OTC over-the-counter PCS Patient Care Sites | NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| PCS Patient Care Sites | NYHA | New York Heart Association |
| | OTC | over-the-counter |
| PD pharmacodynamic | PCS | Patient Care Sites |
| | PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WHO | World Health Organization |
| WT | wild type |

# 1. INTRODUCTION

# 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR.<sup>1,2</sup> The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset.<sup>3</sup> There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC).<sup>4,5,6</sup> The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States.<sup>7,8</sup> The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.<sup>9</sup>

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. <sup>10</sup> The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

# 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in

serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

# 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the circulating amyloidogenic protein could impact the clinical course of the disease. Based on

nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

## • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone mineralization. If there are no medical contraindications, and per investigator judgment and

local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

# 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 \ (\pm 3)$  days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30 \ (\pm 5)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for

which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

## 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

# 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

# 4. SELECTION AND WITHDRAWAL OF PATIENTS

# 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

## 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study

6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

## 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development.<sup>14</sup> It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters,

or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2,

CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

# 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

## **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

# 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

# 6. STUDY DRUG MATERIALS AND MANAGEMENT

# 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# 6.2. Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

# 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

# **6.4.2.** Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every 21 (±3) days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done according to a site-specific plan by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

# 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of

patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

# 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

# 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

# 8. ASSESSMENT OF EFFICACY

# 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

# 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

# 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

# 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

## 8.1.4. Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. <sup>16</sup> This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

# 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

# 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

# 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

#### 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

# 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

## 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

# 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

## **8.1.12.** Pharmacoeconomics Ouestionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

# 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

# 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

## **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.16. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

## 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

# 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

# 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

## 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

## 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

# 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the

Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

# 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

# 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

# **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

#### 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

# 9.1.5.5. Pregnancy Testing

A urine-based pregnancy test will be performed on all females of child-bearing potential prior to dosing at all visits, as specified in Table 1. In cases where a positive urine pregnancy test result is observed, a serum pregnancy test will be administered and the dose will be held. No dose will be administered until a negative pregnancy test is observed. Pregnancy test on the Day 0 Visit does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.

# 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

# 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE

All IRRs will be recorded as AEs.

# 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)

- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

#### 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline

listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

# 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

## 10. STATISTICS

# 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

#### **10.2.1.** Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### 10.2.2. Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

# 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma 5$  NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm SE$ ) values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

# 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### **10.2.5.** Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

# 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

# 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

# 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

# 13. ETHICS

# 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

## 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes
requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

## 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the

drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

#### 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

## 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- 5 Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| inceded. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| | 40 | Disabled; requires special care and assistance. |
| Unable to care for self; requires | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| equivalent of institutional or hospital care; disease may be progressing rapidly. | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

**Appendix 2: New York Heart Association Classification of Heart Failure** 

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

**Appendix 4: Neuropathy Scores and Their Components** 

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NISa) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (18.6)^a$ |
| | | <ul> <li>Sural SNAP, tibial motor n. distal latency, peroneal<br/>SNAP/motor n. conduction velocity/motor n. distal<br/>latency</li> </ul> |
| | | • Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (10)^a$ |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

## **Country-Specific Amendment Summary of Changes for Brazil**

Protocol Version 2.1-Brazil, dated 15 September 2015, compared to Protocol Version 2.0 (Amendment 1.0), dated 08 September 2015

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Version 2.1-Brazil**

Consistent with Brazil-specific protocol ALN-TTR02-004, pregnancy testing for women of child-bearing potential prior to each dose of patisiran has been included in Brazil-specific protocol ALN-TTR02-006.

A detailed summary of changes is provided in Table 1. Corrections to typographical errors, punctuation, grammar, abbreviations, and formatting are not detailed.

## **Table 1: Version 2.1-Brazil Detailed Summary of Changes**

The primary section(s) of the protocol affected by the changes in this amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose: Add pregnancy testing for women of child-bearing potential be performed prior to each dose of patisiran.

Primary change: Section 9.1.5.5 Pregnancy Testing (formerly Pregnancy Screen)

Formerly read:

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is

specified in in Table 1; additional testing may be done any time pregnancy is suspected.

Now reads: A urine-based pregnancy test will be performed on all females of child-bearing potential prior to dosing at all

visits, as specified in Table 1. In cases where a positive urine pregnancy test result is observed, a serum pregnancy test will be administered and the dose will be held. No dose will be administered until a negative pregnancy test is observed. Pregnancy test on the Day 0 Visit does not need to be repeated if the patient had a

negative pregnancy test (urine or serum) within 14 days of the first dose.

Section(s) also containing this change:

• Table 1 Schedule of Assessments

#### ALN-TTR02-006 Protocol Amendment 2

Summary of Changes (dated 05 January 2017) compared to Protocol Version 2.1 France and Germany (dated 17 December 2015)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Protocol Amendment**

The primary purpose of this amendment is to add the Columbia-Suicide Severity Rating Scale (C-SSRS) to the study assessments, which was inadvertently left out of previous versions of the protocol. The inclusion of the C-SSRS addresses a regulatory requirement to prospectively assess suicidality in clinical trials involving all drugs for neurological indications. Overall, this amendment includes the following changes:

- The Columbia-Suicide Severity Rating Scale has been added as an assessment of suicidal ideation and behavior.
- Country-specific versions of the protocol have been integrated in order to increase consistency in the execution of the clinical study globally
- Electroretinograms are now recommended to be performed in the case of suspected retinal disease.
- The premedication regimen has been updated to align with commercially available doses.
- Blood samples for long-term storage have been added in order to permit future exploratory investigations.
- During scheduled phone contact, clinical sites may now ask patients who are receiving home infusions about their general experience receiving these infusions

A detailed summary of the above changes, in addition to changes made for clarity, is provided in Table 1. Corrections to abbreviations, typographical errors and formatting are not detailed.

## **Table 1: Protocol Amendment 2 Detailed Summary of Changes**

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose: Added Columbia-Suicide Severity Rating Scale to the study assessments

The primary change occurs in Table 1 Schedule of Assessments

Added text: Added row to Schedule of Assessments indicating that the Columbia-Suicide Severity Rating Scale is to be

collected at 26 weeks and 52 weeks after baseline and annually thereafter, as well as at the End of Study and Early

Withdrawal visits.

Section(s) also containing this change or similar changes:

Synopsis, Criteria for Evaluation, Safety

• Section 9.1.7 Columbia-Suicide Severity Rating Scale (section added)

Purpose: As part of global protocol integration, specified that home infusions are allowed only where applicable country and local regulations allow.

The primary change occurs in Section 3.1 Overall Study Design

Added text: After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 (±3) days, or.

Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a

healthcare professional trained on the protocol and delivery of premedications and patisiran.

Section(s) also containing this change or similar changes:

- Synopsis, Methodology
- Table 1, Schedule of Assessments
- Section 5.3 Treatment Compliance
- Section 6.4.2 Study Drug Administration

Purpose: As part of global protocol integration, specified that MR neurography is only to be conducted in Germany and France

The primary change occurs in Table 1 Schedule of Assessments, footnote s

Now reads:

MR neurography will only be conducted at sites in Germany and France. In these countries, neurography may be conducted for patients who had MR neurography in the parent study and may be performed for a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Imaging at baseline (Patients who had imaging in the parent study should have Day 0 visit imaging if they did not required for patients who underwent undergo MR neurography in the parent study within the past 3 months

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for evaluation, Efficacy
- Section 8.1 Efficacy Parameters
- Section 8.1.4 Magnetic Resonance Neurography (Germany and France Only)

Purpose: As part of global protocol integration, specified which studies patients may roll in from, and that the ALN-TTR02-003 study is not being conducted in Japan.

The primary change occurs in Section 3.1 Overall Study Design

Added text: Patients in this study will have completed "parent" study ALN-TTR02-003 or ALN-TTR02-004. Note that Study ALN-TTR02-003 is not being conducted in Japan.

Purpose: As part of global protocol integration, added Japan-specific recommendations regarding contraception.

The primary change occurs in Section 4.4 Pregnancy and Breastfeeding Restrictions / Contraception Requirements

Added text: In Japan it is recommended that the Investigators select appropriate contraception methods, as available.

Purpose: As part of global protocol integration, added Japan-specific instructions regarding duties related to study drug accountability.

The primary change occurs in Section 6.5 Study Drug Accountability

Added text: The Investigator or designee (or in Japan, the responsible pharmacist designated according to the Japan local

regulations) will maintain accurate records of receipt and the condition of the patisiran supplied for this study,

including dates of receipt.

Purpose: As part of global protocol integration, added statement on compensation for health damages as per local regulations.

The primary change occurs in Section 13.4 Compensation for Health Damages (section added)

Added text:

#### 13.4 Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required per local regulations

Purpose: To update premedication regimen so that it aligns with commercially available doses.

The primary change occurs in Section 6.4.1 Premedication

Now reads: Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site).

Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg

PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Section(s) also containing this change or similar changes:

• Synopsis, Investigational product, dosage and mode of administration

Purpose: Added recommendation to collect an electroretinogram in the case of suspected retinal injury

The primary change occurs in Section 9.1.6 Ophthalmology Examination

Added text:

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Updated description of statistical analysis to align with currently planned analytic approach.

The primary change occurs in Section 10.2.3 Efficacy Analyses

Now reads:

Efficacy analyses will examine between and within patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm$ SE) values over time for each location (hip, knee, etc.).

Section(s) also containing this change or similar changes:

- Synopsis, Statistical Methods
- Section 10.2.5 Healthcare Utilization Assessments
- Section 10.2.6 Interim Analysis

Purpose: Added blood sampling for long-term storage in order to permit future exploratory investigations.

The primary change occurs in Table 1 Schedule of Assessments

Added text:

Added row to Schedule of Assessments indicating a blood sample for long-term storage is to be collected at each clinic visit.

Section(s) also containing this change or similar changes:

• Section 8.1.18 Blood Sample for Long-term Storage (section added)

Purpose: Added questionnaire regarding experience of home infusions to scheduled phone contact for home infusion patients.

The primary change occurs in Table 1 Schedule of Assessments, footnote x

Added text:

x. Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every  $30 \ (\pm 5)$  days for assessment of adverse events and concomitant medication use. **During phone contact, patients may also be asked additional questions about their general experience receiving infusions at home.** 

Purpose: Added a definition of "woman of child-bearing potential".

The primary change occurs in Section 4.4 Pregnancy and Breastfeeding Restrictions / Contraception Requirements

Added text:

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

Purpose: Clarified language on Vitamin A dosing and added Japan-specific instructions.

The primary change occurs in Section 5.2 Concomitant Medications

Now reads:

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan, the clinical sites will provide patients with a prescription for vitamin

Section(s) also containing this change or similar changes:

- Section 6.4.2 Study Drug Administration
- Section 8.1.16 Vitamin A

Purpose: Clarified procedures for efficacy assessments, adding the location at which to conduct assessments, and removing specified duration.

The primary change occurs in Section 8.1 Efficacy Parameters

Now reads: Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days at the CAS.

Purpose: Removed language indicating that anti-drug antibodies would only be analyzed if clinically indicated.

The primary change occurs in Section 8.1.17 Efficacy Parameters

Deleted text: Serum samples for anti-drug antibodies will be collected as specified in Table 1.—Samples may be analyzed, if

clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Clarified that no study procedures may occur until approval is granted by all appropriate parties.

The primary change occurs in Section 13.1 Ethics Review

Added text: The Investigator should not start any study procedure with the patient until documentation of the approval

by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator

and Alnylam Pharmaceuticals, Inc.

## PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN


Version 2.1 (Incorporating Amendment 1) - France

and Germany

Protocol Date

17 December 2015

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



Date

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

## **INVESTIGATOR'S AGREEMENT**

I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

# **Version History:**

|---|---|---|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 | 17 December 2015 | Incorporating French and German Specific Update |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

## Name of Investigational Product:

Patisiran

#### **Title of Study:**

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

#### Methodology:

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 (±3) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm$ 5) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### **Number of patients (planned):**

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

#### Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### Reference therapy, dosage and mode of administration:

Not applicable.

## Criteria for evaluation:

#### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography
- Cardiac structure and function through echocardiograms and serum levels of terminal

prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid Stimulating Hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | X° | X° |
| Weight | | Prior t | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | $X^d$ | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | $X^d$ | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | $[X]^{f}$ | $[X]^{f}$ |
| Vital Signs <sup>g</sup> | | Prior 1 | X<br>to Each Dose | • | | | |
| Safety Laboratory Assessments <sup>h</sup> | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | $X^k$ | | X | X | X | X | X |
| TTR Protein (ELISA) | X | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TSH and Vitamin A | | | | X | X | X° | X° |
| mNIS+7 <sup>1</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS+7 <sup>m</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS only | | | | | X <sup>n</sup> | $X^{n,p}$ | $X^{n,p}$ |
| Grip Strength Test <sup>q</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| 10-Meter Walk Test <sup>r</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| Ophthalmology Examination <sup>s</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | | X | X | X° | X° |
| MR Neurography <sup>u</sup> | X | | X | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | X° | X° |
| Norfolk QOL-DN <sup>v</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | $[X]^{f}$ | $[X]^f$ |
| R-ODS Disability | $X^d$ | | | X | | $[X]^f$ | $[X]^f$ |
| EQ-5D QOL | $X^d$ | | | X | X | X° | X° |
| Echocardiogram | $X^{d,w}$ | | | X | | $[X]^f$ | $[X]^f$ |
| Troponin I and NT-proBNP | $X^{d}$ | | | X | | $[X]^{f}$ | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>x</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration | X <sup>y</sup> | | $X^{y}$ | • | | | |
| Phone Contact | | | X <sup>z</sup> | | | | |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Wine | ≤45 Days from Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Adverse Events | | | Continuo | X <sup>b</sup><br>ous Monitori | ng | | |
| Concomitant Medications | | X <sup>b</sup> Continuous Monitoring | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- <sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- <sup>d</sup> Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- e mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f Assessment/procedure required only if patient withdraws before the 52-week visit.
- <sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- <sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- <sup>k</sup> Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.
- The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on


separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patient in the patient in the patient in the patient.

- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- P Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.
- Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- <sup>u</sup> Required for patients who had MR neurography in the parent study and may be performed for a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Imaging at baseline (Day 0 visit) is not required for patients who underwent MR neurography in the parent study within the past 3 months.
- <sup>v</sup> Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- w Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>x</sup> Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study within the 21 (±3) days timeframe. Doses may be administered at the clinical site or at home by a healthcare professional trained in the protocol.
- <sup>z</sup> Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use.

# **TABLE OF CONTENTS**

# SYNOPSIS3

| TABLE | OF CONTENTS | 1 |
|---|---|---|
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 2: |
| 4.3. | Patient Withdrawal Criteria | 20 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 20 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 3 |
| 6.1. | Study Drug Packaging and Labeling | 3 |
| 6.2. | Study Drug Storage | 3 |
| 6.3. | Study Drug Preparation | 3 |
| 6.4. | Administration | 32 |

| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | 37 |
| 8.1.4. | Magnetic Resonance Neurography | 37 |
| 8.1.5. | Modified Body Mass Index | 38 |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.11. | Rasch-built Overall Disability Scale | 39 |
| 8.1.12. | Pharmacoeconomics Questionnaire | 39 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | 39 |
| 8.1.15. | Thyroid-Stimulating Hormone | 39 |
| 8.1.16. | Vitamin A | 39 |
| 8.1.17. | Anti-Drug Antibodies | 39 |
| 9. | ASSESSMENT OF SAFETY | 40 |
| 9.1. | Safety Parameters | 40 |
| 9.1.1. | Demographic and Medical History | 40 |
| 9.1.2. | Vital Signs | 40 |

| Chineari | version 2.1 (timenament 1 Trance and Germany) 1 | 7 December 2018 |
|----------|-------------------------------------------------|-----------------|
| 9.1.3. | Weight and Height | 40 |
| 9.1.4. | Physical Examination | 40 |
| 9.1.5. | Laboratory Assessments | 40 |
| 9.1.5.1. | Hematology | 41 |
| 9.1.5.2. | Blood Chemistry | 41 |
| 9.1.5.3. | Urinalysis | 41 |
| 9.1.5.4. | Coagulation | 41 |
| 9.1.5.5. | Pregnancy Screen | 42 |
| 9.1.6. | Ophthalmology Examination | 42 |
| 9.2. | Adverse Events and Serious Adverse Events | 42 |
| 9.2.1. | Definition of Adverse Events | 42 |
| 9.2.1.1. | Adverse Event | 42 |
| 9.2.1.2. | Serious Adverse Event. | 42 |
| 9.3. | Relationship to Study Drug | 43 |
| 9.4. | Recording Adverse Events | 43 |
| 9.5. | Reporting Adverse Events | 44 |
| 9.5.1. | Serious Adverse Event Reporting | 44 |
| 9.5.2. | Pregnancy Reporting | 45 |
| 10. | STATISTICS | 47 |
| 10.1. | Sample Size | 47 |
| 10.2. | Statistical Methodology | 47 |
| 10.2.1. | Populations to be Analyzed | 47 |
| 10.2.2. | Baseline Evaluations. | 47 |
| 10.2.3. | Efficacy Analyses | 47 |
| 10.2.4. | Safety Analyses | 48 |
| 10.2.5. | Healthcare Utilization Assessments | 48 |
| 10.2.6. | Interim Analysis | 48 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 49 |
| 11.1. | Study Monitoring | 49 |

11.2.11.3.

12.13.

Audits and Inspections 49

ETHICS 51

| Clinical Protocol Version 2.1 (Amendment 1 - France and Germany) 17 | | many) 17 December 2015 |
|---|---|---|
| 13.1. | Ethics Review | 51 |
| 13.2. | Ethical Conduct of the Study | |
| 13.2.1. | Financial Disclosure Reporting Obligations | |
| 13.3. | Written Informed Consent | |
| 14. | DATA HANDLING AND RECORD KEEPING | 53 |
| 14.1. | Case Report Forms | 53 |
| 14.2. | Confidentiality | 53 |
| 14.3. | Inspection of Records | 54 |
| 14.4. | Retention of Records | 54 |
| 15. | PUBLICATION POLICY | 55 |
| 16. | LIST OF REFERENCES | 56 |
| 17. | APPENDICES | 57 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| ЕР | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |

WBC

WHO

WT

white blood cell

wild type

World Health Organization
### 1. INTRODUCTION

## 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

## 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated. with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### • Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

#### 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 \ (\pm 3)$  days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30 \ (\pm 5)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for

which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

# 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

#### 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

## 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# **4.4.** Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study conducted with

patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9,

CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

#### 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

## **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

# 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

## 6. STUDY DRUG MATERIALS AND MANAGEMENT

# 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

#### 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

## **6.4.2.** Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every  $21 \ (\pm 3)$  days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done according to a site-specific plan by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

## 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of

patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - 1) If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

# 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

# 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

#### 8. ASSESSMENT OF EFFICACY

# 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

# 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

#### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

#### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

# 8.1.4. Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for a subset of patients providing informed consent who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography. This assessment will be performed serially at 6-month intervals for the first year and then yearly thereafter.

# 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

#### 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

## 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

#### 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

#### 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

# 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

#### 8.1.12. Pharmacoeconomics Questionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

# 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

#### 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

#### **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### **8.1.16.** Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

#### 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

#### 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

# 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

## 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

# 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

## 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

## 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

## **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

## 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

#### 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

#### 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

#### 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to

prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day

should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

# 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within

24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.

```
Medpace SAE hotline – USA:
Telephone: PPD ext. PPD or PPD ext. PPD
Facsimile: PPD or PPD

Medpace SAE hotline – Europe:
Telephone: PPD
Facsimile: PPD
Facsimile: PPD
```

Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

# 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be

discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

## 10. STATISTICS

# **10.1.** Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

#### **10.2.1.** Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### **10.2.2.** Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

#### 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma 5$  NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean  $(\pm SE)$  values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

#### 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### **10.2.5.** Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

#### 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

#### 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

## 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

#### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

#### 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC,

the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

#### 14. DATA HANDLING AND RECORD KEEPING

# 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.
## 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

## 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

#### 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

#### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- 3 Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- 5 Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

## 17. APPENDICES

**Appendix 1: Karnofsky Scale** 

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| assistance needed. | 50 | Requires considerable assistance and frequent medical care. |
| | 40 | Disabled; requires special care and assistance. |
| Unable to care for self; requires | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| equivalent of institutional or hospital care; disease may be progressing rapidly. | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

## **Appendix 2: New York Heart Association Classification of Heart Failure**

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

## **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (18.6)^a$ |
| | | Sural SNAP, tibial motor n. distal latency, peroneal SNAP/motor n. conduction velocity/motor n. distal latency |
| | | Vibration detection threshold (3.7) |
| | | Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (10)^a$ |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

# ALN-TTR02-006 Protocol Version 2.1 – France and Germany Summary of Changes

Protocol Version 2.1 – France and Germany (Incorporating French and German-specific update), dated 17 December 2015, compared to Protocol Version 2.0 (Amendment 1), dated 08 September 2015

A Multicenter, Open-Label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Protocol Amendment**

The primary purpose for this country-specific (France and Germany) protocol amendment is to add two additional MR neurography assessment time points to the schedule of assessments. These additional time points will permit exploration of the effect of patisiran on lower limb nerve injury at 6-month intervals for the first year and then yearly thereafter in patients who elected to undergo serial MR neurography on the parent study or in a subset of patients who provide informed consent to participate for the first time in this assessment on the ALN-TTR02-006 study.

A detailed summary of changes is provided in Table 1. The addition of new reference(s), corrections to typographical errors, punctuation, grammar, abbreviations, and formatting are not detailed.

## **Table 1: Protocol Amendment 6.1 Detailed Summary of Changes**

The primary section(s) of the protocol affected by the changes in Protocol Amendment 2.1 are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose: Addition of timepoints at the Day 0 Visit and at the 26 Week Visit for the MR neurography assessment

The primary change occurs in Table 1, Schedule of Assessments.

Added text: In the table, "X," was added to the row labeled, "MR Neurography," in the corresponding Day 0 and 26 Week columns.

Purpose: To expand information provided in the Table 1 footnote for the MR neurography assessment

The primary change occurs in footnote "u" of Table 1, Schedule of Assessments.

Added text: Required only for patients who had MR neurography in the parent study and may be imaged performed for a subset of consenting patients providing informed consent who did not have MR neurography previously in their parent study. Imaging at baseline (Day 0 visit) not required for patients who underwent MR neurography on the parent study within the past 3 months.

*Purpose:* New text to note the 6-month intervals applied to the MR neurography assessment.

The primary change occurs in Section 8.1.4, Magnetic Resonance Neurography.

Added text: Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting a subset of patients providing informed consent who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography. This assessment will be performed serially at 6-month intervals for the first year and then yearly thereafter.

Purpose: Addition of new references, correct typographical errors, punctuation, grammar, abbreviations, and formatting.

These changes are not listed individually.

#### **ALN-TTR02-006 Protocol Amendment 2**

Summary of Changes (dated 05 January 2017) compared to Protocol Version 2.2 - Japan (dated 14 March 2016)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Protocol Amendment**

The primary purpose of this amendment is to add the Columbia-Suicide Severity Rating Scale (C-SSRS) to the study assessments, which was inadvertently left out of previous versions of the protocol. The inclusion of the C-SSRS addresses a regulatory requirement to prospectively assess suicidality in clinical trials involving all drugs for neurological indications. Overall, this amendment includes the following changes:

- The Columbia-Suicide Severity Rating Scale has been added as an assessment of suicidal ideation and behavior.
- Country-specific versions of the protocol have been integrated in order to increase consistency in the execution of the clinical study globally
- Electroretinograms are now recommended to be performed in the case of suspected retinal disease.
- The premedication regimen has been updated to align with commercially available doses.
- Blood samples for long-term storage have been added in order to permit future exploratory investigations.
- During scheduled phone contact, clinical sites may now ask patients who are receiving home infusions about their general experience receiving these infusions

A detailed summary of the above changes, in addition to changes made for clarity, is provided in Table 1. Corrections to abbreviations, typographical errors and formatting are not detailed.

#### Table 1: Protocol Amendment 2 Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose: As part of global protocol integration, replaced "APOLLO" study with "parent" study, and specified that ALN-TTR02-003 is not being conducted in Japan.

The primary change occurs in Section 3.1 Overall Study Design

Added text:

Patients in this study will have completed "parent" study ALN-TTR02-003 or ALN-TTR02-004. Note that Study ALN-TTR02-003 is not being conducted in Japan.

Section(s) also containing this change or similar changes:

• Throughout protocol wherever "APOLLO" appeared

Purpose: As part of global protocol integration, added magnetic resonance neurography to the protocol as a safety assessment, specifying it is only applicable for patients in Germany and France

The primary change occurs in Table 1 Schedule of Assessments, footnote s

Added text:

s. MR neurography will only be conducted at sites in Germany and France. In these countries, neurography may be conducted for patients who had MR neurography in the parent study and for a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Patients who had imaging in the parent study should have Day 0 imaging if they did not undergo MR neurography within the past 3 months.

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for evaluation, Efficacy
- Section 8.1 Efficacy Parameters
- Section 8.1.4 Magnetic Resonance Neurography (Germany and France Only) (Section has been added)

Purpose: Added Columbia-Suicide Severity Rating Scale to the study assessments

The primary change occurs in Table 1 Schedule of Assessments

Added text:

Added row to Schedule of Assessments indicating that the Columbia-Suicide Severity Rating Scale is to be collected at 26 weeks and 52 weeks after baseline and annually thereafter, as well as at the End of Study and Early

Withdrawal visits.

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for Evaluation, Safety
- Section 9.1.7 Columbia-Suicide Severity Rating Scale (section added)

Purpose: As part of global protocol integration, added the option for home infusions, specifying they may occur only where applicable country and local regulations allow.

The primary change occurs in Section 3.1 Overall Study Design

Added text:

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 (±3) days. Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 (±5) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

Section(s) also containing this change or similar changes:

- Synopsis, Methodology
- Table 1, Schedule of Assessments
- Section 5.3 Treatment Compliance
- Section 6.4.2 Study Drug Administration

Purpose: As part of global protocol integration, added that study will be conducted in accordance with HIPAA in the US.

The primary change occurs in Section 13.2 Ethical Conduct of the Study

Added text:

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Medical Association Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA) in the US, and all other applicable medical privacy laws and regulations.

Purpose: To update premedication regimen so that it aligns with commercially available doses.

The primary change occurs in Section 6.4.1 Premedication

Now reads: Intravenous H1 blocker: di

Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg

PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Section(s) also containing this change or similar changes:

• Synopsis, Investigational product, dosage and mode of administration

Purpose: Added recommendation to collect an electroretinogram in the case of suspected retinal injury

The primary change occurs in Section 9.1.6 Ophthalmology Examination

Added text:

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Updated description of statistical analysis to align with currently planned analytic approach.

The primary change occurs in Section 10.2.3 Efficacy Analyses

Now reads:

Efficacy analyses will examine between and within patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm$ SE) values over time for each location (hip, knee, etc.).

Section(s) also containing this change or similar changes:

- Synopsis, Statistical Methods
- Section 10.2.5 Healthcare Utilization Assessments
- Section 10.2.6 Interim Analysis

Purpose: Added blood sampling for long-term storage in order to permit future exploratory investigations.

The primary change occurs in Table 1 Schedule of Assessments

Added text:

Added row to Schedule of Assessments indicating a blood sample for long-term storage is to be collected at each clinic visit.

Section(s) also containing this change or similar changes:

• Section 8.1.18 Blood Sample for Long-term Storage (section added)

Purpose: Added questionnaire regarding experience of home infusions to scheduled phone contact for home infusion patients.

The primary change occurs in Table 1 Schedule of Assessments, footnote x

Added text: x. Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every

30 (±5) days for assessment of adverse events and concomitant medication use. **During phone contact, patients** 

may also be asked additional questions about their general experience receiving infusions at home.

Purpose: Clarified procedures for efficacy assessments, adding the location at which to conduct assessments, and removing specified duration.

The primary change occurs in Section 8.1 Efficacy Parameters

Now reads: Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days at the CAS.

Purpose: Removed language indicating that anti-drug antibodies would only be analyzed if clinically indicated.

The primary change occurs in Section 8.1.17 Efficacy Parameters

Deleted text: Serum samples for anti-drug antibodies will be collected as specified in Table 1.—Samples may be analyzed, if

clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

## PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

## A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH **PATISIRAN**


Version 2.2-Japan (Incorporating Amendment 1)

Protocol Date

14 March 2016

IND Number:

117395

**EUDRACT Number** 

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



Date

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

## **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to |
|---|
| maintain the confidentiality of all information received or developed in connection with this |
| protocol. |

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

## **Version History:**

|----------------|-------------------|----------------------------------------|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 | 14 October 2015 | Incorporating Japan-Specific Amendment |
| 2.2 | 14 March 2016 | Incorporating Japan-Specific Amendment |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

#### Name of Investigational Product:

Patisiran

#### **Title of Study:**

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

#### Methodology:

This is a multicenter, multinational, open-label, extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study. Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 (±3) days for the duration of the study. In order to maintain the every-21-day dosing schedule from the prior clinical study (APOLLO study), patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the APOLLO study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the APOLLO study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the APOLLO study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter. A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the APOLLO study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### **Number of patients (planned):**

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the APOLLO study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq$  2.5 × the upper limit of normal (ULN), international normalized ratio (INR)  $\leq$  2.0 (patients on anticoagulant therapy with an INR of  $\leq$  3.5 will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the APOLLO study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the APOLLO study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H<sub>2</sub> blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H<sub>2</sub> blocker dose)
- Intravenous H<sub>1</sub> blocker: diphenhydramine 50 mg (or equivalent other IV H<sub>1</sub> blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H<sub>1</sub> blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

#### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS+7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the APOLLO study)
- Cardiac structure and function through echocardiograms and serum levels of terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid Stimulating Hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the APOLLO study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the APOLLO study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | X° | X° |
| Weight | | Prior t | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | $X^d$ | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | $X^d$ | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | $[X]^f$ | $[X]^{f}$ |
| Vital Signs <sup>g</sup> | | Prior t | X<br>to Each Dose | | | | |
| Safety Laboratory Assessments <sup>h</sup> | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | $X^k$ | | X | X | X | X | X |
| TTR Protein (ELISA) | X | | X | X | X | X | X |

| | Day 0 Visit ≤45 Days from Last Dose <sup>a</sup> | 12 Week<br>Visit | 26 Week<br>Visit<br>±4 Weeks | 52 Week<br>Visit<br>±4<br>Weeks | Annual<br>Visit<br>±6<br>Weeks | End of<br>Study<br>4 (+1)<br>Weeks<br>from<br>Last<br>Dose | Early Withdrawal Visit 4 (+1) Weeks from Last Dose |
|---|---|---|---|---|---|---|---|
| Window | | | | | | | |
| Procedure | | | | | | | |
| TSH and Vitamin A | | | | X | X | X° | X° |
| mNIS+7 <sup>1</sup> | X <sup>d</sup> | | | X | | $[X]^{f}$ | $[X]^f$ |
| NIS+7 <sup>m</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS only | | | | | X <sup>n</sup> | $X^{n,p}$ | $X^{n,p}$ |
| Grip Strength Test <sup>q</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| 10-Meter Walk Test <sup>r</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| Ophthalmology Examination <sup>s</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | | X | X | Xº | Xº |
| Pharmacoeconomics Questionnaire | X | | | X | X | X° | X° |
| Norfolk QOL-DN <sup>u</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| COMPASS 31 Questionnaire | $X^d$ | | | X | | $[X]^f$ | $[X]^f$ |
| R-ODS Disability | $X^d$ | | | X | | $[X]^f$ | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | X° | X° |
| Echocardiogram | $X^{d,w}$ | | | X | | $[X]^{f}$ | $[X]^f$ |
| Troponin I and NT-proBNP | $X^d$ | | | X | | $[X]^{f}$ | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>w</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration | X <sup>x</sup> | | X <sup>x</sup> | | | | |
| Adverse Events | X <sup>b</sup> Continuous Monitoring | | | | | | |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Wind | ≤45 Days from<br>Days Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Concomitant Medications | | X <sup>b</sup> Continuous Monitoring | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin


<sup>&</sup>lt;sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the APOLLO study. However, the Day 0 visit may occur within 45 days after the last dose in the APOLLO study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.

<sup>&</sup>lt;sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the APOLLO study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the APOLLO study will be entered into the database.

<sup>&</sup>lt;sup>c</sup> Assessment does not need to be repeated. Information will be obtained from APOLLO study.

<sup>&</sup>lt;sup>d</sup> Assessment/procedure does not need to be repeated if performed during the APOLLO study within 45 days of first dose in this study.

<sup>&</sup>lt;sup>e</sup> mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.

f Assessment/procedure required only if patient withdraws before the 52-week visit.

<sup>&</sup>lt;sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.

<sup>&</sup>lt;sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.

<sup>&</sup>lt;sup>k</sup> Assessment does not need to be repeated if the patient had a negative pregnancy test (urine) within 14 days of the first dose.

<sup>&</sup>lt;sup>1</sup> The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on

492

separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patient in the patient in the patient in the patient.

- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- <sup>p</sup> Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.
- Optional skin biopsies will only be obtained if the patient had skin biopsies in the APOLLO study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- <sup>u</sup> Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- <sup>v</sup> Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>w</sup> Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- x Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the APOLLO study within the 21 (±3) days timeframe. Doses will be administered at the clinical site.

## **TABLE OF CONTENTS**

| S | V | NI | $\cap$ | D | Q. | IQ | -2 |
|----|----|----|--------|---|----|----|----|
| N. | 1. | LΝ | U | 1 | D. | IJ | ני |

| <b>TABLE</b> | E OF CONTENTS | 11 |
|---|---|---|
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 21 |
| 3. | INVESTIGATIONAL PLAN | 21 |
| 3.1. | Overall Study Design | 21 |
| 3.2. | Number of Patients | 22 |
| 3.3. | Treatment Assignment | 22 |
| 3.4. | Criteria for Study Termination | 22 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 23 |
| 4.1. | Patient Inclusion Criteria | 23 |
| 4.2. | Patient Exclusion Criteria | 23 |
| 4.3. | Patient Withdrawal Criteria | 24 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 24 |
| 5. | TREATMENT OF PATIENTS | 27 |
| 5.1. | Description of Study Drug | 27 |
| 5.2. | Concomitant Medications | 27 |
| 5.3. | Treatment Compliance | 28 |
| 5.4. | Randomization and Blinding | 28 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 28 |
| 6.1. | Study Drug Packaging and Labeling | 28 |
| 6.2. | Study Drug Storage | 28 |
| 6.3. | Study Drug Preparation | 29 |
| 6.4. | Administration | 29 |

| 6.4.1. | Premedication | 29 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 30 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 31 |
| 6.5. | Study Drug Accountability | 31 |
| 6.6. | Study Drug Handling and Disposal | 32 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 32 |
| 8. | ASSESSMENT OF EFFICACY | 32 |
| 8.1. | Efficacy Parameters | 32 |
| 8.1.1. | Neurological Testing | 32 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 33 |
| 8.1.1.2. | Neurological Impairment Score | 33 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 33 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | 34 |
| 8.1.4. | Modified Body Mass Index | 34 |
| 8.1.5. | Timed 10-meter Walk Test | 34 |
| 8.1.6. | Grip Strength Test. | 34 |
| 8.1.7. | Composite Autonomic Symptom Score | 34 |
| 8.1.8. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 35 |
| 8.1.9. | EuroQoL Quality of Life Questionnaire | 35 |
| 8.1.10. | Rasch-built Overall Disability Scale | 35 |
| 8.1.11. | Pharmacoeconomics Questionnaire | 35 |
| 8.1.12. | Echocardiogram and Biomarkers of Cardiac Function | 35 |
| 8.1.13. | Transthyretin | 35 |
| 8.1.14. | Thyroid-Stimulating Hormone | 35 |
| 8.1.15. | Vitamin A | 36 |
| 8.1.16. | Anti-Drug Antibodies | 36 |
| 9. | ASSESSMENT OF SAFETY | 36 |
| 9.1. | Safety Parameters | 36 |
| 9.1.1. | Demographic and Medical History | 36 |
| 9.1.2. | Vital Signs | 36 |
| 9.1.3. | Weight and Height | 36 |

| 9.1.4. | Physical Examination | 36 |
|----------|-------------------------------------------|----|
| 9.1.5. | Laboratory Assessments | 37 |
| 9.1.5.1. | Hematology | 37 |
| 9.1.5.2. | Blood Chemistry | 37 |
| 9.1.5.3. | Urinalysis | 37 |
| 9.1.5.4. | Coagulation | 38 |
| 9.1.5.5. | Pregnancy Screen. | 38 |
| 9.1.6. | Ophthalmology Examination | 38 |
| 9.2. | Adverse Events and Serious Adverse Events | 38 |
| 9.2.1. | Definition of Adverse Events | 38 |
| 9.2.1.1. | Adverse Event | 38 |
| 9.2.1.2. | Serious Adverse Event | 38 |
| 9.3. | Relationship to Study Drug | 39 |
| 9.4. | Recording Adverse Events | 39 |
| 9.5. | Reporting Adverse Events | 40 |
| 9.5.1. | Serious Adverse Event Reporting. | 40 |
| 9.5.2. | Pregnancy Reporting | 42 |
| 10. | STATISTICS | 42 |
| 10.1. | Sample Size | 42 |
| 10.2. | Statistical Methodology | 42 |
| 10.2.1. | Populations to be Analyzed | 42 |
| 10.2.2. | Baseline Evaluations | 43 |
| 10.2.3. | Efficacy Analyses | 43 |
| 10.2.4. | Safety Analyses | 43 |
| 10.2.5. | Healthcare Utilization Assessments | 4 |
| 10.2.6. | Interim Analysis | 44 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 44 |
| 11.1. | Study Monitoring. | 44 |
| 11.2. | Audits and Inspections | 44 |
| 11.3. | Institutional Review Board | 44 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 45 |
| 13 | FTHICS | 45 |

| 13.1. | Ethics Review | 45 |
|---------|--------------------------------------------|----|
| 13.2. | Ethical Conduct of the Study | 46 |
| 13.2.1. | Financial Disclosure Reporting Obligations | |
| 13.3. | Written Informed Consent | 46 |
| 13.4. | Compensation for Health Damages | 47 |
| 14. | DATA HANDLING AND RECORD KEEPING | 47 |
| 14.1. | Case Report Forms | 47 |
| 14.2. | Confidentiality | 47 |
| 14.3. | Inspection of Records | 48 |
| 14.4. | Retention of Records | 48 |
| 15. | PUBLICATION POLICY | 48 |
| 16. | LIST OF REFERENCES | 49 |
| 17. | APPENDICES | 50 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| APOLLO | Study name given to the Phase 3 study ALN-TTR02-004 |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| HRdb | heart rate response to deep breathing |
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WHO | World Health Organization |
| WT | wild type |

## 1. INTRODUCTION

#### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

#### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of *in vitro* and *in vivo* studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (> 80% reduction from pretreatment baseline) was observed at doses  $\geq 0.15$  mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated. with maximum TTR knockdown of ~90% and sustained TTR suppression of > 80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of > 80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

#### 1.3. **Study Design Rationale**

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this openlabel study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### 1.4. **Risk-Benefit Assessment**

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and lifethreatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### • Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary among different countries and among different individuals within a country, all patients on the study will be asked to take a daily supplement that contains the recommended daily allowance of vitamin A. Patients should have started an adequate daily intake of vitamin A by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone
mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

## 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

#### 3. INVESTIGATIONAL PLAN

## 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm$  3 days. In order to maintain the every 21-day dosing schedule from the prior clinical study (APOLLO study), patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the APOLLO study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the APOLLO study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the APOLLO study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the APOLLO study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 (\pm 3)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS]"), while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the APOLLO study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on APOLLO study. A combination of the center number, APOLLO study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by Alnylam Pharmaceuticals, Inc.

Alnylam Pharmaceuticals, Inc. reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to Alnylam Pharmaceuticals, Inc. or the CRO, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

## 4. SELECTION AND WITHDRAWAL OF PATIENTS

## 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the APOLLO study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

#### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the APOLLO study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the APOLLO study

6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of Alnylam Pharmaceuticals, Inc., including if Alnylam Pharmaceuticals, Inc. terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with Alnylam Pharmaceuticals, Inc. before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development.<sup>14</sup> It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters,

or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-

dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by *in vitro* human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

It is recommended that the Investigators select appropriate contraception method in Japan as available.

Pregnancy reporting guidelines are provided in Section 9.5.2.

## 5. TREATMENT OF PATIENTS

## 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

## **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is < 20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥ 20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the APOLLO study in accordance with the rules of that study protocol. For patients who did not take these medications while on the APOLLO study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. The Japan clinical sites will provide the subjects with a prescription for vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF.

Similarly, concomitant medications that continue from the APOLLO study will be entered into the database.

## **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the study site for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

## 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

#### 6. STUDY DRUG MATERIALS AND MANAGEMENT

## 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3^{\circ}$ C. Any deviation from the recommended storage conditions must be reported to the CRO and/or Alnylam Pharmaceuticals, Inc. and use of the patisiran halted until authorization for its continued use has been given by Alnylam Pharmaceuticals, Inc. or its designee.

No special procedures for the safe handling of patisiran are required. An Alnylam Pharmaceuticals, Inc. representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

## 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days (±3 days). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

## 6.4. Administration

#### **6.4.1.** Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H<sub>2</sub> blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H<sub>2</sub> blocker dose)
- Intravenous H<sub>1</sub> blocker: diphenhydramine 50 mg (or equivalent other IV H<sub>1</sub> blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H<sub>1</sub> blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

• If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.

- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

## 6.4.2. Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every 21 (±3) days.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the APOLLO study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window ( $\pm 3$  days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. The Japan clinical sites will provide the subjects with a prescription for vitamin A.

#### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H<sub>1</sub>/H<sub>2</sub> receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.
- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - 1) If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The investigator or the responsible pharmacist for study drug (designated according to the Japan local regulations) will maintain accurate records of the receipt and condition of patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed

and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by Alnylam Pharmaceuticals, Inc. or its designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

## 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to Alnylam Pharmaceuticals, Inc. or its designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

## 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

## 8. ASSESSMENT OF EFFICACY

## 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the APOLLO study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

#### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

#### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the APOLLO study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual

Skin biopsies will be performed at a CAS or PCS.

## 8.1.4. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

#### 8.1.5. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

#### 8.1.6. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

## 8.1.7. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

### 8.1.8. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.9. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

### 8.1.10. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

## 8.1.11. Pharmacoeconomics Questionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

## 8.1.12. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

## 8.1.13. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

## **8.1.14.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.15. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A.

#### 8.1.16. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

#### 9. ASSESSMENT OF SAFETY

## 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

## 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the APOLLO study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the APOLLO study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

## 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the APOLLO study.

#### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance;

head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

## 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

### 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

#### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

## **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH

- Leukocytes
- Bilirubin

- Specific gravity
- Ketones
- Protein
- Glucose

- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

## 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

### 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

## 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual

#### 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

Results in death

- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

# 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

#### 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.

```
Medpace SAE hotline – USA:
Telephone: PPD ext. PPD or PPD ext. PPD
Facsimile: PPD or PPD

Medpace SAE hotline – Europe:
Telephone: PPD
Facsimile: PPD
```

Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

Alnylam Pharmaceuticals, Inc. or the CRO will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after Alnylam Pharmaceuticals, Inc. or the CRO has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after Alnylam Pharmaceuticals, Inc. or the CRO has first knowledge of them.

The Investigator may be informed by Alnylam Pharmaceuticals, Inc. or the CRO of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports

should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to Alnylam Pharmaceuticals, Inc. as part of the trial master file on study completion.

## 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

#### 10. STATISTICS

## **10.1.** Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

#### 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### 10.2.2. Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the APOLLO study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

### 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the APOLLO study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the APOLLO study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS+7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma 5$  NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm SE$ ) values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

#### 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

## 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

## 11.1. Study Monitoring

The Clinical Monitor, as a representative of Alnylam Pharmaceuticals, Inc., has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by Alnylam Pharmaceuticals, Inc. or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator and the study site will permit study-related monitoring, audits, and review by the IEC or IRB or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by Alnylam Pharmaceuticals, Inc. or the CRO or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow Alnylam Pharmaceuticals, Inc., the CRO, or regulatory agencies access to all study records.

#### 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

## 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, Alnylam may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to Alnylam Pharmaceuticals, Inc. or its designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by Alnylam Pharmaceuticals, Inc. and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

#### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

The Investigator should not start any study procedure with the patient until documentation of the approval by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator and Alnylam Pharmaceuticals, Inc.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by Alnylam Pharmaceuticals, Inc. or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply Alnylam

Pharmaceuticals, Inc. with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

## 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, and all other applicable medical privacy laws and regulations.

## 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

Alnylam Pharmaceuticals, Inc. or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by Alnylam Pharmaceuticals, Inc. or its designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to Alnylam Pharmaceuticals, Inc. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to Alnylam Pharmaceuticals, Inc.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

## 13.4. Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required.

#### 14. DATA HANDLING AND RECORD KEEPING

## 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

Alnylam Pharmaceuticals, Inc. will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow the CRO and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by Alnylam Pharmaceuticals, Inc. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to Alnylam Pharmaceuticals, Inc. or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to Alnylam Pharmaceuticals, Inc. or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to Alnylam Pharmaceuticals, Inc. (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and Alnylam Pharmaceuticals, Inc., thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. Alnylam Pharmaceuticals, Inc. must approve any transfer of information not directly involved in the study.

## 14.3. Inspection of Records

Alnylam Pharmaceuticals, Inc. will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing Alnylam Pharmaceuticals, Inc. in writing and giving Alnylam Pharmaceuticals, Inc. the opportunity to store the records for a longer period of time at Alnylam Pharmaceuticals, Inc.'s expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

#### 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at Alnylam Pharmaceuticals, Inc. at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by Alnylam Pharmaceuticals, Inc., or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and Alnylam Pharmaceuticals, Inc. confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by Alnylam Pharmaceuticals, Inc.

#### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- 5 Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| inceded. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

**Appendix 2: New York Heart Association Classification of Heart Failure** 

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

**Appendix 4: Neuropathy Scores and Their Components** 

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NISa) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies ∑5 (18.6) <sup>a</sup> |
| | | Sural SNAP, tibial motor n. distal latency, peroneal SNAP/motor n. conduction velocity/motor n. distal latency |
| | | Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies ∑5 (10) <sup>a</sup> |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

## ALN-TTR02-006 Protocol Version 2.2 - Japan

## **Summary of Changes**

Protocol Version 2.2-Japan (Incorporating Japan-specific update), dated 14 March 2016, compared to Protocol Version 2.1-Japan, dated 14 October 2015

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

## Rationale for the Japan Country-specific Protocol Amendment

• The primary purpose of the Japan country-specific protocol amendment is to remove home infusion references and MR neurography scanning as these practices are not applicable in Japan, and to update the vitamin A dispensing requirments to better align with country-specific pharmacy practices.

The following additional change was incorporated:

- Changed reference from "parent study" to "APOLLO study"; this change is being implemented because only Japanese subjects from the APOLLO study (ALN-TTR02-004) will be rolling into this extension study ALN-TTR02-006; none of the subjects participating in the other patisiran parent study (ALN-TTR02-003) are from Japan.
- The name of the Sponsor was added in-text as Alnylam Pharmaceuticals.
- Deleted from Section 13.2, text describing the Health Insurance Portability and Accountability Act of 1996 (HIPAA) that is only applicable in the United States of America.
- New Section 13.4 was added to describe Compensation for Health Damages according to local regulations.

A detailed summary of changes is provided in Table 1. Corrections to typographical errors, punctuation, grammar, abbreviations, and formatting (including administrative changes between protocol amendments 2.1 and 2.2) are not detailed.
#### Table 1: Protocol Amendment 3 Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in this amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

Purpose: Removal of text describing or referencing home infusion

The primary change occurs in Section 3.1, Overall Study Design, paragraph 5.

Deleted text:

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 (±5) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

Sections also containing this change:

- Synopsis, Methodology, paragraph 3
- Table 1, Schedule of Assessment to remove the Phone Contact row and corresponding footnote.
- Section 5.3, Treatment Compliance
- Section 6.4.2, Study Drug Administration

Purpose: Removal of text describing MR neurography scanning assessment

The primary change occurs in Section 8.1, Efficacy Parameters, second paragraph

Deleted text:

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Sections also containing this change:

- Synopsis, Criteria for evaluation, Efficacy, removal of MR neurography bullet
- Table 1, Schedule of Assessment to remove the MR neurography scanning assessment row and corresponding footnote.
- Section 8.1.4, Magnetic Resonance Neurography subsection deleted entirely.

Purpose: Update the vitamin A dispensing requirments

The primary change occurs in Section 5.2, Concomitant Medications, paragraph 4

Deleted text: All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. The Japan clinical sites will provide the subjects with a prescription for vitamin A.

Sections also containing this change:

• Section 6.2.4, Study Drug Administration last paragraph

Purpose: Changed reference from "parent study" to "APOLLO study

The primary change occurs in Section 3.1, Overall Study Design, paragraph 2

Changed Text:

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm$  3 days. In order to maintain the every 21-day dosing schedule from the parent prior clinical study (APOLLO study), patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parentAPOLLO study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parentAPOLLO study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parentAPOLLO study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

Sections also containing this change:

- Synopsis, Methodology, Diagnosis and eligibility criteria, Criteria for (efficacy) evaluation, and Statistical methods sections
- Table 1, Schedule of Assessment footnotes
- Section 3.3, Treatment Assignment
- Section 4.1, Patient Inclusion Criteria
- Section 4.2, Patient Exclusion Criteria
- Section 5.2, Concomitant Medications
- Section 6.4.2, Study Drug Administration
- Section 8.1, Efficacy Parameters
- Section 9.1, Safety Parameters
- Section 10, Statistics

Purpose: The name of the Sponsor was added in-text as Alnylam Pharmaceuticals

The primary change occurs in Section 3.4, Criteria for Study Termination

Changed text:

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the SponsorAlnylam Pharmaceuticals, Inc.

The SponsorAlnylam Pharmaceuticals, Inc. reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representativeAlnylam Pharmaceuticals, Inc. or the CRO, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

Sections also containing this change:

- Synopsis, Methodology, Diagnosis and eligibility
- Section 4.3, Patient Withdrawal Criteria
- Section 6.2, Study Drug Storage
- Section 6.5, 6.5. Study Drug Accountability
- Section 9.5.1, 9.5.1. Serious Adverse Event Reporting
- Section 11, Direct Access to Source Data/Documents
- Section 12, Quality Control and Quality Assurance
- Section 13, Ethics
- Section 14, Data Handling and Record Keeping
- Section 15, Publication Policy

Purpose: Deleted text referring to the HIPAA that is only applicable in the United States of America.

The change occurs in Section 13.2, Ethical Conduct of the Study

#### Deleted text:

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations

Purpose: Provided clarification that written notification of the approval from the IEC/IRB from the head of the study site to the Investigator and Alnylam Pharmaceuticals, Inc.should be provided before the start of study procedures.

The change occurs in Section 13.1, Ethics Review

Added text:

The Investigator should not start any study procedure with the patient until documentation of the approval by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator and Alnylam Pharmaceuticals, Inc.

Purpose: New Section 13.4 was added to describe Compensation for Health Damages according to local regulations

The change occurs in newly added Section 13.4, Compensation for Health Damages

Added text:

#### 13.4. Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required.

Purpose: Correct typographical errors, punctuation, grammar, abbreviations, and formatting[, including administrative changes, if appropriate] These changes are not listed individually.

## PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN

Protocol Version: Version 2.1-Japan (Incorporating Amendment 1)

Protocol Date 14 October 2015

IND Number: 117395

EUDRACT Number 2014-003877-40

Sponsor: Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

# **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to |
|---|
| maintain the confidentiality of all information received or developed in connection with this |
| protocol. |

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date. |

# **Version History:**

|----------------|-------------------|----------------------------------------|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 | 14 October 2015 | Incorporating Japan-Specific Amendment |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

#### **Name of Investigational Product:**

Patisiran

#### Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

#### Methodology:

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every 21 ( $\pm 3$ ) days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm$ 5) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

#### Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

#### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography
- Cardiac structure and function through echocardiograms and serum levels of terminal

prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid Stimulating Hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | X° | X° |
| Weight | | Prior t | X<br>to Each Dose | • | | X° | X° |
| mBMI <sup>e</sup> | $X^d$ | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | $X^d$ | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | $[X]^f$ | $[X]^f$ |
| Vital Signs <sup>g</sup> | | Prior t | X<br>to Each Dose | | | | |
| Safety Laboratory Assessments <sup>h</sup> | $X^d$ | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | $X^k$ | | X | X | X | X | X |
| TTR Protein (ELISA) | X | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TSH and Vitamin A | | | | X | X | X° | X° |
| mNIS+7 <sup>1</sup> | X <sup>d</sup> | | | X | | $[X]^{f}$ | $[X]^{f}$ |
| NIS+7 <sup>m</sup> | $X^d$ | | | X | | $[X]^{f}$ | $[X]^{f}$ |
| NIS only | | | | | $X^n$ | $X^{n,p}$ | $X^{n,p}$ |
| Grip Strength Test <sup>q</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| 10-Meter Walk Test <sup>r</sup> | $X^d$ | | | X | | $[X]^f$ | $[X]^f$ |
| Ophthalmology Examination <sup>s</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | | X | X | X° | X° |
| MR Neurography <sup>u</sup> | | | | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | X° | X° |
| Norfolk QOL-DN <sup>v</sup> | $X^d$ | | | X | X | X° | X° |
| COMPASS 31 Questionnaire | $X^d$ | | | X | | $[X]^f$ | $[X]^f$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | X° | X° |
| Echocardiogram | $X^{d,w}$ | | | X | | $[X]^{f}$ | $[X]^f$ |
| Troponin I and NT-proBNP | $X^{d}$ | | | X | | $[X]^f$ | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>x</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration | X <sup>y</sup> | | X <sup>y</sup> | | | | |
| Phone Contact | | | Xz | | | | |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Wine | ≤45 Days from Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Adverse Events | | X <sup>b</sup> Continuous Monitoring | | | | | |
| Concomitant Medications | | X <sup>b</sup> Continuous Monitoring | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- b Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- d Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- e mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f Assessment/procedure required only if patient withdraws before the 52-week visit.
- <sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- <sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- <sup>k</sup> Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.
- The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on

552

separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patient in the patient in the patient in the patient.

- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- P Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.
- Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- <sup>u</sup> Required only for patients who had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in their parent study.
- <sup>v</sup> Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- w Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>x</sup> Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- <sup>y</sup> Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study within the 21 (±3) days timeframe. Doses may be administered at the clinical site or at home by a healthcare professional trained in the protocol.
- <sup>z</sup> Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use.

# **TABLE OF CONTENTS**

| SYNOR | SIS | 3 |
|---|---|---|
| TABLE | OF CONTENTS | 11 |
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design. | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |

| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | |
| 8.1.4. | Magnetic Resonance Neurography | 37 |
| 8.1.5. | Modified Body Mass Index | 38 |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.11. | Rasch-built Overall Disability Scale | 39 |
| 8.1.12. | Pharmacoeconomics Questionnaire | 39 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | 39 |
| 8.1.15. | Thyroid-Stimulating Hormone | 39 |
| 8.1.16. | Vitamin A | 39 |
| 8.1.17. | Anti-Drug Antibodies | 39 |
| 9. | ASSESSMENT OF SAFETY | 40 |
| 9.1. | Safety Parameters | 40 |
| 9.1.1. | Demographic and Medical History | 40 |
| 9.1.2. | Vital Signs | 40 |

| 9.1.3. | Weight and Height | 40 |
|----------|-------------------------------------------|----|
| 9.1.4. | Physical Examination | 40 |
| 9.1.5. | Laboratory Assessments | 40 |
| 9.1.5.1. | Hematology | 41 |
| 9.1.5.2. | Blood Chemistry | 41 |
| 9.1.5.3. | Urinalysis | 41 |
| 9.1.5.4. | Coagulation | 42 |
| A sample | e for INR assessment will be collected | 42 |
| 9.1.5.5. | Pregnancy Screen | 42 |
| 9.1.6. | Ophthalmology Examination | 42 |
| 9.2. | Adverse Events and Serious Adverse Events | 42 |
| 9.2.1. | Definition of Adverse Events | 42 |
| 9.2.1.1. | Adverse Event | 42 |
| 9.2.1.2. | Serious Adverse Event | 42 |
| 9.3. | Relationship to Study Drug | 43 |
| 9.4. | Recording Adverse Events | 43 |
| 9.5. | Reporting Adverse Events | 44 |
| 9.5.1. | Serious Adverse Event Reporting. | 44 |
| 9.5.2. | Pregnancy Reporting | 46 |
| 10. | STATISTICS | 47 |
| 10.1. | Sample Size | 47 |
| 10.2. | Statistical Methodology | 47 |
| 10.2.1. | Populations to be Analyzed | 47 |
| 10.2.2. | Baseline Evaluations | 47 |
| 10.2.3. | Efficacy Analyses | 47 |
| 10.2.4. | Safety Analyses | 48 |
| 10.2.5. | Healthcare Utilization Assessments | 48 |
| 10.2.6. | Interim Analysis | 48 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 49 |
| 11.1. | Study Monitoring | 49 |
| 11.2. | Audits and Inspections | 49 |
| 11 3 | Institutional Review Board | 40 |

| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 50 |
|---------|--------------------------------------------|----|
| 13. | ETHICS | 51 |
| 13.1. | Ethics Review | 51 |
| 13.2. | Ethical Conduct of the Study | 51 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 51 |
| 13.3. | Written Informed Consent | 51 |
| 14. | DATA HANDLING AND RECORD KEEPING | 53 |
| 14.1. | Case Report Forms | 53 |
| 14.2. | Confidentiality | 53 |
| 14.3. | Inspection of Records | 54 |
| 14.4. | Retention of Records | 54 |
| 15. | PUBLICATION POLICY | 55 |
| 16. | LIST OF REFERENCES | 56 |
| 17. | APPENDICES | 57 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| IB | Investigators Brochure |
|-----------|-----------------------------------------------------|
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WHO | World Health Organization |
| WT | wild type |

#### 1. INTRODUCTION

#### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. <sup>1,2</sup> The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). <sup>4,5,6</sup> The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. <sup>7,8</sup> The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age. <sup>9</sup>

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

#### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated, with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

#### 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

#### • Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

#### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone

mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

#### 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 \ (\pm 3)$  days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every  $30 \ (\pm 5)$  days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for

which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

#### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

# 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

#### 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

#### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study

conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

It is recommended that the Investigators select appropriate contraception method in Japan as available.

Pregnancy reporting guidelines are provided in Section 9.5.2.

#### 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

#### **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

#### 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

#### 6. STUDY DRUG MATERIALS AND MANAGEMENT

## 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

#### 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.
#### 6.4.2. Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every 21 (±3) days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done according to a site-specific plan by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window ( $\pm 3$  days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran.

#### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower

infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - 1) If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

## 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

## 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

## 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

#### 8. ASSESSMENT OF EFFICACY

## 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

#### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

#### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

## 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

#### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

#### 8.1.4. Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

#### 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

#### 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

#### 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

#### 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

#### 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

#### 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

#### 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

#### 8.1.12. Pharmacoeconomics Questionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

## 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

## 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

#### **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.16. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

#### 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

581

#### 9. ASSESSMENT OF SAFETY

## 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

#### 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

#### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

#### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

#### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

#### 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

#### 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

#### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

#### **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

#### 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

#### 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

#### 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

## 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity

- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

## 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

## 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

## 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

#### 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the

completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

#### 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

#### 10. STATISTICS

## 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

## 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

#### 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### 10.2.2. Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

#### 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean  $(\pm SE)$  values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

#### 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

#### 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

#### 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

## 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

## 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

#### 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

## 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

#### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

## 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

#### 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

#### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

#### 14. DATA HANDLING AND RECORD KEEPING

## 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

#### 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

#### 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

#### 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

#### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- 3 Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- 5 Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- 16 Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

## 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| inceded. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

**Appendix 2: New York Heart Association Classification of Heart Failure** 

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

## **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 270 | | Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (18.6)^a$ |
| | | Sural SNAP, tibial motor n. distal latency, peroneal SNAP/motor n. conduction velocity/motor n. distal latency |
| | | • Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (10)^a$ |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

## **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

## Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

#### **Country-Specific Amendment Summary of Changes for Japan**

Protocol Version 2.1-Japan dated 14 October 2015, compared to Protocol Version 2.0 (Amendment 1.0), dated 08 September 2015

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Version 2.1-Japan**

Consistent with Japan-specific protocol ALN-TTR02-004, the following changes have been made to the ALN-TTR02-006 Japan-specific protocol:

- Added the definitions for women of childbearing potential and a post-menopausal women
- Recommended that the Investigators select appropriate contraception method in Japan, as available
- Clarified that patients will receive daily vitamin A supplementation for the duration of their participation in the study while being administered study drug

A detailed summary of changes is provided in Table 1. Corrections to typographical errors, punctuation, grammar, abbreviations, and formatting are not detailed.

1

## **Table 1: Version 2.1-Japan Detailed Summary of Changes**

The primary section(s) of the protocol affected by the changes in this amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by **bold** font.

| Purpose: | Added the definitions for women of childbearing potential and a post-menopausal women |
|---|---|
| Primary change: | Section 4.4 Pregnancy and Breastfeeding Restrictions/Contraception Requirements |
| Added text: | Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy. |
| Purpose: | Recommended that the Investigators select appropriate contraception method in Japan, as available |
| Primary change: | Section 4.4 Pregnancy and Breastfeeding Restrictions/Contraception Requirements |
| Added text: | It is recommended that the Investigators select appropriate contraception method in Japan as available. |
| Purpose: | Clarified that patients will receive daily vitamin $A$ supplementation for the duration of their participation in the study while being administered study drug |
| Primary change: | Section 6.4.2 Study Drug Administration |
| Added text: | In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. |
| Section(s) also containing this change: | Section 5.2 Concomitant Medications |

## PATISIRAN (ALN-TTR02)

#### **ALN-TTR02-006**

# A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH PATISIRAN


Version 2.1-Taiwan (Incorporating Amendment 1)

Protocol Date

10 December 2015

IND Number:

117395

**EUDRACT** Number

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



Date

The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

## **INVESTIGATOR'S AGREEMENT**

| I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree | ree to |
|---|---|
| maintain the confidentiality of all information received or developed in connection with this | S |
| protocol. | |

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

## **Version History:**

|----------------|-------------------|--------------------------------------|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1-Taiwan | 10 Decmeber 2015 | Incorporating Global Amendment 1 and |
| | | Taiwan-specific change |

2

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

#### Name of Investigational Product:

Patisiran

#### Title of Study:

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

#### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

#### Methodology:

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every  $21 \text{ (\pm 3)}$  days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm$ 5) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

3

#### Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

#### Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq$ 2.5 × the upper limit of normal (ULN), international normalized ratio (INR)  $\leq$ 2.0 (patients on anticoagulant therapy with an INR of  $\leq$ 3.5 will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤ 2 X ULN are eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court
### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

## Reference therapy, dosage and mode of administration:

Not applicable.

#### Criteria for evaluation:

## **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography
- Cardiac structure and function through echocardiograms and serum levels of terminal

prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid Stimulating Hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; and ophthalmology examinations.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Efficacy analyses will examine between- and within-subject rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional exploratory analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | X° | X° |
| Weight | | Prior t | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | $X^d$ | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | $[X]^f$ | $[X]^{f}$ |
| Vital Signs <sup>g</sup> | | Prior 1 | X<br>to Each Dose | | | | |
| Safety Laboratory Assessments <sup>h</sup> | $X^d$ | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | $X^k$ | | X | X | X | X | X |
| TTR Protein (ELISA) | X | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TSH and Vitamin A | | | | X | X | Xº | Xº |
| mNIS+7 <sup>1</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^{f}$ |
| NIS+7 <sup>m</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| NIS only | | | | | X <sup>n</sup> | $X^{n,p}$ | $X^{n,p}$ |
| Grip Strength Test <sup>q</sup> | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| 10-Meter Walk Test <sup>r</sup> | X <sup>d</sup> | | | X | | $[X]^{f}$ | $[X]^{f}$ |
| Ophthalmology Examination <sup>s</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>t</sup> | | | | X | X | Xº | X° |
| MR Neurography <sup>u</sup> | | | | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | Xº | X° |
| Norfolk QOL-DN <sup>v</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| COMPASS 31 Questionnaire | $X^d$ | | | X | | $[X]^{f}$ | $[X]^{f}$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | $[X]^f$ | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | X° | X° |
| Echocardiogram | $X^{d,w}$ | | | X | | $[X]^{f}$ | $[X]^f$ |
| Troponin I and NT-proBNP | X <sup>d</sup> | | | X | | $[X]^{\mathrm{f}}$ | $[X]^{f}$ |
| Anti-Drug Antibody Testing <sup>x</sup> | | | X | X | X | X | X |
| Premedication / Patisiran Administration | X <sup>y</sup> | | $X^{y}$ | • | | | |
| Phone Contact | | | Xz | | | | |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Win | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Adverse Events | | X <sup>b</sup> Continuous Monitoring | | | | | |
| Concomitant Medications | | X <sup>b</sup> Continuous Monitoring | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- <sup>a</sup> Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- <sup>b</sup> Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- <sup>c</sup> Assessment does not need to be repeated. Information will be obtained from parent study.
- <sup>d</sup> Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- <sup>e</sup> mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f Assessment/procedure required only if patient withdraws before the 52-week visit.
- <sup>g</sup> Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- <sup>h</sup> Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- <sup>k</sup> Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.
- <sup>1</sup> The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on

616

separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patient in the patient in the patient in the patient.

- <sup>m</sup> The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- <sup>n</sup> One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- <sup>o</sup> Assessment does not need to be repeated if done within the previous 26 weeks.
- P Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- <sup>q</sup> Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- <sup>s</sup> Examination will include visual acuity, visual fields, and slit-lamp evaluation.
- Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- <sup>u</sup> Required only for patients who had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in their parent study.
- <sup>v</sup> Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- w Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- <sup>x</sup> Serum samples for anti-drug antibodies will be collected as specified. Samples may be analyzed, if clinically indicated.
- Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study within the 21 (±3) days timeframe. Doses may be administered at the clinical site or at home by a healthcare professional trained in the protocol.
- <sup>z</sup> Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use.

# **TABLE OF CONTENTS**

| SYNOP | SIS | 3 |
|---|---|---|
| TABLE | OF CONTENTS | 11 |
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance. | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage. | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |

| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | |
| 8.1.4. | Magnetic Resonance Neurography | 37 |
| 8.1.5. | Modified Body Mass Index | |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.11. | Rasch-built Overall Disability Scale | 39 |
| 8.1.12. | Pharmacoeconomics Questionnaire | 39 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | 39 |
| 8.1.15. | Thyroid-Stimulating Hormone | 39 |
| 8.1.16. | Vitamin A | 39 |
| 8.1.17. | Anti-Drug Antibodies | 39 |
| 9. | ASSESSMENT OF SAFETY | 40 |
| 9.1. | Safety Parameters | 40 |
| 9.1.1. | Demographic and Medical History | 40 |
| 9.1.2. | Vital Signs | 40 |

| 9.1.3. | Weight and Height | 40 |
|----------|-------------------------------------------|----|
| 9.1.4. | Physical Examination | 40 |
| 9.1.5. | Laboratory Assessments | 40 |
| 9.1.5.1. | Hematology | 41 |
| 9.1.5.2. | Blood Chemistry | 41 |
| 9.1.5.3. | Urinalysis | 41 |
| 9.1.5.4. | Coagulation | 42 |
| 9.1.5.5. | Pregnancy Screen. | 42 |
| 9.1.6. | Ophthalmology Examination | 42 |
| 9.2. | Adverse Events and Serious Adverse Events | 42 |
| 9.2.1. | Definition of Adverse Events | 42 |
| 9.2.1.1. | Adverse Event | 42 |
| 9.2.1.2. | Serious Adverse Event | 42 |
| 9.3. | Relationship to Study Drug | 43 |
| 9.4. | Recording Adverse Events | 43 |
| 9.5. | Reporting Adverse Events | 44 |
| 9.5.1. | Serious Adverse Event Reporting | 44 |
| 9.5.2. | Pregnancy Reporting | 46 |
| 10. | STATISTICS | 47 |
| 10.1. | Sample Size | 47 |
| 10.2. | Statistical Methodology | 47 |
| 10.2.1. | Populations to be Analyzed | 47 |
| 10.2.2. | Baseline Evaluations. | 47 |
| 10.2.3. | Efficacy Analyses | 47 |
| 10.2.4. | Safety Analyses | 48 |
| 10.2.5. | Healthcare Utilization Assessments | 48 |
| 10.2.6. | Interim Analysis | 48 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 49 |
| 11.1. | Study Monitoring | 49 |
| 11.2. | Audits and Inspections | 49 |
| 11.3. | Institutional Review Board | 49 |
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 50 |

| 13. | ETHICS | 51 |
|---------|--------------------------------------------|----|
| 13.1. | Ethics Review | 51 |
| 13.2. | Ethical Conduct of the Study | 51 |
| 13.2.1. | Financial Disclosure Reporting Obligations | 51 |
| 13.3. | Written Informed Consent | 51 |
| 14. | DATA HANDLING AND RECORD KEEPING | 53 |
| 14.1. | Case Report Forms | 53 |
| 14.2. | Confidentiality | 53 |
| 14.3. | Inspection of Records | 54 |
| 14.4. | Retention of Records | 54 |
| 15. | PUBLICATION POLICY | 55 |
| 16. | LIST OF REFERENCES | 56 |
| 17. | APPENDICES | 57 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | 7 |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| ТР | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WHO | World Health Organization |
| WT | wild type |

# 1. INTRODUCTION

## 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

## 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated. with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran IB.

# 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

# 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and life-threatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the

circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

#### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

#### • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

### • Vitamin A Lowering

The suppression of serum levels of TTR and RBP is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

# Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone

mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the IB.

# 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

# 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 ( $\pm 3$ ) days, or receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm 5$ ) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for

which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

## 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

# 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

# 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor.

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or its representative, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

# 4. SELECTION AND WITHDRAWAL OF PATIENTS

#### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

# 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing at the Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

# 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study

conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9,

CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

Pregnancy reporting guidelines are provided in Section 9.5.2.

# 5. TREATMENT OF PATIENTS

# 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

# **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

# **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

# 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

# 6. STUDY DRUG MATERIALS AND MANAGEMENT

# 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

# **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

# 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

## 6.4. Administration

#### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

# **6.4.2.** Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every  $21 \pm 3$  days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done according to a site-specific plan by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A in an oral supplement.

# 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of

patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

# 6.5. Study Drug Accountability

The Investigator or designee will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

# 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

# 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

# 8. ASSESSMENT OF EFFICACY

# 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

# 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

# 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

# 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

# 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

# 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

### 8.1.4. Magnetic Resonance Neurography

Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity will be imaged for patients who have previously had MR neurography in the parent study and may be imaged for consenting patients who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

# 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

# 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

# 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

# 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

# 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

## 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

# 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

## **8.1.12.** Pharmacoeconomics Ouestionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

# 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

# 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

## **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

#### 8.1.16. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A supplementation.

## 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1. Samples may be analyzed, if clinically indicated.

## 9. ASSESSMENT OF SAFETY

# 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

# 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

# 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

## 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

## 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

## 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.
In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

## 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

## 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

## **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

#### 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

## 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

## 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

## 9.2. Adverse Events and Serious Adverse Events

#### 9.2.1. Definition of Adverse Events

#### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

#### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity

- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

## 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs,

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

# 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).

In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

## 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

### 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

- Patient's study number
- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the

completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or e-mail. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

### 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

### 10. STATISTICS

## 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

## 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

### 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### 10.2.2. Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

## 10.2.3. Efficacy Analyses

Efficacy analyses will examine between- and within-patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post-administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean (±SE) values over time for each location (hip, knee, etc.).

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

## 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

The observed values and changes from baseline in healthcare utilization will be evaluated and summarized using descriptive statistics.

#### 10.2.6. Interim Analysis

There is no formal interim analysis planned for this study. Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

## 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

## 11.2. Audits and Inspections

The Investigator will permit trial-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

## 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

## 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

## 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Health Organization (WHO) Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA), and all other applicable medical privacy laws and regulations.

## 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

### 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

## 14. DATA HANDLING AND RECORD KEEPING

## 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

## 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

## 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

## 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

## 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| necucu. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

## **Appendix 2: New York Heart Association Classification of Heart Failure**

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

### **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

## **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Sensation (32) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies ∑5 (18.6) <sup>a</sup> |
| | | <ul> <li>Sural SNAP, tibial motor n. distal latency, peroneal<br/>SNAP/motor n. conduction velocity/motor n. distal<br/>latency</li> </ul> |
| | | Vibration detection threshold (3.7) |
| | | • Heart rate response to deep breathing (3.7) |
| Modified NIS+7 | 304 | Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS <sup>a</sup> ) |
| | | • Weakness (192) |
| | | • Reflexes (20) |
| | | • Nerve conduction studies $\sum 5 (10)^a$ |
| | | <ul> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP,<br/>peroneal CMAP</li> </ul> |
| | | • Quantitative sensory testing: QST-BSA <sub>TP+HP5</sub> (80) |
| | | Postural blood pressure (2) |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

## **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| Ι | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

## Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

#### ALN-TTR02-006 Protocol Amendment 2

Summary of Changes (dated 05 January 2017) compared to Protocol Version 2.1 Taiwan (dated 10 December 2015)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Protocol Amendment**

The primary purpose of this amendment is to add the Columbia-Suicide Severity Rating Scale (C-SSRS) to the study assessments, which was inadvertently left out of previous versions of the protocol. The inclusion of the C-SSRS addresses a regulatory requirement to prospectively assess suicidality in clinical trials involving all drugs for neurological indications. Overall, this amendment includes the following changes:

- The Columbia-Suicide Severity Rating Scale has been added as an assessment of suicidal ideation and behavior.
- Country-specific versions of the protocol have been integrated in order to increase consistency in the execution of the clinical study globally
- Electroretinograms are now recommended to be performed in the case of suspected retinal disease.
- The premedication regimen has been updated to align with commercially available doses.
- Blood samples for long-term storage have been added in order to permit future exploratory investigations.
- During scheduled phone contact, clinical sites may now ask patients who are receiving home infusions about their general experience receiving these infusions

A detailed summary of the above changes, in addition to changes made for clarity, is provided in Table 1. Corrections to abbreviations, typographical errors and formatting are not detailed.

### Table 1: Protocol Amendment 2 Detailed Summary of Changes

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by bold font.

Purpose: Added Columbia-Suicide Severity Rating Scale to the study assessments

The primary change occurs in Table 1 Schedule of Assessments

Added text: Added row to Schedule of Assessments indicating that the Columbia-Suicide Severity Rating Scale is to be

collected at 26 weeks and 52 weeks after baseline and annually thereafter, as well as at the End of Study and Early

Withdrawal visits.

Section(s) also containing this change or similar changes:

Synopsis, Criteria for Evaluation, Safety

• Section 9.1.7 Columbia-Suicide Severity Rating Scale (section added)

Purpose: As part of global protocol integration, specified that home infusions are allowed only where applicable country and local regulations allow.

The primary change occurs in Section 3.1 Overall Study Design

Added text: After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every  $21 \pm 3$  days, or.

Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a

healthcare professional trained on the protocol and delivery of premedications and patisiran.

Section(s) also containing this change or similar changes:

- Synopsis, Methodology
- Table 1, Schedule of Assessments
- Section 5.3 Treatment Compliance
- Section 6.4.2 Study Drug Administration

Purpose: As part of global protocol integration, specified that MR neurography is only to be conducted in Germany and France

The primary change occurs in Table 1 Schedule of Assessments, footnote s

Now reads: Required only forMR neurography will only be conducted at sites in Germany and France. In these countries,

neurography may be conducted for patients who had MR neurography in the parent study and may be imaged for consenting for a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Patients who had imaging in the parent study should have Day 0 imaging if they did not

 $undergo\ MR\ neurography\ within\ the\ past\ 3\ months.$ 

Section(s) also containing this change or similar changes:

- Synopsis, Criteria for evaluation, Efficacy
- Section 8.1 Efficacy Parameters
- Section 8.1.4 Magnetic Resonance Neurography (Germany and France Only) (Section has been added)

Purpose: As part of global protocol integration, specified which studies patients may roll in from, and that the ALN-TTR02-003 study is not being conducted in Japan.

The primary change occurs in Section 3.1 Overall Study Design

Added text: Patients in this study will have completed "parent" study ALN-TTR02-003 or ALN-TTR02-004. Note that Study ALN-TTR02-003 is not being conducted in Japan.

Purpose: As part of global protocol integration, added Japan-specific recommendations regarding contraception.

The primary change occurs in Section 4.4 Pregnancy and Breastfeeding Restrictions / Contraception Requirements

Added text: In Japan it is recommended that the Investigators select appropriate contraception methods, as available.

Purpose: As part of global protocol integration, added Japan-specific instructions regarding duties related to study drug accountability.

The primary change occurs in Section 6.5 Study Drug Accountability

Added text: The Investigator or designee (or in Japan, the responsible pharmacist designated according to the Japan local

regulations) will maintain accurate records of receipt and the condition of the patisiran supplied for this study,

including dates of receipt.

Purpose: As part of global protocol integration, added statement on compensation for health damages as per local regulations.

The primary change occurs in Section 13.4 Compensation for Health Damages (section added)

Added text:

## 13.4 Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required per local regulations

Purpose: To update premedication regimen so that it aligns with commercially available doses.

The primary change occurs in Section 6.4.1 Premedication

Now reads: Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site).

Hydroxyzine or fexofenadine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg

PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Section(s) also containing this change or similar changes:

• Synopsis, Investigational product, dosage and mode of administration

Purpose: Added recommendation to collect an electroretinogram in the case of suspected retinal injury

The primary change occurs in Section 9.1.6 Ophthalmology Examination

Added text:

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Updated description of statistical analysis to align with currently planned analytic approach.

The primary change occurs in Section 10.2.3 Efficacy Analyses

Now reads:

Efficacy analyses will examine between and within patient rates of change over time. For the subset of patients that have previously received placebo in the parent study, comparisons for the various efficacy assessments will be made between rates of change pre- and post administration of patisiran, and relative to the treatment group in the parent study. Additional analyses will compare rates of change with rates estimated from previous studies, including cross-sectional, natural history, and interventional studies of other drugs. Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma 5$  NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also. Values of the individual components of the mNIS weakness and reflex scores will be depicted graphically by presenting the mean ( $\pm SE$ ) values over time for each location (hip, knee, etc.).

Section(s) also containing this change or similar changes:

- Synopsis, Statistical Methods
- Section 10.2.5 Healthcare Utilization Assessments
- Section 10.2.6 Interim Analysis

Purpose: Added blood sampling for long-term storage in order to permit future exploratory investigations.

The primary change occurs in Table 1 Schedule of Assessments

Added text:

Added row to Schedule of Assessments indicating a blood sample for long-term storage is to be collected at each clinic visit.

Section(s) also containing this change or similar changes:

• Section 8.1.18 Blood Sample for Long-term Storage (section added)

Purpose: Added questionnaire regarding experience of home infusions to scheduled phone contact for home infusion patients.

The primary change occurs in Table 1 Schedule of Assessments, footnote x

Added text:

x. Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every  $30 \ (\pm 5)$  days for assessment of adverse events and concomitant medication use. **During phone contact, patients may also be asked additional questions about their general experience receiving infusions at home.** 

Purpose: Added a definition of "woman of child-bearing potential".

The primary change occurs in Section 4.4 Pregnancy and Breastfeeding Restrictions / Contraception Requirements

Added text:

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

Purpose: Clarified language on Vitamin A dosing and added Japan-specific instructions.

The primary change occurs in Section 5.2 Concomitant Medications

Now reads:

All patients will be asked to continue to take an oral daily supplement containing the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan, the clinical sites will provide patients with a prescription for vitamin A.

Section(s) also containing this change or similar changes:

- Section 6.4.2 Study Drug Administration
  - Section 8.1.16 Vitamin A

Purpose: Clarified procedures for efficacy assessments, adding the location at which to conduct assessments, and removing specified duration.

The primary change occurs in Section 8.1 Efficacy Parameters

Now reads: Efficacy assessments will occur for all patients at the 52-week visit, which will take place over 2 days at the CAS.

Purpose: Removed language indicating that anti-drug antibodies would only be analyzed if clinically indicated.

The primary change occurs in Section 8.1.17 Efficacy Parameters

Deleted text: Serum samples for anti-drug antibodies will be collected as specified in Table 1.—Samples may be analyzed, if

clinically indicated.

Section(s) also containing this change or similar changes:

• Table 1, Schedule of Assessments

Purpose: Clarified that no study procedures may occur until approval is granted by all appropriate parties.

The primary change occurs in Section 13.1 Ethics Review

Added text: The Investigator should not start any study procedure with the patient until documentation of the approval

by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator

and Alnylam Pharmaceuticals, Inc.

## PATISIRAN (ALN-TTR02)

### ALN-TTR02-006

A MULTICENTER, OPEN-LABEL, EXTENSION STUDY TO EVALUATE THE LONG-TERM SAFETY AND EFFICACY OF PATISIRAN IN PATIENTS WITH FAMILIAL AMYLOIDOTIC POLYNEUROPATHY WHO HAVE COMPLETED A PRIOR CLINICAL STUDY WITH **PATISIRAN** 


Version 3.1 – United Kingdom (Incorporating

country-specific request)

Protocol Date

11 May 2017

**IND Number:** 

117395

**EUDRACT Number** 

2014-003877-40

Sponsor:

Alnylam Pharmaceuticals, Inc

300 Third Street

Cambridge, MA 02142 USA

**Sponsor Contact:** 



The concepts and information contained in this document or generated during the study are considered proprietary and may not be disclosed in whole or in part without expressed written authorization of Alnylam Pharmaceuticals, Inc.

The study will be completed according to guidelines of Good Clinical Practice (GCP). Compliance with this practice provides public assurance that the rights, safety, and well-being of study patients are protected consistent with the principles that have their origin in the Declaration of Helsinki.

## **INVESTIGATOR'S AGREEMENT**

I have read the ALN-TTR02-006 protocol and agree to conduct the study as outlined. I agree to maintain the confidentiality of all information received or developed in connection with this protocol.

| Printed Name of Investigator |
|------------------------------|
| Signature of Investigator |
| Date |

## **Version History:**

|---|---|---|
| 1.0 (Original) | 06 November 2014 | Initial Release |
| 2.0 – Global | 08 September 2015 | Incorporating Global Amendment 1 |
| 2.1 – Japan | 14 October 2015 | Incorporating Japan-specific Amendment 1 |
| 2.1 – Taiwan | 10 December 2015 | Incorporating Taiwan-specific Amendment 1 |
| 2.1 – France/Germany | 17 December 2015 | Incorporating France/Germany-specific |
| | | Amendment 1 |
| 2.1 – Brazil | 16 September 2015 | Incorporating Brazil-specific Amendment 1 |
| 2.2 – Japan | 14 March 2016 | Incorporating Japan-specific Amendment 2 |
| 3.0 - Global | 05 January 2017 | Incorporating Global Amendment 2 (including |
| | | Japan-, Taiwan- and France/Germany-specific |
| | | changes) |
| 3.1 – Brazil | 20 January 2017 | Incorporating Global Amendment 2 (including |
| | | Japan-, Taiwan- and France/Germany-specific |
| | | changes) |
| 3.1 – Argentina | 20 January 2017 | Incorporating Global Amendment 2 (including |
| | | Japan-, Taiwan- and France/Germany-specific |
| | | changes) |
| 3.1 – United Kingdom | 11 May 2017 | Incorporating country-specific request |

#### **SYNOPSIS**

#### Name of Sponsor/Company:

Alnylam Pharmaceuticals, Inc

### **Name of Investigational Product:**

Patisiran

#### **Title of Study:**

A Multicenter, Open-Label, Extension Study to Evaluate the Long-term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy Who Have Completed a Prior Clinical Study with Patisiran

### **Study Centers:**

This study will be conducted at multiple sites worldwide that have enrolled patients in a previous patisiran study.

#### **Objectives:**

To assess the safety and efficacy of long-term dosing with patisiran in transthyretin-mediated amyloidosis (ATTR) patients with familial amyloidotic polyneuropathy (FAP).

## **Methodology:**

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran introvenously. (I

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran intravenously (IV) once every  $21 \text{ (\pm 3)}$  days for the duration of the study. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) in this study 3 weeks after their last dose visit in the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

After the Day 0 visit, patients should return to the site for patisiran dosing once every 21 days. Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm 5$ ) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be done at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can also dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments after the 52-week visit may be done at a PCS.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may

occur if deemed necessary by the study personnel.

### Number of patients (planned):

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## Diagnosis and eligibility criteria:

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin ≤2 x ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study
- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

#### Investigational product, dosage and mode of administration:

Patisiran (comprising a small interfering ribonucleic acid [siRNA] targeting mutant and wild type transthyretin [TTR] messenger RNA [mRNA], in a lipid nanoparticle formulation for IV administration), 0.3 mg/kg once every 21 (±3) days administered as an IV infusion over 70 minutes (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion) by a controlled infusion device.

Patients will receive the following premedications at least 60 minutes before the start of the patisiran infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the study site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

#### **Duration of treatment:**

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

### Reference therapy, dosage and mode of administration:

Not applicable.

#### **Criteria for evaluation:**

### **Efficacy:**

The efficacy of patisiran will be assessed by the following evaluations:

- Neurological impairment assessed using the Neuropathy Impairment Score (NIS), Modified NIS (mNIS +7) composite score, and NIS+7
- Patient-reported quality of life (QOL) using the Norfolk Quality of Life-Diabetic Neuropathy (QOL-DN) and the EuroQOL (EQ-5D) questionnaires
- Disability reported by patients using the Rasch-built Overall Disability Scale (R-ODS)
- Autonomic symptoms assessed using the Composite Autonomic Symptom Score (COMPASS 31)
- Motor function assessments, including NIS-Weakness (NIS-W), timed 10-meter walk test, and grip strength test
- Polyneuropathy disability (PND) score and FAP stage
- Nutritional status using modified body mass index (mBMI)
- Pathologic evaluation of sensory and autonomic innervation evaluated by intraepidermal nerve fiber density (IENFD) analysis and quantitation of dermal sweat gland nerve fibers (SGNFD) via tandem 3 mm skin punch biopsies taken from the leg (only for patients having this assessment in the parent study)
- Magnetic resonance (MR) neurography (as regionally applicable)
- Cardiac structure and function through echocardiograms and serum levels of terminal

prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I

- New York Heart Association (NYHA) classification of heart failure
- Serum TTR
- Vitamin A
- Thyroid stimulating hormone
- Disease burden and healthcare utilization assessed using a patient-reported pharmacoeconomics questionnaire

#### Safety:

Safety assessments will include monitoring for AEs (including serious AEs [SAEs]); clinical laboratory tests, including hematology, clinical chemistry, urinalysis, and pregnancy testing; measurement of antidrug antibodies (if clinically indicated); vital signs; physical examinations; ophthalmology examinations; and assessment of suicidal ideation and behavior.

#### **Statistical methods:**

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

Associations between pharmacodynamic and efficacy data will be explored via correlation.

Descriptive statistics will be provided for clinical efficacy data, clinical laboratory data, vital signs data, and ECG interval data, presented as both actual values and changes from baseline relative to each on-study evaluation. Laboratory shift tables from baseline to worst values will be presented.

 Table 1
 Schedule of Assessments

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Windov | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Informed Consent | X | | | | | | |
| Inclusion/Exclusion Criteria | X | | | | | | |
| Medical History | X <sup>b</sup> | | | | | | |
| Demographics | X <sup>c</sup> | | | | | | |
| Physical Examination | X <sup>d</sup> | | | X | X | X° | X° |
| Weight | | Prior 1 | X<br>to Each Dose | | | X° | X° |
| mBMI <sup>e</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Height | X <sup>c</sup> | | | | | | |
| FAP Stage and PND Score | $X^d$ | | | X | X | X° | X° |
| Karnofsky Performance Status | X | | | | | | |
| NYHA Classification | X | | | X | | | $[X]^f$ |
| Vital Signs <sup>g</sup> | | X<br>Prior to Each Dose | | | | | |
| Safety Laboratory Assessments <sup>h</sup> | X <sup>d</sup> | X | X | X | X | X | X |
| INR | X | | | | | | |
| Pregnancy Test (urine) | X <sup>i</sup> | | X | X | X | X | X |
| C-SSRS Questionnaire | | | X | X | X | X | X |

| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| TTR Protein (ELISA) | X <sup>d</sup> | | X | X | X | X | X |
| TSH and Vitamin A | | | | X | X | X° | X° |
| Blood Sample for Long-term Storage | X | X | X | X | X | X | X |
| mNIS+7 <sup>j</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS+7 <sup>k</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| NIS only | | | | | $X^{l}$ | X <sup>m</sup> | X <sup>m</sup> |
| Grip Strength Test <sup>n</sup> | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| 10-Meter Walk Test <sup>p</sup> | X <sup>d</sup> | | | X | | | $[X]^f$ |
| Ophthalmology Examination <sup>q</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| Skin Punch Biopsy (IENFD and SGNFD) <sup>r</sup> | | | | X | X | Xº | X° |
| MR Neurography <sup>s</sup> (Germany & France only) | X | | X | X | X | X° | X° |
| Pharmacoeconomics Questionnaire | X | | | X | X | X° | X° |
| Norfolk QOL-DN <sup>t</sup> | X <sup>d</sup> | | | X | X | X° | X° |
| COMPASS 31 Questionnaire | X <sup>d</sup> | | | X | | | $[X]^{f}$ |
| R-ODS Disability | X <sup>d</sup> | | | X | | | $[X]^f$ |
| EQ-5D QOL | X <sup>d</sup> | | | X | X | X° | X° |
| Echocardiogram | $X^{d,u}$ | | | X | | | $[X]^f$ |
| Troponin I and NT-proBNP | $X^{d}$ | | | X | | | $[X]^f$ |
| Anti-Drug Antibody Testing <sup>v</sup> | | | X | X | X | X | X |
| | Day 0 Visit | 12 Week<br>Visit | 26 Week<br>Visit | 52 Week<br>Visit | Annual<br>Visit | End of<br>Study | Early<br>Withdrawal<br>Visit |
|---|---|---|---|---|---|---|---|
| Window | ≤45 Days from<br>Last Dose <sup>a</sup> | ±4 Weeks | ±4 Weeks | ±4<br>Weeks | ±6<br>Weeks | 4 (+1)<br>Weeks<br>from<br>Last<br>Dose | 4 (+1)<br>Weeks<br>from Last<br>Dose |
| Procedure | | | | | | | |
| Premedication / Patisiran Administration <sup>w</sup> | X | | X | | | | |
| Phone Contact <sup>x</sup> (In applicable regions only) | X | | | | | | |
| Adverse Events | X <sup>b</sup> Continuous Monitoring | | | | | | |
| Concomitant Medications | X <sup>b</sup> Continuous Monitoring | | | | | | |

#### **Table 1 Footnotes:**

Abbreviations: C-SSRS = Columbia-Suicide Severity Rating Scale; COMPASS 31 = Composite Autonomic Symptom Score; ELISA = enzyme linked immunosorbent assay; EQ-5D QOL = EuroQOL; FAP = familial amyloidotic polyneuropathy; IENFD = intraepidermal nerve fiber density; mBMI = modified body mass index; mNIS = Modified Neuropathy Impairment Score; MR = magnetic resonance; NIS = Neuropathy Impairment Score; NT-proBNP = N-terminal prohormone of B-type natriuretic peptide; NYHA = New York Heart Association; PND = polyneuropathy disability; QOL-DN = Quality of Life-Diabetic Neuropathy; R-ODS = Rasch-built Overall Disability Scale; SGNFD = sweat gland nerve fiber density; TSH = thyroid stimulating hormone; TTR = transthyretin

- a. Every effort should be made to perform Day 0 visit 3 weeks (±3 days) from the last dose of study drug in the parent study. However, the Day 0 visit may occur within 45 days after the last dose in the parent study. Exceptions may be made for medical or regulatory considerations only after consultation with the Medical Monitor.
- b. Medical history includes TTR genotype. Ongoing AEs from the parent study will be captured as Medical History on the case report form (CRF). Similarly concomitant medications that continue from the parent study will be entered into the database.
- c. Assessment does not need to be repeated. Information will be obtained from parent study.
- d. Assessment/procedure does not need to be repeated if performed during the parent study within 45 days of first dose in this study.
- e. mBMI will be calculated within the clinical database; this calculation does not need to be performed at the study center.
- f. Assessment/procedure required only if patient withdraws before the 52-week visit.
- g. Vital signs include blood pressure, heart rate, body temperature, and respiratory rate. Collected supine using an automated instrument after patient rests for 10 minutes. Must be performed pre-dose.
- h. Includes serum chemistry, hematology, and urinalysis. Refer to Section 9.1.5 for specific laboratory assessments.
- i. Assessment does not need to be repeated if the patient had a negative pregnancy test (urine or serum) within 14 days of the first dose.

- j. The mNIS+7 consists of the modified NIS tool (weakness and reflexes), nerve conduction studies (NCS) 5 attributes (Σ5), quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP), and postural blood pressure. Two assessments of the mNIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- k. The NIS+7 consists of the NIS tool (weakness, sensation, and reflexes), NCS Σ5, vibration detection threshold (VDT), and heart rate response to deep breathing (HRdB). Two assessments of the NIS+7 will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled.
- 1. One assessment of the NIS will be performed at each specified visit and must be performed by a neurologist.
- m. Assessment of NIS only does not need to be repeated if done as part of the NIS+7 at the End of Study or Early Withdrawal visit or if done within the previous 26 weeks.
- n. Grip strength will be measured in triplicate using a dynamometer held in the dominant hand. Every effort will be made to use the same device for a patient throughout the duration of the study. Two assessments of the grip strength will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) after the first assessment, but not more than 7 days apart.
- o. Assessment does not need to be repeated if done within the previous 26 weeks.
- p. The patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded. Two assessments of the 10-meter walk test will be performed on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.
- q. Examination will include visual acuity, visual fields, and slit-lamp evaluation. An electroretinogram may also be performed, as described in Section 9.1.6
- r. Optional skin biopsies will only be obtained if the patient had skin biopsies in the parent study and has provided separate informed consent for the skin biopsies in this study. Each skin biopsy assessment will include 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total), including 1 set of biopsies taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.
- s. MR neurography will only be conducted at sites in Germany and France. In these countries, neurography may be conducted for patients who had MR neurography in the parent study and for a subset of patients providing informed consent who did not have MR neurography previously in their parent study. Patients who had imaging in the parent study should have Day 0 imaging if they did not undergo MR neurography within the past 3 months.
- t. Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) do not have to complete this assessment.
- u. Patients entering this study from study ALN-TTR02-003, who were not previously participating in the cardiac subgroup, will be required to have an echocardiogram before dosing on Day 0.
- v. Serum samples for anti-drug antibodies will be collected as specified.
- w. Patisiran will be administered once every 21 (±3) days. Every effort should be made to continue dosing from the parent study in the 21 (±3) day timeframe. Doses may be administered at the clinical site or, where applicable country and local regulations allow, at home by a healthcare professional trained in the protocol.
- x. Patients who are receiving patisiran infusions at home must be contacted by the clinical site a minimum of every 30 (±5) days for assessment of adverse events and concomitant medication use. During phone contact, patients may also be asked additional questions about their general experience receiving infusions at home.

## **TABLE OF CONTENTS**

| SYNOP | SIS | 3 |
|---|---|---|
| TABLE | OF CONTENTS. | 11 |
| LIST O | F ABBREVIATIONS AND DEFINITIONS OF TERMS | 15 |
| 1. | INTRODUCTION | 18 |
| 1.1. | Disease Overview | 18 |
| 1.2. | Patisiran | 18 |
| 1.3. | Study Design Rationale | 19 |
| 1.4. | Risk-Benefit Assessment | 19 |
| 2. | STUDY OBJECTIVES | 22 |
| 3. | INVESTIGATIONAL PLAN | 23 |
| 3.1. | Overall Study Design | 23 |
| 3.2. | Number of Patients | 24 |
| 3.3. | Treatment Assignment | 24 |
| 3.4. | Criteria for Study Termination | 24 |
| 4. | SELECTION AND WITHDRAWAL OF PATIENTS | 25 |
| 4.1. | Patient Inclusion Criteria | 25 |
| 4.2. | Patient Exclusion Criteria | 25 |
| 4.3. | Patient Withdrawal Criteria | 26 |
| 4.4. | Pregnancy and Breastfeeding Restrictions / Contraception Requirements | 26 |
| 5. | TREATMENT OF PATIENTS | 29 |
| 5.1. | Description of Study Drug | 29 |
| 5.2. | Concomitant Medications | 29 |
| 5.3. | Treatment Compliance | 30 |
| 5.4. | Randomization and Blinding | 30 |
| 6. | STUDY DRUG MATERIALS AND MANAGEMENT | 31 |
| 6.1. | Study Drug Packaging and Labeling | 31 |
| 6.2. | Study Drug Storage | 31 |
| 6.3. | Study Drug Preparation | 31 |
| 6.4. | Administration | 32 |

| 6.4.1. | Premedication | 32 |
|---|---|---|
| 6.4.2. | Study Drug Administration | 33 |
| 6.4.3. | Suggested Guidelines for Management of Infusion-Related Reactions | 33 |
| 6.5. | Study Drug Accountability | 34 |
| 6.6. | Study Drug Handling and Disposal | 34 |
| 7. | PHARMACOKINETIC ASSESSMENTS | 35 |
| 8. | ASSESSMENT OF EFFICACY | 36 |
| 8.1. | Efficacy Parameters | 36 |
| 8.1.1. | Neurological Testing | 36 |
| 8.1.1.1. | Modified Neurological Impairment Score +7 and Neurological Impairment Score +7 | 36 |
| 8.1.1.2. | Neurological Impairment Score | 37 |
| 8.1.2. | Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score | 37 |
| 8.1.3. | Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density | 37 |
| 8.1.4. | Magnetic Resonance Neurography (Germany and France Only) | 37 |
| 8.1.5. | Modified Body Mass Index | 38 |
| 8.1.6. | Timed 10-meter Walk Test | 38 |
| 8.1.7. | Grip Strength Test | 38 |
| 8.1.8. | Composite Autonomic Symptom Score | 38 |
| 8.1.9. | Norfolk Quality of Life - Diabetic Neuropathy Questionnaire | 38 |
| 8.1.10. | EuroQoL Quality of Life Questionnaire | 38 |
| 8.1.11. | Rasch-built Overall Disability Scale | 39 |
| 8.1.12. | Pharmacoeconomics Questionnaire | 39 |
| 8.1.13. | Echocardiogram and Biomarkers of Cardiac Function | 39 |
| 8.1.14. | Transthyretin | |
| 8.1.15. | Thyroid-Stimulating Hormone | 39 |
| 8.1.16. | Vitamin A | 39 |
| 8.1.17. | Anti-Drug Antibodies | 39 |
| 8.1.18. | Blood Sample for Long-term Storage | 39 |
| 9. | ASSESSMENT OF SAFETY | |
| 9.1. | Safety Parameters | 41 |
| 9.1.1. | Demographic and Medical History | |

| 9.1.2. | Vital Signs | 41 |
|----------|-------------------------------------------|----|
| 9.1.3. | Weight and Height | 41 |
| 9.1.4. | Physical Examination | 41 |
| 9.1.5. | Laboratory Assessments | 41 |
| 9.1.5.1. | Hematology | 42 |
| 9.1.5.2. | Blood Chemistry | 42 |
| 9.1.5.3. | Urinalysis | 42 |
| 9.1.5.4. | Coagulation | 43 |
| 9.1.5.5. | Pregnancy Screen | 43 |
| 9.1.6. | Ophthalmology Examination | 43 |
| 9.1.7. | Columbia-Suicide Severity Rating Scale | 43 |
| 9.2. | Adverse Events and Serious Adverse Events | 43 |
| 9.2.1. | Definition of Adverse Events | 43 |
| 9.2.1.1. | Adverse Event | 43 |
| 9.2.1.2. | Serious Adverse Event | 44 |
| 9.3. | Relationship to Study Drug | 44 |
| 9.4. | Recording Adverse Events | 44 |
| 9.5. | Reporting Adverse Events | 45 |
| 9.5.1. | Serious Adverse Event Reporting | 45 |
| 9.5.2. | Pregnancy Reporting | 47 |
| 10. | STATISTICS | 48 |
| 10.1. | Sample Size | 48 |
| 10.2. | Statistical Methodology | 48 |
| 10.2.1. | Populations to be Analyzed | 48 |
| 10.2.2. | Baseline Evaluations | 48 |
| 10.2.3. | Efficacy Analyses | 48 |
| 10.2.4. | Safety Analyses | 49 |
| 10.2.5. | Healthcare Utilization Assessments | 49 |
| 10.2.6. | Interim Analysis | 49 |
| 11. | DIRECT ACCESS TO SOURCE DATA/DOCUMENTS | 50 |
| 11.1. | Study Monitoring | 50 |
| 11.2. | Audits and Inspections | 50 |

| 11.3. | Institutional Review Board | 50 |
|---------|----------------------------------------------|----|
| 12. | QUALITY CONTROL AND QUALITY ASSURANCE | 51 |
| 13. | ETHICS | |
| 13.1. | Ethics Review | 52 |
| 13.2. | Ethical Conduct of the Study | 52 |
| 13.2.1. | . Financial Disclosure Reporting Obligations | |
| 13.3. | Written Informed Consent | |
| 13.4. | Compensation for Health Damages | 53 |
| 14. | DATA HANDLING AND RECORD KEEPING | 54 |
| 14.1. | Case Report Forms | 54 |
| 14.2. | Confidentiality | 54 |
| 14.3. | Inspection of Records | 55 |
| 14.4. | Retention of Records | 55 |
| 15. | PUBLICATION POLICY | 56 |
| 16. | LIST OF REFERENCES | 57 |
| 17. | APPENDICES | 58 |
| | LIST OF TABLES | |
| Table 1 | Schedule of Assessments | |

## LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviation | Definition |
|--------------|-------------------------------------------------------------|
| AE | adverse event |
| ALT | alanine transaminase |
| AST | aspartate transaminase |
| ATTR | transthyretin-mediated amyloidosis |
| BUN | blood urea nitrogen |
| CAS | Central Assessment Sites |
| CFR | Code of Federal Regulations |
| COMPASS 31 | Composite Autonomic Symptom Score |
| CRF | case report form |
| CRO | clinical research organization |
| СҮР | cytochrome P450 |
| DLin-MC3-DMA | 1,2-Dilinoleyloxy-N,N-dimethylpropylamine |
| DN | diabetic neuropathy |
| DSPC | 1,2-Distearoyl-sn-glycero-3-phosphocholine |
| EDC | electronic data capture |
| ELISA | enzyme linked immunosorbent assay |
| EP | European Pharmacopoeia |
| EQ-5D | EuroQOL |
| EU | European Union |
| Σ5 | 5 attributes |
| FAC | familial amyloidotic cardiomyopathy |
| FAP | familial amyloidotic polyneuropathy |
| GCP | Good Clinical Practice |
| GMP | Good Manufacturing Practice |
| HEENT | head, ears, eyes, nose, and throat |
| HIPAA | Health Insurance Portability and Accountability Act of 1996 |
| HP | heat pain |
| HRdb | heart rate response to deep breathing |

| Abbreviation | Definition |
|--------------|-----------------------------------------------------|
| IB | Investigators Brochure |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | Independent Ethics Committee |
| IENFD | intraepidermal nerve fiber density |
| INN | International Nonproprietary Name |
| INR | international normalized ratio |
| IRB | Institutional Review Board |
| IRR | infusion-related reaction |
| IRS | interactive response system |
| IUD | intrauterine device |
| IUS | intrauterine system |
| IV | intravenous |
| LNP | lipid nanoparticle |
| mBMI | modified body mass index |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mNIS | Modified Neuropathy Impairment Score |
| mRNA | messenger RNA |
| MR | magnetic resonance |
| NCS | nerve conduction studies |
| NHP | non-human primate |
| NIS | Neuropathy Impairment Score |
| NIS-W | Neuropathy Impairment Score- Weakness |
| NSAID | nonsteroidal anti-inflammatory drug |
| NT-proBNP | N-terminal prohormone of B-type natriuretic peptide |
| NYHA | New York Heart Association |
| OTC | over-the-counter |
| PCS | Patient Care Sites |
| PD | pharmacodynamic |

| Abbreviation | Definition |
|---|---|
| PEG <sub>2000</sub> -C-DMG | (R)-methoxy-PEG <sub>2000</sub> -carbamoyl-di-O-myristyl-sn-glyceride |
| PK | pharmacokinetic |
| PND | polyneuropathy disability |
| PO | per os (orally) |
| QOL | quality of life |
| QOL-DN | Quality of Life-Diabetic Neuropathy |
| QST | quantitative sensory testing |
| RBC | red blood cell |
| RBP | retinol binding protein |
| RNAi | ribonucleic acid interference |
| R-ODS | Rasch-built Overall Disability Scale |
| SAE | serious adverse event |
| SGNFD | sweat gland nerve fiber density |
| siRNA | small interfering ribonucleic acid |
| SUSAR | Suspected Unexpected Serious Adverse Reaction |
| TP | touch pressure |
| TSH | thyroid stimulating hormone |
| TTR | transthyretin |
| TUDCA | tauroursodeoxycholic acid |
| ULN | upper limit of normal |
| USP | United States Pharmacopeia |
| V30M | Val30Met |
| VDT | vibration detection threshold |
| WBC | white blood cell |
| WT | wild type |

### 1. INTRODUCTION

### 1.1. Disease Overview

Transthyretin-mediated amyloidosis (ATTR) is a hereditary, autosomal dominant, systemic disease caused by a mutation in the transthyretin (TTR) gene leading to the extracellular deposition of amyloid fibrils containing both mutant and wild type (WT) TTR. The particular TTR mutation and site of amyloid deposition determines the clinical manifestations of the disease, which include sensory and motor neuropathy, autonomic neuropathy, and/or cardiomyopathy. ATTR is a progressive disease associated with severe morbidity, with a life expectancy limited to 5 to 15 years from symptom onset. There are over 100 reported TTR mutations which are associated with 2 clinical syndromes: familial amyloidotic polyneuropathy (FAP) and familial amyloidotic cardiomyopathy (FAC). The estimated worldwide prevalence of FAP is 5,000 to 10,000, with the majority of cases in Portugal, Sweden, France, Japan, Brazil, and the United States. The most common causative mutation of FAP is TTR Val30Met (V30M), with the onset of symptoms typically occurring between 30 and 55 years of age.

Reduction of circulating amyloidogenic TTR improves outcomes in patients with FAP. Orthotopic liver transplantation, which eliminates mutant TTR from the circulation, has improved survival in early stage FAP patients. The TTR tetramer stabilizer tafamidis (Vyndaqel®) was approved in the European Union (EU) for the treatment of stage 1 FAP based on evidence that it may slow neuropathy progression in these patients, but has not been approved for use in other regions of the world. Diflunisal, a generic, nonsteroidal anti-inflammatory drug (NSAID) that is also a tetramer stabilizer, exhibits slowing of neuropathy progression in FAP patients, but is not standardly used among practitioners. Thus, there remains an unmet medical need for a potent and effective therapy for FAP that will have an impact on patients across a broad range of neurologic impairment, regardless of their mutation.

### 1.2. Patisiran

Patisiran (the International Nonproprietary Name [INN] name for the drug product also referred to as ALN-TTR02) is a novel investigational agent being developed for the treatment of ATTR patients with symptomatic FAP. Patisiran comprises a small interfering ribonucleic acid (siRNA) which is specific for TTR, and is formulated in a hepatotropic lipid nanoparticle (LNP) for intravenous (IV) administration. <sup>11</sup> It is designed to significantly suppress liver production of both WT and all mutant forms of TTR, thereby having the potential to reduce amyloid formation and provide clinical benefit to patients with FAP.

The nonclinical pharmacology, pharmacokinetics (PK), and toxicology of patisiran were evaluated in a series of in vitro and in vivo studies that have enabled chronic dosing in clinical studies. A summary of the nonclinical data can be found in the patisiran Investigators Brochure (IB).

In a Phase 1 study of patisiran in healthy volunteers (Study ALN-TTR02-001), patisiran was generally well tolerated. Significant pharmacology in terms of TTR protein lowering (>80% reduction from pretreatment baseline) was observed at doses ≥0.15 mg/kg. TTR levels showed evidence of recovery at Day 28 and return to baseline by Day 70. A Phase 1 study in healthy

subjects of Japanese origin (Study ALN-TTR02-005) also showed dose dependent reduction in serum TTR, similar to that observed in Study ALN-TTR02-001 in Caucasian subjects; patisiran was safe and well tolerated up to 0.3 mg/kg. An open-label Phase 2 multiple ascending dose study of patisiran in ATTR patients with FAP (Study ALN-TTR02-002) was conducted to determine the safety and tolerability, PK, and pharmacodynamics (PD) of a 60 or 70 minute IV infusion of patisiran administered once every 3 or 4 weeks for 2 doses. The top dose of 0.3 mg/kg administered every 3 or 4 weeks was found to be generally safe and well tolerated. with maximum TTR knockdown of ~90% and sustained TTR suppression of >80% most consistently observed with every 3 week dosing. Twenty seven of the 29 patients treated on the Phase 2 trial enrolled in an open-label extension study (ALN-TTR02-003) to evaluate safety and tolerability of long-term dosing with patisiran for approximately 2 years. Multiple doses of patisiran have been generally safe and well-tolerated on the -003 study, with preliminary data indicating no changes in liver function tests, renal function, or hematologic parameters, and no treatment-related discontinuations. Sustained suppression of serum TTR of >80% has been observed in the open-label extension study, and preliminary clinical data at 6 months showed evidence for disease stabilization. <sup>12</sup> A randomized, double-blind, placebo-controlled Phase 3 study of patisiran (ALN-TTR02-004; APOLLO) is ongoing worldwide. The main objectives of the study are to demonstrate the clinical efficacy of patisiran and to establish the safety of chronic dosing in ATTR patients with FAP. Further details on the clinical studies of patisiran can be found in the patisiran Investigator's Brochure.

## 1.3. Study Design Rationale

This is a multicenter, open-label extension study designed to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have completed a prior study with patisiran.

The nonclinical data and clinical experience with patisiran support the continuation of patisiran treatment in this long-term extension study for ATTR patients with FAP. All patients will receive patisiran at 0.3 mg/kg administered IV every 3 weeks, which is the dose and regimen employed in the ongoing Phase 3 study with patisiran. Various clinical evaluations will be performed periodically as outlined in Table 1 to continue to assess the effect of patisiran beyond the duration of the ongoing clinical studies, and will enable all patients who have completed a prior study with patisiran (provided they meet the eligibility criteria of this study), including those previously on placebo, to receive open-label patisiran. Patients coming on to this open-label study from a blinded study will remain blinded to their previous treatment assignment until at least database lock has occurred in that study. The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

### 1.4. Risk-Benefit Assessment

Patisiran is a novel investigational agent intended for the treatment of FAP, a serious and lifethreatening orphan disease with limited treatment options. The therapeutic hypothesis that systemic amyloidoses can be managed by reducing circulating levels of amyloidogenic protein has been established in other acquired and hereditary amyloidoses. The experience from these systemic amyloidotic disorders, as well as the liver transplant data in FAP, suggest that lowering of the circulating amyloidogenic protein could impact the clinical course of the disease. Based on nonclinical and clinical data that showed suppression in levels of WT and mutant TTR upon administration of 0.3 mg/kg patisiran once every 21 days, it is possible that long term treatment with patisiran may have a clinical benefit in FAP patients with mild to moderate polyneuropathy and that further study is warranted.

In completed and ongoing clinical studies (ALN-TTR02-001, ALN-TTR02-002 and ALN-TTR02-003), single and multiple doses of patisiran have been generally well tolerated. Potential risks of patisiran include the following:

### • Infusion-Related Reactions

Infusion-related reactions (IRRs) can occur with systemic administration of certain biological agents such as liposomes or monoclonal antibodies. In order to reduce the potential for an IRR with patisiran, all patients in this study will be premedicated prior to dosing with patisiran. The step-wise infusion regimen over approximately 70 minutes (starting with a slower infusion rate of approximately 1 mL/minute for the first 15 minutes before increasing to 3 mL/minute for the remainder of the infusion), may further reduce the risk of an IRR.

### • Liver function test abnormalities

In preclinical studies, patisiran-related increased serum liver markers and histopathology in the liver were observed at dosages > 0.1 mg/kg in rats and > 1.0 mg/kg in monkeys. In general, all of the findings were not observed or were observed at lower severity at the end of the 60-90 day dose free period, indicating that the toxicities were reversible. In clinical studies to date, there have been no clinically significant changes in liver function tests in either the single-dose or multiple-dose studies. Patients in the study are monitored for liver function via serial laboratory assessments.

### • Vitamin A Lowering

The suppression of serum levels of TTR and retinol binding protein (RBP) is expected to result in the lowering of circulating vitamin A levels. Preclinical and clinical data have shown that the lowering of circulating vitamin A associated with suppression of RBP does not result in severe vitamin A deficiency. Furthermore, there are individuals with RBP/TTR mutations who have life-long low levels of circulating vitamin A and are essentially in good health, suggesting that there are compensatory transport mechanisms for vitamin A that are yet undescribed. This has also been confirmed in TTR knockout mice, which do not exhibit any manifestations of vitamin A deficiency, with vitamin A uptake by most tissues continuing in the absence of RBP. Provided there is adequate vitamin A in the diet, tissue stores of vitamin A should not be affected by the lowering of TTR and RBP. However, as the vitamin A content of the diet may vary between different countries and different individuals within a country, all patients on the study will be asked to take a daily supplement containing the recommended daily allowance of vitamin A. Patients should have started vitamin A supplementation by the time they start his/her first dose of patisiran.

### Osteoporosis

Patients with FAP may be at risk for osteoporosis. <sup>15</sup> In addition, as part of the premedication regimen administered prior to patisiran dosing every three weeks, FAP patients participating in this study are given glucocorticoids, a drug known to have the potential to reduce bone

mineralization. If there are no medical contraindications, and per investigator judgment and local standard of care, study participants should, if appropriate, receive therapy for the prevention and early treatment of osteoporosis such as: calcium and vitamin D supplementation, bisphosphonates, calcitonin, parathyroid hormone, estrogen agonist/antagonist or combination therapies.

Further guidance to the investigator can be found in the Investigator's Brochure.

## 2. STUDY OBJECTIVES

The objective of this study is to assess the safety and efficacy of long-term dosing with patisiran in ATTR patients with FAP.

### 3. INVESTIGATIONAL PLAN

## 3.1. Overall Study Design

This is a multicenter, multinational, open-label extension study to evaluate the long-term safety and efficacy of patisiran in patients with FAP who have previously completed a patisiran study. Patients in this study will have completed "parent" study ALN-TTR02-003 or ALN-TTR02-004. Note that Study ALN-TTR02-003 is not being conducted in Japan.

Consented eligible patients will enroll in this study and receive 0.3 mg/kg patisiran IV once every 21 days for the duration of the study. All dosing visits have a window of  $\pm 3$  days. In order to maintain the every 21-day dosing schedule from the parent study, patients are expected to have their first visit (Day 0) on this study 3 weeks after their last dose visit on the parent study. However, if necessary, a patient may initiate dosing in this study up to 45 days from the time of the last dose in the parent study. Exceptions to this timing may be allowed for medical or regulatory considerations only after consultation with the Medical Monitor. The last testing visit in the parent study will serve as the baseline for this study, unless more than 45 days have elapsed, in which case the baseline tests will need to be repeated on Day 0. Eligibility for this study will be confirmed before administration of the first dose on Day 0.

The duration of the study has been determined to allow the collection of long-term safety, tolerability and efficacy data of patisiran in patients with FAP who have completed a prior study with patisiran. The estimated duration of the study is 5 years.

In order to reduce the potential for an IRR with patisiran, all patients on this study will receive premedications at least 60 minutes before the start of the patisiran infusion. Patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15-minutes followed by approximately 3 mL/minute for the remainder of the infusion). If the infusion duration for a patient was lengthened beyond 70 minutes due to the occurrence of an IRR while on the parent study, that infusion duration may be continued on this study for that particular patient. Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor.

After the Day 0 visit, patients should return to the clinical site for patisiran dosing once every 21 ( $\pm 3$ ) days. Where applicable country and local regulations allow, patients may receive the patisiran infusions at home by a healthcare professional trained on the protocol and delivery of premedications and patisiran. Patients who are receiving patisiran infusions at home will have a phone contact with the site at least every 30 ( $\pm 5$ ) days. Patients will also have visits at the clinical site at approximately 12, 26 and 52 weeks, and yearly thereafter.

A complete set of efficacy assessments will be performed at 52 weeks, followed by more limited efficacy assessments yearly thereafter. In order to decrease the variability in the efficacy assessment testing at the 52-week visit, there will be a limited number of sites within any one territory that conduct these efficacy assessments (referred to as "Central Assessment Sites [CAS]"); these sites can dose and manage patients. There will also be sites that can dose and manage the patients ("Patient Care Sites [PCS])", while sending the patients to the nearest CAS for their 52-week efficacy assessments. Every effort should be made for the patient to return to the same CAS center that the patient went to in the parent study. Yearly efficacy assessments

after the 52-week visit may be done at a PCS. Prior to starting the study, the CAS and PCS will create a delegation of responsibilities document that clearly details which site is responsible for which efficacy tests and safety parameters to ensure adherence to the protocol. This document will become part of the study site specific documentation.

Safety will be assessed throughout the study. Patients will return to the clinical site for safety evaluations at 12, 26 and 52 weeks during the first year and yearly thereafter. Patients will be continually assessed throughout the study for adverse events (AEs). Unscheduled visits for study assessments may occur if deemed necessary by the study personnel.

### 3.2. Number of Patients

All patients who have previously completed a patisiran study may be enrolled if they meet the eligibility criteria for this study.

## 3.3. Treatment Assignment

All patients enrolled in this study will receive open-label patisiran at 0.3 mg/kg administered IV once every 21 (±3) days.

The Investigator or his/her delegate will contact the interactive response system (IRS) (via phone or web) after confirming that the patient fulfills all the inclusion criteria and none of the exclusion criteria. The patient will then be assigned a patient number that corresponds to their current patient number on the parent study. A combination of the center number, parent study number, enrollment number, and patient initials will create the unique patient identifier. In countries with regulations prohibiting the use of patient initials, a strategy consistent with local regulations will be used to generate replacement values for the patient initials.

## 3.4. Criteria for Study Termination

The study may be terminated if patisiran does not obtain marketing approval or the development of patisiran is no longer being pursued by the Sponsor (Alnylam Pharmaceuticals, Inc).

The Sponsor reserves the right to discontinue the study for clinical or administrative reasons at any time. Should the study be terminated and/or the site closed for whatever reason, all documentation and patisiran supplied for the study must be returned to the Sponsor or Medpace, and the Investigators, Independent Ethics Committee (IEC) / Institutional Review Board (IRB) and Regulatory Authorities will be promptly informed of the termination and the reason for the decision. The Investigator should promptly inform the patients and assure appropriate therapy and follow-up.

### 4. SELECTION AND WITHDRAWAL OF PATIENTS

### 4.1. Patient Inclusion Criteria

To be enrolled in the study, patients must meet the following criteria before administration of patisiran on Day 0:

- 1. Have completed a patisiran study (ie, completed the last efficacy visit in the parent study) and, in the opinion of the investigator, tolerated study drug
- 2. Be considered fit for the study by the Investigator
- 3. Have aspartate transaminase (AST) and alanine transaminase (ALT) levels  $\leq 2.5 \times$  the upper limit of normal (ULN), international normalized ratio (INR)  $\leq 2.0$  (patients on anticoagulant therapy with an INR of  $\leq 3.5$  will be allowed)
- 4. Have a total bilirubin within normal limits. A patient with total bilirubin  $\leq 2$  X ULN is eligible if the elevation is secondary to documented Gilbert's syndrome (elevation of unconjugated bilirubin with normal conjugated bilirubin) and the patient has ALT and AST levels within normal ranges.
- 5. Have a serum creatinine  $\leq 2 \times ULN$
- 6. Women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing in this study and agree to use 2 highly effective methods of contraception throughout study participation and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control are defined in Section 4.4.
- 7. Males with partners of child-bearing potential must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicide) of contraception throughout study participation and for 75 days after the last dose of patisiran in this study; males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study
- 8. Be willing and able to comply with the protocol-required visit schedule and visit requirements and provide written informed consent

### 4.2. Patient Exclusion Criteria

A patient will be excluded if they meet any of the following criteria before dosing on Day 0:

- 1. Has an active infection requiring systemic antiviral or antimicrobial therapy that will not be completed before the first dose of patisiran administration
- 2. Has poorly controlled diabetes mellitus
- 3. Has uncontrolled cardiac arrhythmia or unstable angina
- 4. Is currently taking tafamidis, diflunisal, doxycycline, or tauroursodeoxycholic acid (TUDCA), unless previously allowed per the parent study

- 5. Is unable to take the required premedications, unless modifications to the premedication regimen were previously allowed per the parent study
- 6. Is under legal protection (defined as "any person who becomes incapable of protecting his/her interests due to a medically diagnosed impairment of his/her mental faculties that may limit or prevent the expression of his will"), decided by a court

### 4.3. Patient Withdrawal Criteria

Patients are free to withdraw from the study at any time and for any reason, without penalty to their continuing medical care. For those patients who withdraw, every effort will be made to determine their reason for dropping out, and to complete the Early Withdrawal visit.

The Investigator may withdraw a patient from the study if the patient:

- Is in violation of the protocol
- Experiences a serious or intolerable AE
- Becomes pregnant
- Requires a prohibited medication (see Section 5.2)
- Requests to be withdrawn from the study
- Is found to be considerably noncompliant with the protocol-required patisiran dosing visits

The Investigator will withdraw patients from the study upon the request of the Sponsor, including if the Sponsor terminates the study. Upon occurrence of a serious or intolerable AE, the Investigator will confer with the Sponsor before discontinuing the patient.

Missing an occasional dose of patisiran will not necessarily result in the patient being withdrawn from the study. However, if a patient misses 3 consecutive doses of patisiran, the Investigator at the clinical site and the Medical Monitor will determine whether the patient should be withdrawn from the study. If the patient is withdrawn from the study, the reason will be noted in the patient medical record and on the case report form (CRF).

In the event a patient is withdrawn from the study, the clinical research organization (CRO) Medical Monitor must be informed immediately.

# 4.4. Pregnancy and Breastfeeding Restrictions / Contraception Requirements

TTR transports vitamin A in plasma; therefore, reductions in circulating vitamin A levels accompany reductions in TTR caused by patisiran. Vitamin A deficiency has known effects on both male and female reproductive performance and embryo/fetal development. It is not known whether decreased levels of vitamin A at efficacious patisiran doses in ATTR patients who are male or who are women of child bearing potential will affect reproduction. Histopathological evaluations of all of the reproductive organs have been conducted in the rat and non-human primate (NHP) toxicology studies including a chronic NHP study in sexually mature animals, where there were no adverse effects in males (including sperm analyses and spermatogenic staging) or females. In a dose range-finding rat embryo/fetal development study

conducted with patisiran, there were no effects on mating, fertility, ovarian or uterine parameters, or fetal development despite reductions (-88% from baseline) in serum vitamin A in the dams dosed with the rat-specific TTR surrogate siRNA.

Women of child-bearing potential are defined as any woman or adolescent who has begun menstruation. A post-menopausal woman is defined as a woman who has 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.

In this study, women of child-bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be using 2 highly effective methods of contraception prior to dosing on Day 0, throughout study participation, and for 75 days after last dose of patisiran in this study. Highly effective methods of birth control result in a low failure rate (ie, less than 1% per year). Acceptable forms of effective contraception are defined as follows:

- Hormonal: established use of oral, implantable, injectable, or transdermal hormonal methods of conception
- Placement of an intrauterine device (IUD)
- Placement of an intrauterine system (IUS)
- Mechanical/barrier method of contraception: condom or occlusive cap (diaphragm or cervical/vault cap) in conjunction with spermicide (foam, gel, film, cream or suppository)

Note: Failure rates indicate that, when used alone, the diaphragm and condom are not highly effective forms of contraception. Therefore the use of additional spermicides does confer additional theoretical contraceptive protection. However, spermicides alone are inefficient at preventing pregnancy when the whole ejaculate is spilled. Therefore, spermicides are not a barrier method of contraception and should not be used alone.

- Surgical sterilization of male partner (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate; for female patients on the study, the vasectomized male partner should be the sole partner for that patient);
- Sexual true abstinence: when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Patients should be instructed to use 2 different forms of effective contraception from the list above. Examples of 2 forms of highly effective contraception are as follows:

- Oral, implantable, injectable, or transdermal contraceptives in conjunction with condom or diaphragm and spermicide
- IUD in conjunction with condom or diaphragm and spermicide
- Surgical sterilization of partner in conjunction with condom or diaphragm and spermicide

Interaction between patisiran and hormonal contraceptives is not anticipated. The patisiran drug substance ALN-18328 (siRNA), and the 2 novel lipid excipients 1,2-Dilinoleyloxy-N,N-dimethylpropylamine (DLin-MC3-DMA) and (R)-methoxy-PEG<sub>2000</sub>-carbamoyl-di-O-myristyl-sn-glyceride (PEG-<sub>2000</sub>-C-DMG), were evaluated by in vitro human microsomal incubations to determine if any had inhibitory effects on cytochrome P450 (CYP) activity. None of the components displayed an inhibitory effect on any of the CYPs investigated (CYP1A2, CYP2C9, CYP2C19, CYP2D6 and CYP3A4/5). In addition, there was no induction of CYP1A2, CYP2B6, or CYP3A4 at any of the concentrations studied. These data suggest a low likelihood of patisiran to interfere with the metabolism of hormonal contraceptives.

Males (including men who have had vasectomies) with partners of child-bearing potential, must agree to use 1 barrier method (eg, condom) and 1 additional method (eg, spermicidal foam, gel, film, cream, or suppository) of contraception throughout study participation and for 75 days (ie, a whole spermatogenic cycle) after the last dose of patisiran in this study. Males must also abstain from sperm donation after the first dose of patisiran through study participation and for 75 days after last dose of patisiran in this study.

In Japan it is recommended that the Investigators select appropriate contraception methods, as available.

Pregnancy reporting guidelines are provided in Section 9.5.2.

### 5. TREATMENT OF PATIENTS

## 5.1. Description of Study Drug

Patisiran Solution for Injection is a ribonucleic acid interference (RNAi) therapeutic consisting of an siRNA targeting TTR messenger RNA (mRNA) formulated in a LNP. The patisiran drug product is a sterile formulation of ALN-18328, an siRNA targeting TTR, formulated as LNPs siRNA with lipid excipients (DLin-MC3-DMA, 1,2-Distearoyl-sn-glycero-3-phosphocholine [DSPC], cholesterol, and PEG<sub>2000</sub>-C-DMG in isotonic phosphate buffered saline. Patisiran Solution for Injection contains 2 mg/mL of the TTR siRNA drug substance.

### **5.2.** Concomitant Medications

Use of the following medications/treatments is prohibited during study participation:

- Any investigational agent other than patisiran
- Corticosteroids other than those administered as premedications prior to the dose of patisiran, those used to treat an infusion reaction, or topical or inhaled corticosteroids. However, for patients with chronic inflammatory disorders (eg, asthma, rheumatoid arthritis), systemically administered steroids may be permitted provided that: 1) the dose is <20 mg/day prednisone or equivalent if administered chronically, or 2) for doses ≥20 mg/day, administration is limited to no more than 5 consecutive days.

Use of the medications/treatments listed below is permitted in patients who were already taking such medications while on the parent study in accordance with the rules of that study protocol. For patients who did not take these medications while on the parent study, use of these medications is permitted, if necessary, only after the patient has completed the 52-week visit.

- Tafamidis
- Diflunisal
- Doxycycline/TUDCA

Medications and treatments other than those specified above, including palliative and supportive care approved by the Investigator for disease-related symptoms, are permitted during the study.

All patients will be asked to continue to take the recommended daily allowance of vitamin A. Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan, the clinical sites will provide patients with a prescription for vitamin A.

Any concomitant medication or treatment that is required for the patient's welfare may be given by the Investigator. Use of all concomitant medications and treatments will be recorded on the patient's CRF through the end of the patient's participation in the study. This will include all prescription drugs, herbal preparations, over-the-counter (OTC) medications, vitamins, and minerals. Any changes in medications during the study will also be recorded on the CRF. Similarly, concomitant medications that continue from the parent study will be entered into the database.

## **5.3.** Treatment Compliance

Compliance with patisiran administration is dependent on the proper preparation and administration of IV infusions by trained personnel and attendance by the patient at the clinic for scheduled assessment visits. Compliance with patisiran administration will be verified through observation by study staff or (in applicable regions) trained home healthcare professionals. A dose will be considered completed if 80% or more of the total volume of the IV solution was administered to the patient. Patients will be permitted to miss an occasional dose of patisiran; however, if a patient misses 3 consecutive doses, the Investigator, in consultation with the Medical Monitor, will discuss whether the patient will be able to continue on the study.

## 5.4. Randomization and Blinding

This is an open-label study; however, patients rolling over into this study from a previously blinded study will remain blind to their previous treatment assignment until database lock has occurred in that study.

### 6. STUDY DRUG MATERIALS AND MANAGEMENT

## 6.1. Study Drug Packaging and Labeling

All packaging, labeling, and the preparation of patisiran will be in compliance with Good Manufacturing Practice (GMP) specifications, as described in the Manufacture of Investigational Medicinal Products Volume 4 Annex 13, and any other or local applicable regulations.

Patisiran labels will include all appropriate local labeling requirements on the vial and external label. Sample labels will be submitted to health authorities, per local country submission requirements.

The patisiran drug product is packaged in 10 mL glass vials with a fill volume of 5.5 mL. The container closure system consists of a United States Pharmacopeia/European Pharmacopoeia (USP/EP) Type I borosilicate glass vial, a Teflon-faced butyl rubber stopper, and an aluminium flip-off cap.

## **6.2.** Study Drug Storage

Patisiran will be stored upright and refrigerated at approximately  $5 \pm 3$  °C. Any deviation from the recommended storage conditions must be reported to the CRO and/or the Sponsor and use of the patisiran halted until authorization for its continued use has been given by the Sponsor or designee.

No special procedures for the safe handling of patisiran are required. A Sponsor representative or designee will be permitted, upon request, to audit the supplies, storage, dispensing procedures, and records.

Patisiran supplied for this study may not be administered to any person not enrolled in the study.

## 6.3. Study Drug Preparation

Staff at each clinical site or the healthcare professional administering patisiran will be responsible for preparation of patisiran doses, according to procedures detailed in the Pharmacy Manual.

All patients in this study will receive 0.3 mg/kg patisiran once every 21 days ( $\pm 3 \text{ days}$ ). The amount (mg) of patisiran to be administered will be based on the patient's body weight (kg). For each dose administered, the weight obtained during the previous dosing visit will be used to calculate the dose of patisiran. In the event that the weight obtained on the previous dosing day is not available, the weight obtained pre-dose on the current dosing day can be used for dose calculation. Patients who weigh 105 kg or more will receive patisiran dosing based on an assumption of a body weight of 104 kg.

Patisiran will be prepared under aseptic conditions. The total amount to be infused into each patient at each dosing visit will be 200 mL. Sterile normal saline (0.9% NaCl) will be added to a sterile infusion bag, and the calculated volume of patisiran will be withdrawn from the vials and injected into the infusion bag.

### 6.4. Administration

### 6.4.1. Premedication

Prior to each dose of patisiran, patients will receive the following premedications in order to reduce the risk of experiencing an IRR at least 60 minutes before the infusion:

- Intravenous dexamethasone (10 mg) or equivalent
- Oral paracetamol/acetaminophen (500 mg) or equivalent
- Intravenous H2 blocker (ranitidine 50 mg, famotidine 20 mg, or equivalent other H2 blocker dose)
- Intravenous H1 blocker: diphenhydramine 50 mg (or equivalent other IV H1 blocker available at the clinical site). Hydroxyzine 25 mg per os (PO, orally) or fexofenadine 30 mg or 60 mg PO or cetirizine 10 mg PO may be substituted for any patient who does not tolerate IV diphenhydramine or other IV H1 blocker.

Further details (including a table of equivalent premedications) can be found in the patisiran Pharmacy Manual.

Patients will be started on the above premedication regimen. However, modifications may be made to the premedication regimen after consultation with the medical monitor either due to a patient's inability to tolerate one or more of the premedications or to the occurrence of IRRs unresponsive to slowing of the infusion rate.

- If a patient is having difficulty tolerating the steroid premedication regimen (e.g., patient develops uncontrolled hyperglycemia, altered mental status, or other complication), then lowering of the steroid premedication may be allowed for that patient after consultation with the medical monitor.
- If after consultation with the medical monitor, it is agreed that an individual patient's steroid premedication will be lowered, then the following steps **must be followed**:
  - 1) If the current steroid dosage is 10 mg or less of intravenous dexamethasone or equivalent, then the patient may be lowered in increments no greater than 2.5 mg intravenous dexamethasone or equivalent.
  - 2) After each incremental lowering of intravenous dexamethasone or equivalent, the patient must receive three consecutive intravenous doses of patisiran without IRR and continued signs or symptoms of steroid intolerance before further reductions in steroid premedications.
  - 3) The premedication steroid dosage should not be reduced below 5 mg intravenous dexamethasone or equivalent.

Alternatively if a patient experiences an IRR when 10 mg or less of IV dexamethasone or equivalent is used as the steroid premedication, then proceed to Section 6.4.3.

If a patient's premedication regimen was modified prior to enrollment in Study TTR02-006, the patient may continue on that modified premedication regimen.

### **6.4.2.** Study Drug Administration

Patisiran will be administered under the supervision of the site personnel every  $21 (\pm 3)$  days. Patients who have received at least 3 doses of patisiran on this study at the clinical site with no evidence of IRRs or other adverse effects may have patisiran administered at home, where applicable country and local regulations allow. Home administration of patisiran will be done by a healthcare professional trained on the protocol and delivery of premedications and patisiran.

On all dosing days, patisiran will be administered as a 70-minute IV infusion (approximately 1 mL/minute for the first 15 minutes followed by approximately 3 mL/minute for the remainder of the infusion).

- If the patient experiences an IRR the infusion time may be extended up to 3 hours in the event of a mild or moderate IRR.
  - 1) If the patient experiences a mild or moderate IRR that resolves by slowing the infusion rate then no further premedication changes are recommended.
  - 2) If the patient experiences a severe IRR, then patisiran administration will not be resumed until the case is discussed with the Medical Monitor (see Section 6.4.3).
- If the infusion time for a patient was already extended on the parent study due to an IRR, that modified infusion duration may be continued on this study for that particular patient.

  Returning the patient's infusion duration to 70 minutes will require a discussion with the Medical Monitor
- For the first 3 infusions of patisiran on this study, the patient's infusion site should be assessed for signs of any localized reaction during the infusion and for 30 minutes after the end of the infusion, and the patient will remain at the clinical site for 1 hour following completion of dosing.

If a patient does not receive a dose of patisiran within the dosing window (±3 days), the dose will be considered missed and not administered.

Additional details can be found in the patisiran Pharmacy Manual.

In addition to study treatment, patients will receive the recommended daily allowance of vitamin A . Patients will receive this daily dose for the duration of their participation in the study while being administered patisiran. In Japan the clinical sites will provide the subjects with a prescription for vitamin A..

### 6.4.3. Suggested Guidelines for Management of Infusion-Related Reactions

Criteria for categorizing IRRs are provided in Appendix 3.

- In the event of an IRR, the infusion of patisiran may be stopped and the patient closely monitored until resolution of the reaction. Drugs that may be used to facilitate resolution and permit resumption of patisiran administration include, but are not limited to: paracetamol/acetaminophen (or equivalent), additional histamine H1/H2 receptor antagonists (eg, ranitidine), NSAIDs, adrenaline, supplemental oxygen, IV fluids, and/or corticosteroids.
- Following resolution of a mild or moderate IRR that required interruption of the patisiran infusion, resumption of administration may occur at the Investigator's discretion at a slower

infusion rate (but not to exceed 3 hours) for that dose and for all subsequent doses of patisiran. If the infusion is delayed, the administration of the infusion should be completed no more than 6 hours from the initial start of the infusion.

- Patisiran administration will not be resumed for any patient following a severe IRR until the case is discussed with the Medical Monitor.
- If after consultation with the Medical Monitor it is agreed that an individual patient's steroid premedication will be increased then the following steps are **recommended**:
  - If the IRR occurred while the patient received 10 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and did not resolve with slowing of the infusion rate, then the patient should be increased by multiples of 5 mg intravenous dexamethasone or equivalent at least 60 minutes before the infusion and/or 5 mg oral dexamethasone or equivalent the night before the intravenous infusion.
  - 2) Increased dose of premedication steroids should NOT exceed the combination of 20 mg intravenous dexamethasone or equivalent on the day of infusion and 8 mg oral dexamethasone or equivalent taken the night before the infusion.
  - 3) If the IRR occurred while the patient received less than 10 mg intravenous dexamethasone or equivalent, then the patient should return to the prior dose of intravenous dexamethasone or equivalent that did not result in an IRR.

Patients will be instructed to call the Investigator if they experience symptoms such as fever, chills, myalgia, or nausea/vomiting after discharge from the site.

## 6.5. Study Drug Accountability

The Investigator or designee (or in Japan, the responsible pharmacist designated according to the Japan local regulations) will maintain accurate records of receipt and the condition of the patisiran supplied for this study, including dates of receipt. In addition, accurate records will be kept of the weight used to calculate each dispensed patisiran dose, and when and how much patisiran is dispensed and used by each patient in the study. Any reasons for departure from the protocol dispensing regimen must also be recorded.

Drug accountability records and inventory will be available for verification by the Sponsor or designee.

Further instructions about drug accountability are detailed in the patisiran Pharmacy Manual.

## 6.6. Study Drug Handling and Disposal

All used, partially used, and unused vials of patisiran will be returned to the Sponsor or its specified designee/depot or destroyed at the site according to applicable regulations.

Patisiran supplied for this study must not be used for any purpose other than the present study. Drug that has been dispensed for a patient and returned unused must not be redispensed.

## 7. PHARMACOKINETIC ASSESSMENTS

No PK assessments will be performed in this study.

### 8. ASSESSMENT OF EFFICACY

## 8.1. Efficacy Parameters

Efficacy assessments may be performed at Day 0 if not performed during the parent study within 45 days of the first dose in this study. Efficacy assessments will occur for all patients at the 52-week visit, which will take place at the CAS. Patients will not receive study drug at this visit. A subset of the efficacy assessments performed at 52 weeks will be performed annually thereafter. The specific timing for each assessment is presented in Table 1.

For the 52-week time point, a central neurologic testing core facility will review the data derived from the various neuropathy measures at each participating site to ensure compliance with testing procedures and quality of the data. A central echocardiography core lab will analyze the echocardiogram data. A core lab will be responsible for processing and analyzing skin punch biopsy samples. Magnetic resonance (MR) neurography data (when performed) will also be centrally read.

Further details on performing the efficacy assessments will be provided in the Study Reference Manual.

### 8.1.1. Neurological Testing

Neurological testing will be performed and the results of these tests will be used to calculate the Neuropathy Impairment Score (NIS), modified NIS (mNIS+7), and NIS+7, at the time points specified in Table 1.

## 8.1.1.1. Modified Neurological Impairment Score +7 and Neurological Impairment Score +7

The mNIS+7 assessment tool is a composite measure of neurologic impairment which includes the following measures:

- Clinical exam-based NIS (weakness and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - Nerve conduction studies (NCS) 5 attributes ( $\Sigma$ 5)
  - Quantitative sensory testing (QST) by body surface area including touch pressure (TP) and heat pain (HP)
- Autonomic function (postural blood pressure)

Neurologic impairment will also be assessed by NIS+7. The NIS+7 consists of the following measures:

- Full NIS (including weakness, sensation, and reflexes)
- Electrophysiologic measures of small and large nerve fiber function (+7) including:
  - NCS  $\Sigma 5$
  - Vibration detection threshold (VDT)
- Heart rate response to deep breathing (HRdb)

The scoring and components of the mNIS+7 and NIS+7 are summarized in Appendix 4. Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

Every effort will be made to use the same devices for NCS, QST, and VDT for a patient throughout the duration of the study.

For each patient, 2 independent assessments of the mNIS+7 and NIS+7 will be performed at each time point at a CAS. Assessments are to be performed at least 24 hours (approximately) apart from each other but no greater than 7 days apart. In order to limit potential intra-operator bias, results of any of the prior assessments will not be available to the examiner when performing the second assessment. Each site will make every effort to have these assessments at the Week 52 visit performed by the same study personnel who performed the assessments for the patient in the patisiran study in which they were previously enrolled. Assessments of the NIS during the annual visit (after the Week 52 visit) must be performed by a neurologist.

### 8.1.1.2. Neurological Impairment Score

At each time point when only the full NIS is required, 1 assessment of the NIS will be performed at a CAS or PCS.

## 8.1.2. Familial Amyloidotic Polyneuropathy Stage and Polyneuropathy Disability Score

Changes in ambulation will be evaluated through the polyneuropathy disability (PND) score and FAP stage (see Appendix 5 and Appendix 6, respectively).

### 8.1.3. Intraepidermal Nerve Fiber Density and Sweat Gland Nerve Fiber Density

Quantification of nerve fibers in skin will be assessed via intraepidermal nerve fiber density (IENFD) and sweat gland nerve fiber density (SGNFD). For patients who had skin biopsies on the parent study and who have provided additional voluntary consent for skin biopsy on this study, 2 sets of tandem 3-mm skin punch biopsies (4 biopsies total) for IENFD and SGNFD will be obtained at each time point. One set of biopsies will be taken from the distal lower leg, when a patient's clinical status allows, and 1 set from the distal thigh.

Details on sample collection, processing, and storage will be provided in the Study Laboratory Manual.

Skin biopsies will be performed at a CAS or PCS.

### 8.1.4. Magnetic Resonance Neurography (Germany and France Only)

Magnetic resonance (MR) neurography will only be performed at sites in Germany and France. Magnetic resonance neurography enables direct high-resolution longitudinal and cross-sectional images for the evaluation of peripheral nerve disorders. <sup>16</sup> This procedure produces detailed images of nerve morphology to evaluate degeneration and regeneration. Nerves in the lumbar plexus and lower extremity may be imaged for patients in Germany and France who have previously had MR neurography in the parent study and for a subset of patients providing informed consent who did not have MR neurography previously in the parent study. A central reader will be used for MR neurography.

### 8.1.5. Modified Body Mass Index

Sites will measure body weight on all dosing days. Using that data, the modified body mass index (mBMI) will be calculated (BMI × albumin) programmatically in the clinical database and does not need to be performed at the study center.

### 8.1.6. Timed 10-meter Walk Test

To perform the timed 10-meter walk test, the patient will be asked to walk 10 meters. The walk must be completed without assistance from another person; ambulatory aids such as canes and walkers are permitted. The time required for the patient to walk 10 meters will be recorded.

Two assessments of the 10-meter walk test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment. Each site will make every effort to have this assessment performed by the same Investigator.

## 8.1.7. Grip Strength Test

Hand grip strength is to be measured by dynamometer. Sites will be trained on dynamometer and testing for the study. When performing the test, patients will stand, holding the dynamometer in their dominant hand, with their arm parallel to the body without squeezing the arm against the body. Tests will be performed in triplicate for each assessment. Two assessments of the grip strength test are to be conducted on separate days (1 assessment on each day). The second (repeat) assessment must be conducted at least 24 hours (approximately) but not more than 7 days after the first assessment.

Every effort will be made to use the same dynamometer for a patient on both assessment days.

### 8.1.8. Composite Autonomic Symptom Score

To evaluate changes in autonomic symptoms, patients will complete the Composite Autonomic Symptom Score (COMPASS 31) questionnaire. The questionnaire consists of 31 clinically selected questions evaluating 6 autonomic domains (orthostatic intolerance, secretomotor, gastrointestinal, bladder, and pupillomotor).

### 8.1.9. Norfolk Quality of Life - Diabetic Neuropathy Questionnaire

Quality of life will be assessed through the Norfolk Quality of Life - Diabetic Neuropathy (QOL-DN) questionnaire, a standardized 47-item patient-reported outcomes measure that is sensitive to the different features of diabetic neuropathy (DN)-small fiber, large fiber, and autonomic nerve function.

Patients who are entering this study from a protocol that does not include the Norfolk QOL-DN questionnaire (eg, ALN-TTR02-003) will not complete this assessment.

### 8.1.10. EuroQoL Quality of Life Questionnaire

Quality of life will also be assessed through the use of the EuroQOL (EQ-5D) questionnaire, a standardized 5 question instrument for use as a measure of health outcomes.

### 8.1.11. Rasch-built Overall Disability Scale

An assessment of the disability each patient experiences will be assessed through the Rasch-built Overall Disability Scale (R-ODS). The R-ODS consists of a 24-item linearly weighted scale that specifically captures activity and social participation limitations in patients.

### **8.1.12.** Pharmacoeconomics Ouestionnaire

The burden of disease and healthcare utilization will be assessed using a patient-reported pharmacoeconomics questionnaire. This assessment will be performed at the location of the patient's scheduled visit.

### 8.1.13. Echocardiogram and Biomarkers of Cardiac Function

Cardiac structure and function will be assessed through echocardiograms and measurement of serum levels of the cardiac biomarkers N-terminal prohormone of B-type natriuretic peptide (NT-proBNP) and troponin I.

Echocardiograms will be performed and interpreted at a central echocardiography core laboratory. Patients entering this study from Study ALN-TTR02-003 who were not previously participating in the cardiac subgroup study will also be required to have an echocardiogram performed before dosing on Day 0. Image acquisition, storage, and transfer guidelines will be provided in a Study Manual.

Blood samples will be drawn to measure levels of NT-proBNP and troponin I. Details on sample collection, processing, and storage will be provided in a Study Laboratory Manual.

### 8.1.14. Transthyretin

Blood for serum TTR levels will be collected at scheduled time points before the administration of patisiran. Serum TTR will be assessed using enzyme linked immunosorbent assay (ELISA).

### **8.1.15.** Thyroid-Stimulating Hormone

Blood for TSH levels will be collected at scheduled visits.

### 8.1.16. Vitamin A

Blood for serum vitamin A levels will be collected at scheduled visits before the administration of vitamin A

### 8.1.17. Anti-Drug Antibodies

Serum samples for anti-drug antibodies will be collected as specified in Table 1.

### 8.1.18. Blood Sample for Long-term Storage

To permit exploratory investigations and the application of novel approaches to bioanalysis that may further elucidate the outcomes of this study, or potentially advance understanding of the safety, mechanism of action and/or efficacy of patisiran, blood samples will be collected for long-term storage. These samples will be securely stored in a central biorepository for up to 10

years following the last patient last visit in this clinical study. After 10 years have elapsed, samples will be destroyed.

Details regarding the collection, processing, storage, and shipping of samples will be provided in the Laboratory Manual.

Exploratory analysis of these biospecimens will be performed by Alnylam Pharmaceuticals or its designees.

All study participants will be advised during the informed consent process of these biobanking details and the potential for exploratory investigation of their samples. Those who do not wish to contribute specimens to the biorepository will be asked to sign an "opt out" form. Moreover, patients who subsequently decide to withdraw consent for the utilization of such stored samples will be able to do so, with the understanding that any data arising from samples already analyzed will be the property of Alnylam Pharmaceuticals.

### 9. ASSESSMENT OF SAFETY

### 9.1. Safety Parameters

All safety assessment measures will be recorded in the patient's medical record and CRF. Refer to Table 1 for the timing of each safety assessment.

### 9.1.1. Demographic and Medical History

Patient demographic data will be obtained from the parent study.

The Investigator will assess all patients according to the Karnofsky Scale (see Appendix 1) and the New York Heart Association Classification of Heart Failure (NYHA; see Appendix 2).

For all patients, a complete medical history will be obtained, including TTR genotype. Any AEs from the parent study that are ongoing on Day 0 will be considered as part of the medical history.

### 9.1.2. Vital Signs

Vital signs will be measured pre-dose on all dosing days. Vital signs include systolic/diastolic blood pressure, heart rate, respiratory rate, and body temperature, and will be measured in the supine position using an automated instrument after the patient has rested comfortably for 10 minutes. Each patient's blood pressure should be taken using the same arm. Temperature will be recorded in Celsius or Fahrenheit. Heart rate will be counted for a full minute and recorded in beats per minute. Respirations will be counted for a full minute and recorded in breaths per minute.

For the safety of the patient, additional vital signs may be obtained at the discretion of the Investigator.

### 9.1.3. Weight and Height

Body weight will be measured on all dosing days to inform the next infusion dosing calculation. The rules for using body weight to calculate dose are described in Section 6.4.2.

Height will be measured only if it was not obtained in the parent study.

### 9.1.4. Physical Examination

A physical examination will be performed by a physician before dosing at scheduled time points. The physical examinations will include the examination of the following: general appearance; head, ears, eyes, nose, and throat; cardiovascular; dermatologic; abdominal; genito-urinary; lymph nodes; hepatic; musculoskeletal; respiratory; and neurological.

### 9.1.5. Laboratory Assessments

Blood samples for clinical laboratory testing will be collected before patisiran dosing at the time points listed in Table 1. All samples will be sent to a central laboratory for analysis. Details on sample collection, processing, and shipping will be provided in a Laboratory Manual.

In the event of an unexplained clinically relevant abnormal laboratory test occurring after patisiran administration, the test should be repeated and followed up at the discretion of the Investigator until it has returned to the normal range or stabilized, and/or a diagnosis is made to adequately explain the abnormality.

### 9.1.5.1. Hematology

Blood samples will be collected for evaluation of the following hematology parameters:

- Hematocrit
- Hemoglobin
- Red blood cell (RBC) count
- White blood cell (WBC) count
- Mean corpuscular volume
- Mean corpuscular hemoglobin
- Mean corpuscular hemoglobin concentration

- Neutrophils, absolute and %
- Lymphocytes, absolute and %
- Monocytes, absolute and %
- Eosinophils, absolute and %
- Basophils, absolute and %
- Platelet count

### 9.1.5.2. Blood Chemistry

Blood samples will be collected for evaluation of the following chemistry parameters:

- Aspartate transaminase (AST)
- Alanine transaminase (ALT)
- Sodium
- Potassium
- Blood urea nitrogen (BUN)
- Creatinine

- Alkaline phosphatase
- Bilirubin (total and direct)
- Glucose
- Phosphate
- Albumin
- Calcium

### **9.1.5.3.** Urinalysis

Urine samples will be collected for evaluation of the following urinalysis parameters:

- Visual inspection for color and appearance
- pH
- Specific gravity
- Ketones
- Protein
- Glucose

- Leukocytes
- Bilirubin
- Nitrite
- Urobilinogen
- Microscopic inspection of sediment

### 9.1.5.4. Coagulation

A sample for INR assessment will be collected.

### 9.1.5.5. Pregnancy Screen

Urine pregnancy tests are to be performed for all women of child-bearing potential. The timing of the tests is specified in in Table 1; additional testing may be done any time pregnancy is suspected.

### 9.1.6. Ophthalmology Examination

Ophthalmology examinations will include assessment of visual acuity, visual fields, and slitlamp evaluation. Visual acuity should be evaluated at the beginning of each specified visit in the study (ie, prior to slit-lamp examination). Manifest refraction will be performed at each specified visit before visual acuity testing and will be used to obtain a correction for visual acuity evaluations. Visual acuity testing should be done with best (most recent) correction.

An electroretinogram (ERG) is a test to evaluate the retinal response to light. It is done to determine if there is damage to rods and cones. ERG testing should be performed if visual changes raise the suspicion for this sort of retinal disease and if clinically indicated.

Further details regarding the ophthalmology examinations will be provided in the Study Reference Manual.

### 9.1.7. Columbia-Suicide Severity Rating Scale

The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess each patient's mental status as it relates to suicidal ideation and behavior. If a patient's C-SSRS raises concern of suicidal ideation or behavior, the Investigator must ensure prompt and appropriate mental health interventions in accordance with standard of care.

### 9.2. Adverse Events and Serious Adverse Events

### 9.2.1. Definition of Adverse Events

### 9.2.1.1. Adverse Event

An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Disease progression (including worsening of neuropathy impairment) will not be considered an AE.

All IRRs will be recorded as AEs.

### 9.2.1.2. Serious Adverse Event

A serious AE (SAE) is any untoward medical occurrence that at any dose:

- Results in death
- Is life-threatening (an event which places the patient at immediate risk of death from the event as it occurred; it does not include an event that had it occurred in a more severe form might have caused death)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly or birth defect
- An important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the other outcomes listed in the definition above (eg, such events include allergic bronchospasm, blood dyscrasias or convulsions, or the development of drug dependency or abuse)

## 9.3. Relationship to Study Drug

Causal relationship assessment to drug treatments is required for purposes of reporting AEs. To promote consistency, the following guidelines should be taken into consideration along with good clinical and scientific judgment when determining the relationship of drug treatments to an AE:

Definitely Related: A clinical event, including laboratory test abnormality, occurring in a

plausible time relationship to the medication administration, and which cannot be explained by concurrent disease or other drugs or chemicals. The response to withdrawal of the drug should be clinically plausible.

Possibly Related: A clinical event, including laboratory test abnormality, with a reasonable

time sequence to the medication administration, but which could also be explained by concurrent disease or other drugs or chemicals. Information

on the drug withdrawal may be lacking or unclear.

Unlikely Related: A clinical event, including laboratory test abnormality, with little or no

temporal relationship to medication administration, and which other drugs.

chemicals, or underlying disease provide plausible explanations.

Not Related: A clinical event, including laboratory test abnormality, that has no

temporal relationship to the medication or has more likely alternative

etiology.

## 9.4. Recording Adverse Events

The patient should be asked about medically relevant changes in his/her health since the last visit. The patient should also be asked if he/she has been hospitalized, had any accidents, used any new medications, or changed concomitant medication routines (both prescription and OTC).
In addition to patient observations, AEs will be documented from any clinically relevant laboratory findings, physical examination findings, or other findings.

Adverse events are to be graded according to the categories detailed below.

Mild: Mild events are those which are easily tolerated with no disruption of normal

daily activity.

Moderate: Moderate events are those which cause sufficient discomfort to interfere with

daily activity.

Severe: Severe events are those which incapacitate and prevent usual activity.

Changes in severity should be documented in the medical record to allow assessment of the duration of the event at each level of severity. Adverse events characterized as intermittent require documentation of the start and stop of each incidence. When changes in the severity of an AE occur more frequently than once a day, the maximum severity for the experience that day should be noted. If the severity category changes over a number of days, then those changes should be recorded separately (with distinct onset dates).

# 9.5. Reporting Adverse Events

The Investigator is responsible for reporting all AEs that are observed or reported after the first dose of patisiran regardless of their relationship to patisiran administration through the end of the study.

Any medical condition that is present when the patient enters this extension study and does not deteriorate should not be reported as an AE. However, if it does deteriorate at any time during the study, it should be reported as an AE.

All AEs must be fully recorded in the site's source records and in the patients' CRF, whether or not they are considered to be drug-related. Each AE should be described in detail: onset time and date, description of event, severity, relationship to investigational product, action taken, and outcome (including time and date of resolution, if applicable).

Adverse events should be followed through the end of study visit or until recovery to the normal state has been achieved, whichever occurs first. In the event of a patient not returning to the clinical unit, the outcome of this event will be recorded as lost to follow-up.

For patients who withdraw from the study early, ongoing AEs will be followed until resolution or 28 days from last dose, whichever occurs first. SAEs will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable.

# 9.5.1. Serious Adverse Event Reporting

An assessment of the seriousness of each AE will be made by the Investigator. Any AE and laboratory abnormality that meets the above seriousness criteria (Section 9.2.1.2) must be reported immediately to the CRO, always within 24 hours from the time that site personnel first learn of the event. All SAEs must be reported regardless of the relationship to patisiran.

The initial report should include at least the following information:

• Patient's study number

- Description and date of onset of the event
- Criterion for serious
- Preliminary assignment of causality

Serious AE reporting will be via electronic data capture (EDC).

To report the SAE, complete the SAE form electronically in the EDC system for the study. If the event meets serious criteria and it is not possible to access the EDC system, send an email to Medpace Safety at PPD or call the Medpace SAE hotline listed below (country-specific phone number will be provided in the Study Manual), and fax the completed back-up paper SAE form to Medpace (country-specific fax number will be provided in the Study Manual) within 24 hours of awareness. When the form is completed, Medpace Safety personnel will be notified electronically and will retrieve the form. When the EDC system becomes available, the SAE information must be entered into the EDC system within 24 hours of the system becoming available. Medpace Safety personnel will be available for SAE reporting on a 24 hour basis. Incoming reports will be reviewed during normal business hours.



Within 24 hours of receipt of follow-up information, the investigator must update the SAE form electronically in the EDC system for the study and submit any supporting documentation (eg, patient discharge summary or autopsy reports) to Medpace Safety personnel via fax or email. If it is not possible to access the EDC system, refer to the procedures outlined above for initial reporting of SAEs.

Appropriate remedial measures should be taken by the Investigator using his/her best medical judgment to treat the SAE. These measures and the patient's response to these measures should be recorded. All SAEs, regardless of causality, will be followed by the Investigator until satisfactory resolution or the Investigator deems the SAE to be chronic or stable. Clinical, laboratory, and diagnostic measures should be employed by the Investigator as needed to adequately determine the etiology of the event.

The Investigator will be responsible for reporting all SAEs to the local IEC or IRB when required by national regulations.

The Sponsor or its representative will be responsible for the reporting of all relevant events to the concerned regulatory authorities according to all applicable regulations.

In Europe, in accordance with the Directive 2001/20/EC, the Competent Authorities and the Ethics Committees in the concerned Member States will be notified of fatal and life-threatening Suspected Unexpected Serious Adverse Reactions (SUSARs) as soon as possible but no later than 7 calendar days after the Sponsor or its representative has first knowledge of the minimum criteria for expedited reporting. Non-fatal and non-life-threatening SUSARs should be reported no later than 15 calendar days after the Sponsor or its representative has first knowledge of them.

The Investigator may be informed by the Sponsor or its representative of SAEs from other Investigators or clinical studies which may have relevance to this clinical study. These SAEs should also be reported promptly to the IEC/IRB that approved the study. All SAE reports should be transmitted to the IEC/IRB with a cover letter or transmittal form, and a copy of that transmittal should be maintained in the Investigator's files and forwarded to the Sponsor as part of the trial master file on study completion.

### 9.5.2. Pregnancy Reporting

A female patient must have a negative pregnancy test within 14 days before the first dose of patisiran on this study. If a female patient is found to be pregnant during the course of the study or during the first month after receiving the last dose of patisiran, the Investigator should report the pregnancy to the CRO within 24 hours of being notified of the pregnancy. Details of the pregnancy will be recorded on the pregnancy reporting form. Treatment with patisiran will be discontinued in any patient who is found to be pregnant during the study. The patient should receive any necessary counseling regarding the risks of continuing the pregnancy and the possible effects on the fetus.

The pregnancy should be followed by the Investigator until completion. At the completion of the pregnancy, the Investigator will document the outcome of the pregnancy. If the outcome of the pregnancy meets the criteria for an SAE (ie, postpartum complication, spontaneous abortion, stillbirth, neonatal death, or congenital anomaly), then the Investigator should follow the procedures for reporting an SAE outlined above.

Pregnancy occurring in the partner of a patient participating in the study should also be reported to the Investigator, who will then report this to the CRO and follow to outcome as described above.

### 10. STATISTICS

# 10.1. Sample Size

This is an open-label extension study enrolling patients who have previously completed a patisiran study; the size of the study is not determined via power analysis of particular hypotheses tests.

# 10.2. Statistical Methodology

Statistical analyses will be primarily descriptive in nature.

For categorical variables, summary tabulations of the number and percentage of patients within each category (with a category for missing data) will be presented. For continuous variables, the number of patients, mean, median, standard deviation, minimum, and maximum values will be presented.

All data will be provided in by-patient listings.

### 10.2.1. Populations to be Analyzed

The following patient populations (ie, analysis sets) may be evaluated and used for presentation of the data:

- Full Analysis Set: All patients who were enrolled will be included in the full analysis set. The full analysis set will be the primary set for the analysis of efficacy data.
- Safety Analysis Set: All patients in the full analysis set who received patisiran. The safety analysis set will be used for the analysis of safety assessments.

#### 10.2.2. Baseline Evaluations

Demographic information and baseline disease characteristic data collected in the parent study will be summarized. Data to be tabulated will include sex, age, and race, as well as disease-specific information.

#### 10.2.3. Efficacy Analyses

Associations between PD (serum TTR) and efficacy data will be explored via correlation.

Summary statistics of observed values and changes from baseline will be provided for the mNIS +7 composite score. Summaries will also be provided for the components of the composite score (ie, the NIS weakness and reflex scores, the  $\Sigma$ 5 NCS, and QST values). The NIS+7 score (including full NIS, NCS, VDT, and HRdb), and full NIS will be summarized also.

Patient reported quality of life and disease burden will be assessed by summary statistics for the EQ5D and R-ODS. Summary statistics will be provided for observed values and changes from baseline. Patient reported autonomic neuropathy symptoms will be assessed by descriptive statistics for the COMPASS 31.

Descriptive statistics will also be provided for observed values and changes from baseline in motor function (10-meter walk test and test of grip strength), nutritional status (mBMI), sensory

and autonomic innervation (IENFD and SGNFD), VDT, and ambulation (FAP stage and PND score).

Summary tables and graphical displays of observed values and changes from baseline in serum TTR will be used to assess the durability of suppression over the course of the study.

Descriptive statistics will be provided for actual values and changes from baseline in serum levels of troponin I and NT-proBNP in the subset of patients with evidence of pre-existing cardiac amyloid involvement. Results of echocardiograms will be summarized.

#### 10.2.4. Safety Analyses

A summary of exposure to patisiran, including the durations of the infusions and doses, and the proportions of patients with modifications in the durations of infusions will be produced.

Adverse events will be summarized by the Medical Dictionary for Regulatory Activities (MedDRA) system organ class and preferred term. Separate tabulations will be produced for all treatment emergent AEs, treatment-related AEs (those considered by the Investigator as at least possibly drug related), SAEs, and discontinuations due to AEs, and AEs by severity. By-patient listings will be provided for deaths, SAEs, and events leading to discontinuation of treatment.

Descriptive statistics will be provided for clinical laboratory data and vital signs data, presented as both actual values and changes from baseline relative to each on-study evaluation and to the last evaluation on study. Laboratory shift tables from baseline to worst values will be presented.

#### 10.2.5. Healthcare Utilization Assessments

A listing of healthcare utilization data will be presented.

#### 10.2.6. Interim Analysis

Interim data examinations may be performed, but these will be of a descriptive nature and will not involve any formal hypothesis testing.

723

## 11. DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

# 11.1. Study Monitoring

The Clinical Monitor, as a representative of the Sponsor, has an obligation to follow the study closely. In doing so, the Monitor will visit the Investigators and sites periodically and maintain frequent telephone and written contact. The Monitor will maintain current personal knowledge of the study through observation, review of study records and source documentation and discussion of the conduct of the study with the Investigator and staff.

All aspects of the study will be carefully monitored by the Sponsor or its designee for compliance with applicable government regulations in respect to Good Clinical Practice (GCP) and current standard operating procedures.

# 11.2. Audits and Inspections

The Investigator and the site will permit study-related monitoring, audits and review by the IEC or IRB and/or Regulatory Authorities, providing direct access to source data/documents. The study may be subject to audit by the Sponsor or its representatives or by regulatory authorities. If such an audit occurs, the Investigator must agree to allow access to the required patient records. In the event of an audit, the Investigator agrees to allow the Sponsor, representatives from the Sponsor, or regulatory agencies access to all study records.

## 11.3. Institutional Review Board

The Investigator must obtain IRB or IEC approval for the investigation. Initial IRB approval, and all materials approved by the IRB for this study including the patient consent form and recruitment materials must be maintained by the Investigator and made available for inspection.

# 12. QUALITY CONTROL AND QUALITY ASSURANCE

Study personnel are expected to adhere to the following practices, governed by GCP and all applicable regulatory requirements. To ensure these practices are in place, the Sponsor may conduct a quality assurance audit.

The Investigator will submit reports of SAEs as outlined in this protocol. In addition, the Investigator agrees to submit progress reports to his/her IRB or IEC per their local reporting requirements, or at least annually and at the conclusion of the study. The reports will be made available to the Sponsor or designee.

Deviations from the protocol necessary to protect patient safety should be reported to the CRO within 24 hours of knowledge of the event.

Any communications from regulatory agencies in regard to inspections, other studies that impact this protocol or the qualifications of study personnel should be promptly reported to the CRO.

Major changes in this research activity, except those to remove an apparent immediate hazard to the patient, must be reviewed and approved by the Sponsor and the IRB or IEC that approved the study. Amendments to the protocol must be submitted in writing to the Investigator's IRB or IEC and the Regulatory Authority for approval before patients are enrolled under the amended protocol.

Regulatory authorities will receive the protocol, amendments, reports on SAEs, and the Integrated Clinical Trial Report according to national and any local regulations.

### 13. ETHICS

#### 13.1. Ethics Review

National regulations and International Conference on Harmonization (ICH) require that approval be obtained from an IRB or an IEC prior to participation of patients in research studies. Prior to the study onset, the protocol, any protocol amendments, informed consent forms (ICFs), and any other written information regarding this study to be provided to a patient or patient's legal guardian must be approved by the IRB or IEC.

All IRB and IEC approvals must be dated and contain IRB/IEC Chairman or designee authorization and must identify the IRB/IEC (eg, name and address), the clinical protocol by title and/or protocol number, and the date of approval or favorable opinion was granted for the clinical research.

The Investigator should not start any study procedure with the patient until documentation of the approval by the IEC/IRB and written notification of the approval from the head of the study site to the Investigator and Alnylam Pharmaceuticals, Inc.

No drug will be released to the site to dose a patient until written IRB/IEC authorization has been received by the Sponsor or designee.

The Investigator is responsible for obtaining continuing review of the clinical research at least annually or more often if specified by the IRB or IEC. The Investigator must supply the Sponsor with written documentation of the approval of the continued clinical research.

The Investigator will make all attempts to ensure that the IRB or IEC is constituted and operates in accordance with Federal and ICH GCP and any local regulations.

# 13.2. Ethical Conduct of the Study

This study will be performed in accordance with the clinical trial agreement, the protocol, all applicable government laws, regulations, and guidances where the study is being conducted including policies with foundations in the World Medical Association Declaration of Helsinki, the ICH of Technical Requirements for Registration of Pharmaceuticals for Human Use, the Health Insurance Portability and Accountability Act of 1996 (HIPAA) in the US, and all other applicable medical privacy laws and regulations.

#### 13.2.1. Financial Disclosure Reporting Obligations

Each Investigator (including Principal and any Sub Investigators) directly involved in the treatment or evaluation of study patients is required to provide financial disclosure information according to all applicable legal requirements. In addition, Investigators must commit to promptly updating this information if any relevant changes occur during the study and for a period of one year after the completion of the study.

## 13.3. Written Informed Consent

Written informed consent in compliance with 21 Code of Federal Regulations (CFR) § 50 and ICH will be obtained from each patient before undergoing any protocol-specific tests or procedures that are not part of routine care.

The Sponsor or the CRO designee will provide an ICF template to the Investigator for use in developing a site-specific ICF. Prior to submission of the site-specific ICF to the IRB or IEC, the site-specific ICF must be reviewed and approved by the Sponsor or designee. Any changes requested by the IRB or IEC must also be agreed upon. The final IRB/IEC approved ICF must be provided to the Sponsor. Revisions to the ICF required during the study must be agreed upon, and a copy of the revised ICF provided to the Sponsor.

At the time of recruitment, each prospective patient (or legal guardian) will be given a full explanation of the study and be allowed to read the ICF. Once the Investigator is assured that the patient/legal guardian understands the commitments of participating in the study, the patient/legal guardian will be asked to sign and date the ICF. A copy of the fully signed and dated ICF will be given to the patient. The original ICF will be maintained in the patient's medical record at the site. All active patients will sign an updated ICF if revisions are made to the ICF during the course of the study.

Prior to dosing in this study, the patient will sign and date the ICF and receive a copy of the signed ICF. No study procedures should be performed before informed consent is obtained. The Investigator or another person authorized by the Investigator will also sign and date the informed consent before giving a copy to the patient. The ICF will be filed in the patient's medical record.

# 13.4. Compensation for Health Damages

A copy of the certificate of insurance as a measure to compensation for health damages will be submitted to the IRB/IEC if required per local regulations.

727

## 14. DATA HANDLING AND RECORD KEEPING

## 14.1. Case Report Forms

The Investigator and designees agree to maintain accurate CRFs and source documentation as part of these case histories. Source documents are the originals of any documents used by the Investigator or hospital/institution that allow verification of the existence of the patient and substantiate the integrity of the data collected during the trial.

The Sponsor will supply CRFs for each patient. Case report forms must be completed only by persons designated by the Investigator. Corrections must be made so as not to obliterate original data and must be identified and dated by the person who made the correction. All data entered into the CRF must also be available in the source documents. The Investigator will allow designated Sponsor representatives and regulatory bodies to have direct access to the source documents to verify the data reported in the CRFs.

Each completed CRF must be reviewed and signed by the Investigator or designee in a timely manner. The completed CRF will be the records maintained by the Sponsor. A copy of the CRF will remain in the Investigator's files.

# 14.2. Confidentiality

The Investigator must ensure that the patients' anonymity will be maintained. On the CRFs or other documents submitted to the Sponsor or designees, patients should not be identified by their names, but by the assigned patient number and initials. If patient names are included on copies of documents submitted to the Sponsor or designees, the names (except for initials) will be obliterated and the assigned patient number added to the document. Documents not for submission to the Sponsor (eg, signed ICFs) should be maintained by the Investigator in strict confidence.

Following the principles of the GCP, if local regulations specify a patient's number and initials will be used to identify the patient on their study records. Laboratory samples may be labeled with an independent numbering code, and the label will not contain any other personal identification information. The numbering code associated with these labels will be held by the study CRO and the Sponsor, thereby allowing no unwarranted access to the information. The numbering code will also be held for samples in storage until marketing approval of patisiran in the countries where this study was conducted, or until clinical development of patisiran is halted. Throughout sample collection, storage (limited, staff only access area containing locked sample storage, and limited access sample tracking) and processing, the samples will only be handled by appropriate personnel per the laboratory's standard operating procedures.

The Investigator must treat all of the information related to the study and the compiled data as confidential, whose use is for the purpose of conducting the study. The Sponsor must approve any transfer of information not directly involved in the study.

# 14.3. Inspection of Records

The Sponsor will be allowed to conduct site visits to the investigation facilities for the purpose of monitoring any aspect of the study. The Investigator agrees to allow the Monitor to inspect the drug storage area, drug stocks, drug accountability records, patient charts and study source documents, and other records relative to study conduct.

#### 14.4. Retention of Records

Essential documents should be retained for the period of time required by applicable local law. The essential documents include the signed and dated final protocol, signed and dated amendments(s), if applicable, signed and dated curricula vitae of the Investigators, copies of the completed CRFs, signed ICFs, IEC/IRB approval and all related correspondence, financial agreements, regulatory approval, drug accountability, study correspondence, and patient identification codes. Records will not be destroyed without informing the Sponsor in writing and giving the Sponsor the opportunity to store the records for a longer period of time at the Sponsor's expense.

The ICH requires that patient identification codes be retained for at least 15 years after the completion or discontinuation of the study.

## 15. PUBLICATION POLICY

Following completion of the study, the data may be considered for publication in a scientific journal or for reporting at a scientific meeting. A copy of the manuscript must be provided and confirmed received at the Sponsor at least 30 days before its submission.

No submission of a manuscript may be made until the results from all of the clinical sites have been received and analyzed by the Sponsor, or the study has been terminated at all centers. A separate, individual publication of the results of the study will be delayed until initial publication of the results of the multicenter study, or a decision not to publish is made. If an initial draft is not produced within 18 months of completion of the study at all centers, or the timeframe for publication is not satisfactory, the Investigator may disclose the results after providing a copy and the Sponsor confirms receipt of the manuscript 30 days before submission.

Research ancillary to this main protocol may not be performed by individual sites without prior discussion and approval by the Sponsor.

### 16. LIST OF REFERENCES

Yazaki M., Tokuda T, et al. Cardiac amyloid in patients with familial amyloid polyneuropathy consists of abundant wild-type transthyretin. Biochem Biophys Res Commun. 2000; 274(3):702-706.

- 2 Gillmore JD, Hawkins PN. Drug Insight: emerging therapies for amyloidosis. Nat Clin Pract Nephrol. 2006. 2(5):263-70.
- Suhr OB, Herlenius G, et al. Liver transplantation for hereditary transthyretin amyloidosis. Liver Transpl. 2000;6(3): 263-276.
- 4 Benson MD. Familial amyloidotic polyneuropathy. Trends Neurosci. 1989;12(3):88-92.
- Connors LH, Yamashita T, et al. A rare transthyretin mutation (Asp18Glu) associated with cardiomyopathy. Amyloid. 2004;11(1):61-66.
- Buxbaum JN. (2007). Transthyretin and the Transthyretin Amyloidoses. Protein Reviews: Protein Misfolding, Aggregation, and Conformational Diseases. V. N. a. F. Uversky, A. New York, Springer US. 7: 259-283.
- Suhr OB. Impact of liver transplantation on familial amyloidotic polyneuropathy (FAP) patients' symptoms and complications. Amyloid. 2003;10 (Suppl 1):77-83.
- 8 Ando Y, Nakamura M, et al. Transthyretin-related familial amyloidotic polyneuropathy. Arch Neurol. 2005;62(7):1057-1062.
- 9 Coelho T, Adams D, Silva A, et al. Safety and Efficacy of an RNAi Therapeutic Targeting Transthyretin (TTR) for TTR Amyloidosis. NEJM. 2013, accepted for publication.
- Stangou AJ and Hawkins PN. Liver transplantation in transthyretin-related familial amyloid polyneuropathy. Current Opinion in Neurology. 2004;17(5):615-620.
- Akinc A, Zumbuehl A, et al. A combinatorial library of lipid-like materials for delivery of RNAi therapeutics. Nat Biotechnol. 2008;26(5):561-569.
- Adams D, Suhr O, Coelho T, et al. Phase 2 open-label extension study of patisiran, an RNAi therapeutic for the treatment of familial amyloidotic polyneuropathy. Presented at: Annual Meeting of the American Neurological Association; 2014 Oct 12; Baltimore, MD.
- Biesalski, H.K., et al., Biochemical but not clinical vitamin A deficiency results from mutations in the gene for retinol binding protein. Am J Clin Nutr, 1999. 69(5): p. 931-6.
- Episkopou, V., et al., Disruption of the transthyretin gene results in mice with depressed levels of plasma retinol and thyroid hormone. Proc Natl Acad Sci U S A, 1993. 90: p. 2375-2379.
- 15 Conceiciao IM, Miranda LC, et al. Bone mineral density in familial amyloid polyneuropathy and in other neuromuscular disorders. Eur J Neurol. 2005;12(6):480-2.
- Kollmer J, Hund E, Hornung B, Schönland S, et al. MR-neurography: In-vivo detection of nerve injury in systemic light chain (AL) amyloidosis. XIVth International Symposium on Amyloidosis, 2014.

731

# 17. APPENDICES

Appendix 1: Karnofsky Scale

| | 100 | Normal no complaints; no evidence of disease. |
|---|---|---|
| Able to carry on normal activity and to work; no special care needed. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| noodo. | 80 | Normal activity with effort; some signs or symptoms of disease. |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work. |
| home and care for most personal needs; varying amount of assistance needed. | 60 | Requires occasional assistance, but is able to care for most of his personal needs. |
| | 50 | Requires considerable assistance and frequent medical care. |
| Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly. | 40 | Disabled; requires special care and assistance. |
| | 30 | Severely disabled; hospital admission is indicated although death not imminent. |
| | 20 | Very sick; hospital admission necessary; active supportive treatment necessary. |
| | 10 | Moribund; fatal processes progressing rapidly. |
| | 0 | Dead |

# **Appendix 2: New York Heart Association Classification of Heart Failure**

| Class | Symptomatology |
|---|---|
| I | No symptoms. Ordinary physical activity such as walking and climbing stairs does not cause fatigue or dyspnea. |
| II | Symptoms with ordinary physical activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, in cold weather, in wind or when under emotional stress causes undue fatigue or dyspnea. |
| III | Symptoms with less than ordinary physical activity. Walking one to two blocks on the level and climbing more than one flight of stairs in normal conditions causes undue fatigue or dyspnea. |
| IV | Symptoms at rest. Inability to carry on any physical activity without fatigue or dyspnea. |

## **Appendix 3: Categorization of Infusion-Related Reactions**

Signs and symptoms of an infusion-related reaction (IRR) usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion. Signs/symptoms may include: allergic reaction/hypersensitivity (including drug fever), arthralgia (joint pain), bronchospasm, cough, dizziness, dyspnea (shortness of breath), fatigue (asthenia, lethargy, malaise), headache, hypertension, hypotension, myalgia (muscle pain), nausea, pruritus/itching, rash/desquamation, rigors/chills, sweating (diaphoresis), tachycardia, urticaria (hives, welts, wheals), vomiting.

Categorization of IRRs is as follows:

| Categorization | Description |
|---|---|
| Mild | Mild reaction: infusion may be continued; if intervention is indicated it is minimal and additional treatment (other than paracetamol for delayed reactions) is not required. |
| Moderate | Moderate reaction: requires treatment including more intensive therapy (eg, IV fluids, nonsteroidal anti-inflammatory drug [NSAIDs]) in addition to infusion interruption but responds promptly to medication. Treatment is indicated for ≤24 hours. |
| Severe | More than moderate reaction: not rapidly responsive to medication or to interruption of infusion; and/ or prolonged (treatment is indicated for >24 hours); recurrence of severe symptoms following initial improvement. |

# **Appendix 4: Neuropathy Scores and Their Components**

| Assessment Tool | Total<br>Points | Components (points) |
|---|---|---|
| NIS+7 | 270 | <ul> <li>Neurologic exam of lower limbs, upper limbs and cranial nerves (NIS<sup>a</sup>)</li> <li>Weakness (192)</li> <li>Sensation (32)</li> <li>Reflexes (20)</li> <li>Nerve conduction studies ∑5 (18.6)<sup>a</sup></li> <li>Sural SNAP, tibial motor n. distal latency, peroneal CMAP/motor n. conduction velocity/motor n. distal latency</li> <li>Vibration detection threshold (3.7)</li> <li>Heart rate response to deep breathing (3.7)</li> </ul> |
| Modified NIS+7 | 304 | <ul> <li>Neurologic exam of lower limbs, upper limbs and cranial nerves (mNIS<sup>a</sup>)</li> <li>Weakness (192)</li> <li>Reflexes (20)</li> <li>Nerve conduction studies ∑5 (10)<sup>a</sup></li> <li>Ulnar CMAP and SNAP, sural SNAP, tibial CMAP, peroneal CMAP</li> <li>Quantitative sensory testing: QST-BSA<sub>TP+HP5</sub> (80)</li> <li>Postural blood pressure (2)</li> </ul> |

a Components that are shared between the mNIS+7 and NIS+7 (including NIS and NCS) will be performed once at each assessment.

# **Appendix 5: Polyneuropathy Disability Score**

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Sensory disturbances but preserved walking capability |
| II | Impaired walking capacity but ability to walk without a stick or crutches |
| IIIA | Walking with the help of one stick or crutch. |
| IIIB | Walking with the help of two sticks or crutches. |
| IV | Confined to a wheelchair or bedridden. |

# Appendix 6: Familial Amyloidotic Polyneuropathy Stage

| Stage | Description |
|---|---|
| 0 | No symptoms |
| I | Unimpaired ambulation; mostly mild sensory, motor, and autonomic neuropathy in the lower limbs |
| II | Assistance with ambulation required, mostly moderate impairment progression to the lower limbs, upper limbs, and trunk. |
| III | Wheelchair-bound or bedridden; severe sensory, motor, and autonomic involvement of all limbs. |

## **ALN-TTR02-006 Protocol Version 3.1 United Kingdom**

Summary of Changes (dated 11 May 2017) compared to Protocol Version 3.0 (dated 05 January 2017)

A Multicenter, Open-label, Extension Study to Evaluate the Long-Term Safety and Efficacy of Patisiran in Patients with Familial Amyloidotic Polyneuropathy who have Completed a Prior Clinical Study with Patisiran

#### **Rationale for Protocol Amendment**

The purpose of this country-specific protocol amendment is to address comments (dated 28 February 2017) from the United Kingdom's National Health Service Ethics Committee

PPD Text has been added to the protocol detailing that if a patient's Columbia-Suicide Severity Rating Scale (C-SSRS) score raises concern of suicidal ideation or behavior, the Investigator must ensure prompt and appropriate mental health interventions in accordance with standard of care.

A detailed summary of changes is provided in Table 1.

1

## **Table 1: Protocol Amendment 2 Detailed Summary of Changes**

The primary section(s) of the protocol affected by the changes in the protocol amendment are indicated. The corresponding text has been revised throughout the protocol. Deleted text is indicated by strikeout; added text is indicated by bold font.

Purpose: Added text that if a patient's Columbia-Suicide Severity Rating Scale (C-SSRS) score raises concern of suicidal ideation or behavior, the Investigator must ensure prompt and appropriate mental health interventions in accordance with standard of care

The primary change occurs in Section 9.1.7, Columbia-Suicide Severity Rating Scale

Added text:

The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess each patient's mental status as it relates to suicidal ideation and behavior. If a patient's C-SSRS raises concern of suicidal ideation or behavior, the Investigator must ensure prompt and appropriate mental health interventions in accordance with standard of care.